CLINICAL TRIAL: NCT00809354
Title: A PHASE 3, MULTI-CENTER, RANDOMIZED, DOUBLE-BLIND, CONTROLLED STUDY OF THE LONG-TERM ANALGESIC EFFICACY AND SAFETY OF TANEZUMAB ALONE OR IN COMBINATION WITH NON-STEROIDAL ANTI-INFLAMMATORY DRUGS (NSAIDS) VERSUS NSAIDS ALONE IN PATIENTS WITH OSTEOARTHRITIS OF THE KNEE OR HIP
Brief Title: Long-Term Analgesic Efficacy And Safety Of Tanezumab Alone Or In Combination With Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) Versus NSAIDs Alone In Patients With Osteoarthritis Of The Knee Or Hip
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4091025; 2008-004815-37 (EudraCT Number); OA CONTROLLED SAFETY STUDY (Other: Alias Study Number)
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Osteoarthritis; Arthritis
Keywords: monoclonal antibody; nerve growth factor (NGF); anti-NGF; tanezumab; PF-04383119; RN624; osteoarthritis (OA)
MeSH Terms: conditions — Osteoarthritis; Arthritis; Hereditary Sensory and Autonomic Neuropathies | interventions — Anti-Inflammatory Agents, Non-Steroidal; tanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- IV Placebo + NSAID (Active Comparator): Oral NSAID
  Interventions: Drug: NSAID
- Tanezumab 5 mg (Experimental): IV tanezumab 5 mg every 8 weeks (through Week 48)
  Interventions: Biological: tanezumab
- Tanezumab 10 mg (Experimental): IV tanezumab 10 mg every 8 weeks (through Week 48)
  Interventions: Biological: tanezumab
- Tanezumab 5 mg + NSAID (Experimental): IV doses of tanezumab 5 mg every 8 weeks (through Week 48) plus oral naproxen 500 mg BID for 56 weeks or oral celecoxib 100 mg BID for 56 weeks
  Interventions: Biological: tanezumab; Drug: NSAID
- Tanezumab 10 mg + NSAID (Experimental): IV doses of tanezumab 10 mg every 8 weeks (through Week 48) plus oral naproxen 500 mg BID for 56 weeks or oral celecoxib 100 mg BID for 56 weeks
  Interventions: Biological: tanezumab; Drug: NSAID

INTERVENTIONS:
Drug: NSAID — IV doses of placebo (to match tanezumab) every 8 weeks (through Week 48) plus oral naproxen 500 mg BID for 56 weeks or oral celecoxib 100 mg BID for 56 weeks
  Arms: IV Placebo + NSAID
Biological: tanezumab — IV tanezumab 5 mg every 8 weeks (through Week 48) and oral placebo for NSAID BID from Weeks 2 through 56
  Arms: Tanezumab 5 mg
Biological: tanezumab — IV tanezumab 10 mg every 8 weeks (through Week 56) and oral placebo for NSAID BID from Weeks 2 through 56
  Arms: Tanezumab 10 mg
Biological: tanezumab — IV tanezumab 5 mg every 8 weeks (through Week 48)
  Arms: Tanezumab 5 mg + NSAID
Drug: NSAID — Oral naproxen 500 mg BID for 56 weeks or oral celecoxib 100 mg BID for 56 weeks
  Arms: Tanezumab 5 mg + NSAID
Biological: tanezumab — IV tanezumab 10 mg every 8 weeks (through Week 48)
  Arms: Tanezumab 10 mg + NSAID
Drug: NSAID — Oral naproxen 500 mg BID for 56 weeks or oral celecoxib 100 mg BID for 56 weeks
  Arms: Tanezumab 10 mg + NSAID

SUMMARY:
The purpose of this study is to investigate the long-term analgesic efficacy and safety of tanezumab for patients with osteoarthritis (OA) of the knee or hip currently experiencing partial benefit from, and are tolerating, non-steroidal anti-inflammatory drug (NSAID) therapy.

DETAILED DESCRIPTION:
This study was terminated on 28 October 2010 following a US FDA clinical hold for tanezumab osteoarthritis clinical studies which halted dosing and enrollment of patients on 23 June 2010 for potential safety issues.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee or hip according to ACR criteria with Kellgren-Lawrence x-ray grade equal to, or greater than, 2.
* Patients must be experiencing some benefit from their current stable dose regimen of oral NSAID therapy of either naproxen 500-1000 mg/day or celecoxib 200 mg/day (either 100 mg BID or 200 mg QD) and be tolerating their NSAID regimen.
* Pain level and function levels as required by the protocol at Screening and Baseline.
* Willing to discontinue all non-study pain medications for osteoarthritis except rescue medication (acetaminophen) and not use prohibited pain medications throughout the duration of the study except as permitted per protocol.
* Willing and able to comply with lifestyle guidelines, scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

* Pregnant women.
* BMI greater than 39.
* Fibromyalgia, regional pain caused by lumbar or cervical compression with radiculopathy or other moderate to sever pain that may confound assessments or self-evaluation of the pain associated with OA.
* Signs and symptoms of clinically significant cardiac disease with 6 months prior to screening.
* Diagnosis of TIA within 6 months prior to screening or diagnosis of stroke with residual deficits that would preclude completion of required study activities.
* History, diagnosis, signs or symptoms of clinically significant neurological and/or psychiatric disease/disorder.
* At Screening: uncontrolled hypertension, hemoglobin A1c greater than or equal to 10%, ALT or AST greater than or equal to 3X upper limit of normal, creatinine exceeding 1.7 mg/dL (men) or 1.5 mg/dL (women).
* Patients on warfarin or other coumadin anticoagulant therapy and/or lithium therapy within 30 days prior to screening.
* Known hypersensitivity to NSAIDs or cyclooxygenase inhibitors.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2720 (Actual)
Dates: Start 2009-02-12 (Actual); Primary Completion 2010-10-28 (Actual); Study Completion 2011-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (331):
- United States (248):
  - Rheumatology Associates, P.C., Birmingham, Alabama
  - Radiant Research, Birmingham, Alabama
  - Alliance Clinical Research, Birmingham, Alabama
  - Shades Mountain Imaging, Birmingham, Alabama
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Saadat Ansari, MD Office, Huntsville, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Office of Vaughn H. Mancha, Jr., MD, Montgomery, Alabama
  - Radiant Research - Phoenix Southeast, Chandler, Arizona
  - Dedicated Clinical Research, Goodyear, Arizona
  - Eclipse Clinical Research, Green Valley, Arizona
  - Midwest Internal Medicine, PLLC, Lake Havasu City, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C., Mesa, Arizona
  - Pivotal Research Centers, Mesa, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Paradise Valley, Arizona
  - Pivotal Research Centers, Peoria, Arizona
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Associates, P.C., Phoenix, Arizona
  - Cochise Clinical Research, Sierra Vista, Arizona
  - Premiere Phamaceutical Research, LLC, Tempe, Arizona
  - Radiant Research, Tucson, Arizona
  - Arizona Research Associates, Tucson, Arizona
  - Quality of Life Medical and Research Center, Tucson, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Little Rock Diagnostic Clinic, PA, Little Rock, Arkansas
  - Little Rock Family Practice Clinic, Little Rock, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - Orange County Clinical Trials, Inc., Anaheim, California
  - Med Center, Carmichael, California
  - eStudySite, Chula Vista, California
  - Med Investigations, Inc., Fair Oaks, California
  - Triwest Research, La Mesa, California
  - Lakewood Orthopedic Medical & Surgical Group, Lakewood, California
  - Premier Clinical Research LLC., Lakewood, California
  - Prohealth Partners, Long Beach, California
  - Peak Health Medical Group, Inc., Los Angeles, California
  - Synergy Clinical Research Center, National City, California
  - eStudySite, Oceanside, California
  - Desert Medical Group Inc., Desert Oasis Healthcare, Palm Springs, California
  - Advances in Medicine, Rancho Mirage, California
  - Mercy Imaging Center, Sacramento, California
  - Northern Clinical Research, Sacramento, California
  - California Research Foundation, San Diego, California
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - eStudySite, San Jose, California
  - Trinity Clinical Trials, Santa Ana, California
  - Apex Research Institute, Santa Ana, California
  - St. Joseph Medical Associates, Stockton, California
  - Westlake Medical Center, Westlake Village, California
  - Colorado Springs Family Practice, Colorado Springs, Colorado
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Colorado Arthritis Center, PC, Englewood, Colorado
  - Joao MA Nascimento, MD, Bridgeport, Connecticut
  - New England Research Associates, LLC, Trumbull, Connecticut
  - Rheumatology Consultants of Delaware/Delaware Arthritis, Lewes, Delaware
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - International Physicans Research, Aventura, Florida
  - Surgery Center of Aventura, Aventura, Florida
  - HeartCare, Bradenton, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Nature Coast Clinical Research, Crystal River, Florida
  - Homestead Clinical Research Group, P.A., Cutler Bay, Florida
  - Covance CRU, Inc., Daytona Beach, Florida
  - Robert W. Levin MD, Dunedin, Florida
  - Internal Medicine Associates, Fort Myers, Florida
  - Clinical Physiology Associates, Clinical Study Center, Fort Myers, Florida
  - Research Consultants Group, Hialeah, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Florida Arthritis, Lake Mary, Florida
  - Pharmax Research Clinic, Inc., Miami, Florida
  - Community Research Foundation, Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - Jeffrey Alper MD Research, Naples, Florida
  - American Family Medicine, Ocala, Florida
  - Renstar Medical Research, Ocala, Florida
  - Sunshine Research Center, Opa-locka, Florida
  - Arthritis Associates, Orlando, Florida
  - Arthritis Research of Florida, Inc., Palm Harbor, Florida
  - University Clinical Research, Pembroke Pines, Florida
  - Pembroke Clinical Trials, Pemkbroke Pines, Florida
  - Advent Clinical Research Center Inc, Pinellas Park, Florida
  - Advent Clinical Research Centers, Pinellas Park, Florida
  - Berma Research Group, Plantation, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - HeartCare Research, Sarasota, Florida
  - Kennedy-White Orthopaedic Center, Sarasota, Florida
  - Sarasota Center for Clinical Research, Sarasota, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - The Arthritis Specialty Centre, Sarasota, Florida
  - Dale G. Bramlet, MD, P.L., St. Petersburg, Florida
  - Soutwest Florida Clinical Research Center, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Tampa Medical Group, PA, Tampa, Florida
  - Florida Medical Clinic, PA, Zephyrhills, Florida
  - Perimeter Institute for Clinical Reseach, Inc., Atlanta, Georgia
  - Laureate Clinical Research Group, Atlanta, Georgia
  - ACCR/Internal Medicine, Roswell, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Idaho Arthritis & Osteoporosis Center, PC, Meridian, Idaho
  - Saltzer Medical Group PA, Nampa, Idaho
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Rockford Orthopedic Associates, Rockford, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Clinical Research Department, Springfield, Illinois
  - Deerbrook Medical Associates, Vernon Hills, Illinois
  - American Health Network of Indiana, LLC, Avon, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Integrated Clinical Trial Services, Inc, West Des Moines, Iowa
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Center for Arthritis and Osteoporosis, Elizabethtown, Kentucky
  - Pain Treatment Center of the Bluegrass, Lexington, Kentucky
  - Pasadena Pharmacy, Lexington, Kentucky
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - Multicare Specialists, Madisonville, Kentucky
  - Gulf Coast Research, LLC, Baton Rouge, Louisiana
  - The Bone and Joint Clinic, Baton Rouge, Louisiana
  - MD Medical Research, Oxon Hill, Maryland
  - Beacon Clinical Research, Brockton, Massachusetts
  - Berkshire Rheumatology, Pittsfield, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Quest Research Institute, Bingham Farms, Michigan
  - Rheumatology PC, Kalamazoo, Michigan
  - Justus J Fiechtner, MD, Lansing, Michigan
  - PCM Medical Services, Lansing, Michigan
  - Medical Research Associates, Traverse City, Michigan
  - The Center for Clinical Trials, Biloxi, Mississippi
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Highland Community Hospital, Picayune, Mississippi
  - Mississippi Medical Research, Picayune, Mississippi
  - No. County Internal Medicine & Rheumatology, Florissant, Missouri
  - Dynamic Clinical Research, Inc., Kansas City, Missouri
  - Joan Prouty Moore, Kansas City, Missouri
  - Orthopaedic & Occupational Medicine, Kansas City, Missouri
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - Rheumatology and Internal Medicine Associates of West County, P.C., St Louis, Missouri
  - A & A Pain Institute, St Louis, Missouri
  - Arthritis Consultants Inc., St Louis, Missouri
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Westroads Medical Group, Omaha, Nebraska
  - Anderson and Collins Clinical Research Inc., Edison, New Jersey
  - Central Jersey Medical Research Center, Elizabeth, New Jersey
  - Arthritis & Osteoporosis Associates, P.A., Freehold, New Jersey
  - Mark Fisher, MD, FACRUC, Haddon Heights, New Jersey
  - New Jersey Physicians, LLC, Passaic, New Jersey
  - Rheumatology Associates of North Jersey, Teaneck, New Jersey
  - Arthritis & Osteoporosis Associates, Toms River, New Jersey
  - Premier Research, Trenton, New Jersey
  - Arthritis, Rheumatic & Back Disease Associates, Voorhees Township, New Jersey
  - The Center for Rheumatology, LLP, Albany, New York
  - Arthritis and Osteoporosis Associates of Brooklyn Heights, Brooklyn, New York
  - NYU Hospital for Joint Diseases, New York, New York
  - Prem C. Chatpar, MD, LLC, Plainview, New York
  - SPRI Bronx LLC, The Bronx, New York
  - Southgate Medical Group, West Seneca, New York
  - Physicians East P. A., Greenville, North Carolina
  - Physicians East, PA, Greenville, North Carolina
  - Clinical Trials of America, Inc, Hickory, North Carolina
  - Piedmont Rheumatology, Hickory, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Wake Internal Medicine Consultants Inc, Raleigh, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Crescent Medical Research, Salisbury, North Carolina
  - Internal Medicine Associates, Fargo, North Dakota
  - Lillestol Research, LLC, Fargo, North Dakota
  - Daystar Clinical Research, Inc., Akron, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Doctor's Urgent Care Offices, Cincinnati, Ohio
  - Sterling Research Group, Cincinnati, Ohio
  - Columbus Clinical Research, Inc., Columbus, Ohio
  - Optimed Research, LTD, Columbus, Ohio
  - STAT Research, Inc., Dayton, Ohio
  - Dayton Science Institute (DSI), Dayton, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - PHP - Center for Clinical Research, Dayton, Ohio
  - David R. Mandel, MD, Inc, Mayfield, Ohio
  - Southwest Rheumatology and Research Group, LLC, Middleburg Heights, Ohio
  - Integris Family Care of Norman, Norman, Oklahoma
  - LION Research, Norman, Oklahoma
  - Central Sooner Research, Norman, Oklahoma
  - Elise Wiesner, MD, Norman, Oklahoma
  - McBride Clinic, Inc, Norman, Oklahoma
  - McBride Clinic, Norman, Oklahoma
  - McBride Clinic, Inc, Oklahoma City, Oklahoma
  - Bone and Joint Hospital at St. Anthony, Oklahoma City, Oklahoma
  - Christine Codding, MD, Oklahoma City, Oklahoma
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Mc Bride Clinic, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Associated Orthopedics, Inc., Oklahoma City, Oklahoma
  - Hillcrest Clinical Research, Oklahoma City, Oklahoma
  - Rheumatology Associates Inc, Tulsa, Oklahoma
  - Aquilo Clinical Research, Yukon, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - Blair Orthopedics Associates, Altoona, Pennsylvania
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - The Family Healthcare Center, PA, Clinton, South Carolina
  - Columbia Arthritis Center P.A., Columbia, South Carolina
  - Southern Orthopaedic Sports Medicine, Columbia, South Carolina
  - Radiant Research Inc, Greer, South Carolina
  - The Carolina Center for Rheumatology and Arthritis Care, PA, Rock Hill, South Carolina
  - Regional Health Clinical Research, Rapid City, South Dakota
  - Regional Medical Clinical-Rheumatology, Rapid City, South Dakota
  - Arthritis Clinic, Jackson, Tennessee
  - Ramesh C. Gupta, M.D., Memphis, Tennessee
  - Abilene Arthritis Center, Abilene, Texas
  - Tekton Research, Inc., Austin, Texas
  - Dr. Paul K. Pickrell (Physician's Office), Austin, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - One Step Diagnostic, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Miracle Medical Center, Houston, Texas
  - DM Clinical Research, Houston, Texas
  - Gill Orthopedic Center, Lubbock, Texas
  - Robert R. King, M.D., Lubbock, Texas
  - Southwest Rheumatology, PA, Mesquite, Texas
  - Hill Country Medical Associates, New Braunfels, Texas
  - Neurology Clinic of Central Texas, New Braunfels, Texas
  - Philip Blum, Pasadena, Texas
  - Pearland Primary Care Associates, Pearland, Texas
  - Southwest Clinical Research Centers, LLC, Pearland, Texas
  - Plano Primary Care Clinic, Plano, Texas
  - Advanced Family Medical Care, Plano, Texas
  - Alamo Clinical Research Associates, San Antonio, Texas
  - Alamo Clinical Research Consultants, San Antonio, Texas
  - Texas Arthritis Research Center, PA, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Radiant Research San Antonio, San Antonio, Texas
  - SAM Clinical Research Center, San Antonio, Texas
  - San Antonio Preventive & Diagnostic Medicine, PA, San Antonio, Texas
  - South Texas Radiology Imaging Center, San Antonio, Texas
  - The Rehab Group, San Antonio, Texas
  - Sugar Land Med-Ped, PA, Sugar Land, Texas
  - Scott & White Healthcare, Temple, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - Pivotal Research Centers, Midvale, Utah
  - Optimum Clinical Research, Inc., Salt Lake City, Utah
  - Radiant Research, Inc., Salt Lake City, Utah
  - Doris M. Rice, M.D., F.A.C.R., Portsmouth, Virginia
  - National Clinical Research Richmond Inc., Richmond, Virginia
  - Hypothe Test, LLC, Roanoke, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Tacoma Center for Arthritis Research, PS, Tacoma, Washington
  - Gundersen Clinic Ltd., Onalaska, Wisconsin
- Canada (12):
  - Office of Diane Wilson, Lunenburg, Nova Scotia
  - MAC Research Inc., Hamilton, Ontario
  - KW Musculoskeletal Research Inc., Kitchener, Ontario
  - The Arthritis Program Research Group, Newmarket, Ontario
  - SKDS Research Inc., Newmarket, Ontario
  - Dr. Saeed Shaikh, St. Catharines, Ontario
  - Dr. Anil Gupta, Toronto, Ontario
  - Groupe de Recherche en Rhumatologie et Maladies Osseuses, Québec, Quebec
  - Clinique Medicale St-Louis, Québec, Quebec
  - Polyclinique St. Eustache, Saint-Eustache, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec
- Colombia (5):
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Centro Integral de Reumatologia e Inmunologia CIREI, Bogota, Cundinamarca
  - Riesgo de Fractura S.A., Bogota-Cundinamarca
  - Clinica Las Americas, Medellín
  - Reumatologya S.A., Medellín
- India (8):
  - Krishna Institute of Medical Sciences Ltd., Department of Rheumatology, Secunderabad, Andhra Pradesh
  - St. Johns Medical College Hospital, Department of Orthopaedics, Bangalore, Karnataka
  - M.S. Ramaiah Memorial Hospital, Department of Orthopaedics, Bangalore, Karnataka
  - ChanRe Rheumatology & Immunology Center & Research, Bangalore, Karnataka
  - KMC Hospital, Department of Orthopaedics, Mangalore, Karnataka
  - Sancheti Hospital, Pune, Maharashtra
  - PSG Institute of Medical Sciences and Research, Coimbatore, Tamil Nadu
  - CSM Medical University, Department of Rheumatology, Lucknow, Uttar Pradesh
- Mexico (5):
  - URHIA(Unidad de Investigacion en Reumatologia)Hospital Civil de Guadalajara"Fray Antonio Alcalde", Guadalajara, Jalisco
  - Unidad de Enfermedades Reumaticas y Cronico Degenerativas S.C., Coahuila
  - Hospital General de Culiacan, S.S., "Dr. Bernardo Gastelum"., Culiacan Sinaloa
  - Hospital Aranda de la Parra, Leon Gto
  - Beneficencia Espanola de la Laguna, Torreon Coahuila
- Netherlands (3):
  - READE, Amsterdam
  - UMC St. Radboud, Nijmegen
  - UMC Utrecht, Utrecht
- Philippines (8):
  - Cebu Orthopedic Institute, Cebu City
  - Chong Hua Hospital, Medical Arts Center, Cebu City
  - Diaz Building, Cebu City
  - Asian Hospital and Medical Center, City of Muntinlupa
  - Davao Doctors Hospital, Medical Tower, Davao City
  - Davao Doctors Hospital, Davao City
  - Rayuma Clinic, OPD , Jose Reyes Memorial Medical Center, Manila
  - Chinese General Hospital and Medical Center, Out Patient Department, Manila
- Russia (6):
  - State Healthcare Institution Moscow City Clinical Hospital #4, Moscow
  - State Healthcare Institution: Moscow City Clinical Hospital #7, Moscow
  - Institution Of Russian Academy of Medical Sciences, Moscow
  - Federal State Healthcare Institution Clinical Hospital #122 n.a.Sokolov, Saint Petersburg
  - Saint-Petersburg State Healthcare Institution "City Hospital #26", Saint Petersburg
  - Saint Petersburg State Medical University named after Pavlov, Saint Petersburg
- South Africa (14):
  - 136 Panorama Medical Center, Panorama, CAPE TOWN
  - Phelang Private Hospital Research Unit, Mamelodi East, Pretoria
  - Tiervlei Trial Center, Bellville
  - Worthwhile Clinical Trials, Benoni
  - Josha Research, Bloemfontein
  - Vincent Pallotti Hospital, Cape Town
  - Private Practice, Durban
  - Randles Road Medical Center, Durban
  - A. Briel, Durbanville
  - Origin Clinical Research, Johannesburg
  - Clinresco Centres (Pty) Ltd, Kempton Park
  - Paarl Research Center, Paarl
  - TREAD Research, Parrowvalley
  - Clinical Research Unit, Pretoria
- South Korea (5):
  - Kyungpook National University Hospital, Daegu
  - Inha University Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
- Spain (9):
  - Corporacio Sanitaria Parc Tauli de Sabadell, Servicio de Reumatologia, Sabadell, Barcelona
  - Hospital El Tomillar, Dos Hermanas, Sevilla
  - Complejo Hospitalario Universitario de A Coruna, A Coruña
  - Hospital de Cruces, Servicio de Reumatologia, Barakaldo (Vizcaya)
  - Clinica CIMA, Barcelona
  - Servicio de Reumatologia,Institut Ferran de Reumatologia-Clinica CIMA, Barcelona
  - Hospital Universitario La Paz, Servicio de Reumatologia, Madrid
  - Hospital Nuestra Senora de la Esperanza, Servicio de Reumatologia, Santiago de Compostela, A Coruna
  - Hospital Nuestra Senora de Valme, Servicio de Reumatologia, Seville
- Ukraine (8):
  - Chernivtsi Regional Clinical Hospital, Chernivtsi
  - City Clinical Hospital #5, Donetsk
  - V.K. Gusak Institute of Urgent and Recovery Surgery, Donetsk
  - Kiev City Oleksandrivska Clinical Hospital, Kiev
  - Kiev City Clinical Hospital #3, Kiev
  - State Institution "Research Centre for Radiation Medicine AMS of Ukraine", Kiev
  - State Institution "Institute of Gerontology AMS of Ukraine", Kiev
  - Municipal institution :Zaporizhzhya Regional Clinical Hospital, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Tive L, Bello AE, Radin D, Schnitzer TJ, Nguyen H, Brown MT, West CR. Pooled analysis of tanezumab efficacy and safety with subgroup analyses of phase III clinical trials in patients with osteoarthritis pain of the knee or hip. J Pain Res. 2019 Mar 19;12:975-995. doi: 10.2147/JPR.S191297. eCollection 2019. PMID 30936738
- [Derived] Hochberg MC, Tive LA, Abramson SB, Vignon E, Verburg KM, West CR, Smith MD, Hungerford DS. When Is Osteonecrosis Not Osteonecrosis?: Adjudication of Reported Serious Adverse Joint Events in the Tanezumab Clinical Development Program. Arthritis Rheumatol. 2016 Feb;68(2):382-91. doi: 10.1002/art.39492. PMID 26554876
- [Derived] Schnitzer TJ, Ekman EF, Spierings EL, Greenberg HS, Smith MD, Brown MT, West CR, Verburg KM. Efficacy and safety of tanezumab monotherapy or combined with non-steroidal anti-inflammatory drugs in the treatment of knee or hip osteoarthritis pain. Ann Rheum Dis. 2015 Jun;74(6):1202-11. doi: 10.1136/annrheumdis-2013-204905. Epub 2014 Mar 13. PMID 24625625
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091025&StudyName=Long-Term%20Analgesic%20Efficacy%20And%20Safety%20Of%20Tanezumab%20Alone%20Or%20In%20Combination%20With%20Non-Steroidal%20Anti-Inflammatory%20Drugs%20%28NSAIDs%29%20Versus%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Tanezumab 5 mg (Naproxen Exposure): Participants received tanezumab 5 milligram (mg) intravenously (IV) infusion, once every 8 weeks up to Week 48, beginning from Day 1 of Week 1. Additionally, participants received naproxen 500 mg tablet orally twice daily on Days 1-7, naproxen 500 mg tablet orally once daily in the morning of Days 8-14 and placebo matching to naproxen tablet once daily in the evening of Days 8-14. From Day 15, participants received placebo matched to naproxen 500 mg tablet orally twice daily up to Week 48.
- Tanezumab 10 mg (Naproxen Exposure): Participants received tanezumab 10 mg IV infusion, once every 8 weeks up to Week 48, beginning from Day 1 of Week 1. Additionally, participants received naproxen 500 mg tablet orally twice daily on Days 1-7, naproxen 500 mg tablet orally once daily in the morning of Days 8-14 and placebo matching to naproxen tablet once daily in the evening of Days 8-14. From Day 15, participants received placebo matched to naproxen 500 mg tablet orally twice daily up to Week 48.
- Tanezumab 5 mg + Naproxen 500 mg: Participants received tanezumab 5 mg IV infusion, once every 8 weeks up to Week 48, beginning from Day 1 of Week 1 and naproxen 500 mg tablet orally twice daily from Day 1 of Week 1 up to Week 48.
- Tanezumab 10 mg + Naproxen 500 mg: Participants received tanezumab 10 mg IV infusion, once every 8 weeks up to Week 48, beginning from Day 1 of Week 1 and naproxen 500 mg tablet orally twice daily from Day 1 of Week 1 up to Week 48.
- Naproxen 500 mg: Participants received naproxen 500 mg tablet orally twice daily from Day 1 of Week 1 up to Week 48 and placebo matched to tanezumab infusion, IV once every 8 weeks up to Week 48, beginning from Day 1 of Week 1.
- Tanezumab 5 mg (Celecoxib Exposure): Participants received tanezumab 5 mg IV infusion, once every 8 weeks up to Week 48, beginning from Day 1 of Week 1. Additionally, participants received celecoxib 100 mg tablet orally twice daily on Days 1-7, celecoxib 100 mg tablet orally once daily in the morning of Days 8-14 and placebo matched to celecoxib tablet once daily in the evening of Days 8-14. From Day 15, participants received placebo matched to celecoxib 100 mg tablet orally twice daily up to Week 48.
- Tanezumab 10 mg (Celecoxib Exposure): Participants received tanezumab 10 mg IV infusion, once every 8 weeks up to Week 48, beginning from Day 1 of Week 1. Additionally, participants received celecoxib 100 mg tablet orally twice daily on Days 1-7, celecoxib 100 mg tablet orally once daily in the morning of Days 8-14 and placebo matched to celecoxib tablet once daily in the evening of Days 8-14. From Day 15, participants received placebo matched to celecoxib 100 mg tablet orally twice daily up to Week 48.
- Tanezumab 5 mg + Celecoxib 100 mg: Participants received tanezumab 5 mg IV infusion, once every 8 weeks, beginning from Day 1 of Week 1 and celecoxib 100 mg tablet orally twice daily from Day 1 of Week 1 up to Week 48.
- Tanezumab 10 mg + Celecoxib 100 mg: Participants received tanezumab 10 mg IV infusion, once every 8 weeks up to Week 48, beginning from Day 1 of Week 1 and celecoxib 100 mg tablet orally twice daily from Day 1 of Week 1 up to Week 48.
- Celecoxib 100 mg: Placebo matched to tanezumab infusion, IV once every 8 weeks plus celecoxib 100 mg tablet orally twice daily up to Week 48.
Period: Overall Study
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Started | 288 | 289 | 286 | 288 | 288 | 256 | 255 | 257 | 256 | 257
Treated | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
Completed | 33 | 31 | 32 | 32 | 32 | 31 | 32 | 19 | 28 | 31
Not Completed | 255 | 258 | 254 | 256 | 256 | 225 | 223 | 238 | 228 | 226
Not completed — Adverse Event | 32 | 45 | 37 | 53 | 26 | 33 | 44 | 40 | 46 | 26
Not completed — Lack of Efficacy | 23 | 23 | 22 | 15 | 40 | 19 | 21 | 15 | 18 | 38
Not completed — Lost to Follow-up | 10 | 11 | 8 | 13 | 6 | 2 | 0 | 5 | 4 | 0
Not completed — Protocol Violation | 7 | 14 | 14 | 12 | 14 | 6 | 4 | 6 | 9 | 3
Not completed — Withdrawal by Subject | 32 | 27 | 31 | 33 | 34 | 29 | 27 | 19 | 18 | 20
Not completed — Other | 10 | 2 | 7 | 10 | 5 | 3 | 2 | 3 | 4 | 3
Not completed — Study terminated by sponsor | 138 | 134 | 129 | 120 | 126 | 133 | 124 | 148 | 127 | 135
Not completed — Withdrawn due to pregnancy | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but not Treated | 3 | 1 | 6 | 0 | 5 | 0 | 1 | 1 | 2 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) analysis set included all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg | Total
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256 | 2700
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 20 | 16 | 18 | 18 | 14 | 8 | 3 | 11 | 7 | 3 | 118
  45 to 64 years | 168 | 181 | 157 | 171 | 195 | 134 | 117 | 139 | 133 | 144 | 1539
  greater than or equal to (>=) 65 years | 97 | 91 | 105 | 99 | 74 | 114 | 134 | 106 | 114 | 109 | 1043
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 208 | 184 | 192 | 199 | 192 | 184 | 179 | 177 | 189 | 1904
  Male | 85 | 80 | 96 | 96 | 84 | 64 | 70 | 77 | 77 | 67 | 796

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 16
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis of index joint (knee or hip). The WOMAC pain subscale was a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis of index joint (knee or hip) during past 48 hours. It was calculated as mean of the scores from 5 individual questions scored on a numerical rating scale (NRS) of 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Total score range for WOMAC pain subscale score was 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain.
Time Frame: Baseline, Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (tanezumab or matching placebo). Missing values were imputed using baseline observation carried forward (BOCF). Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 287 | 280 | 286 | 282 | 254 | 254 | 256 | 254 | 255
units on a scale
  Baseline | 6.39 (1.61) | 6.50 (1.57) | 6.52 (1.65) | 6.33 (1.65) | 6.32 (1.64) | 6.49 (1.55) | 6.44 (1.53) | 6.41 (1.66) | 6.27 (1.64) | 6.29 (1.60)
  Change at Week 16 | -1.80 (2.20) | -1.97 (2.35) | -2.09 (2.19) | -2.26 (2.31) | -1.34 (2.08) | -2.11 (2.51) | -2.12 (2.36) | -2.28 (2.43) | -2.41 (2.54) | -1.48 (2.07)
Statistical Analysis 1: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; Analysis was based on analysis of co-variance (ANCOVA) model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; Least Square (LS) Mean Difference = -0.92, 95% CI 2-sided [-1.28 to -0.57], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.70, 95% CI 2-sided [-1.06 to -0.33], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.001, ANCOVA; LS Mean Difference = -0.58, 95% CI 2-sided [-0.94 to -0.23], Standard Error of Mean 0.18
Statistical Analysis 4: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.015, ANCOVA; LS Mean Difference = -0.45, 95% CI 2-sided [-0.81 to -0.09], Standard Error of Mean 0.18
Statistical Analysis 5: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.453, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.49 to 0.22], Standard Error of Mean 0.18
Statistical Analysis 6: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.177, ANCOVA; LS Mean Difference = -0.25, 95% CI 2-sided [-0.61 to 0.11], Standard Error of Mean 0.18
Statistical Analysis 7: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.062, ANCOVA; LS Mean Difference = -0.34, 95% CI 2-sided [-0.70 to 0.02], Standard Error of Mean 0.18
Statistical Analysis 8: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.212, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.59 to 0.13], Standard Error of Mean 0.18
Statistical Analysis 9: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.94, 95% CI 2-sided [-1.34 to -0.54], Standard Error of Mean 0.20
Statistical Analysis 10: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.75, 95% CI 2-sided [-1.15 to -0.35], Standard Error of Mean 0.20
Statistical Analysis 11: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.004, ANCOVA; LS Mean Difference = -0.58, 95% CI 2-sided [-0.98 to -0.18], Standard Error of Mean 0.20
Statistical Analysis 12: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.007, ANCOVA; LS Mean Difference = -0.55, 95% CI 2-sided [-0.95 to -0.15], Standard Error of Mean 0.20
Statistical Analysis 13: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.879, ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.43 to 0.37], Standard Error of Mean 0.20
Statistical Analysis 14: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.330, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.60 to 0.20], Standard Error of Mean 0.20
Statistical Analysis 15: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.083, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.75 to 0.05], Standard Error of Mean 0.20
Statistical Analysis 16: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.360, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.59 to 0.21], Standard Error of Mean 0.20

2. Primary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Score at Week 16
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis of index joint (knee or hip).The WOMAC physical function subscale was comprised of 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis of index joint (knee or hip) during past 48 hours. It was calculated as mean of the scores from 17 individual questions scored on a NRS of 0 (minimum difficulty) to 10 (maximum difficulty), where higher scores indicated worse physical function. Total score range for WOMAC physical function subscale score was 0 (minimum difficulty) to 10 (maximum difficulty), where higher scores indicated worse physical function. Physical function refers to participant's ability to move around and perform usual activities of daily living.
Time Frame: Baseline, Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo). Missing values were imputed using BOCF. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 284 | 287 | 280 | 286 | 282 | 255 | 253 | 255 | 253 | 254
units on a scale
  Baseline | 6.46 (1.72) | 6.47 (1.61) | 6.57 (1.67) | 6.39 (1.62) | 6.32 (1.62) | 6.67 (1.60) | 6.58 (1.58) | 6.57 (1.72) | 6.39 (1.62) | 6.47 (1.59)
  Change at Week 16 | -1.80 (2.15) | -1.84 (2.13) | -2.12 (2.19) | -2.18 (2.31) | -1.28 (1.96) | -2.13 (2.34) | -2.09 (2.34) | -2.27 (2.40) | -2.41 (2.43) | -1.42 (2.03)
Statistical Analysis 1: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.88, 95% CI 2-sided [-1.23 to -0.53], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.78, 95% CI 2-sided [-1.13 to -0.43], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-0.87 to -0.17], Standard Error of Mean 0.18
Statistical Analysis 4: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.007, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-0.83 to -0.13], Standard Error of Mean 0.18
Statistical Analysis 5: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.824, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.39 to 0.31], Standard Error of Mean 0.18
Statistical Analysis 6: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.100, ANCOVA; LS Mean Difference = -0.29, 95% CI 2-sided [-0.64 to 0.06], Standard Error of Mean 0.18
Statistical Analysis 7: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.044, ANCOVA; LS Mean Difference = -0.36, 95% CI 2-sided [-0.70 to -0.01], Standard Error of Mean 0.18
Statistical Analysis 8: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.565, ANCOVA; LS Mean Difference = -0.10, 95% CI 2-sided [-0.45 to 0.25], Standard Error of Mean 0.18
Statistical Analysis 9: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.01, 95% CI 2-sided [-1.40 to -0.62], Standard Error of Mean 0.20
Statistical Analysis 10: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.81, 95% CI 2-sided [-1.20 to -0.42], Standard Error of Mean 0.20
Statistical Analysis 11: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.63, 95% CI 2-sided [-1.02 to -0.24], Standard Error of Mean 0.20
Statistical Analysis 12: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.63, 95% CI 2-sided [-1.02 to -0.24], Standard Error of Mean 0.20
Statistical Analysis 13: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.980, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.39 to 0.40], Standard Error of Mean 0.20
Statistical Analysis 14: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.383, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.56 to 0.22], Standard Error of Mean 0.20
Statistical Analysis 15: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.057, ANCOVA; LS Mean Difference = -0.38, 95% CI 2-sided [-0.77 to 0.01], Standard Error of Mean 0.20
Statistical Analysis 16: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.312, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.59 to 0.19], Standard Error of Mean 0.20

3. Primary Outcome: Change From Baseline in the Patient Global Assessment (PGA) of Osteoarthritis at Week 16
Description: Patient global assessment of osteoarthritis was assessed by asking a question from participants: "Considering all the ways your osteoarthritis in your knee or hip affects you, how are you doing today?" Participants responded by using a 5-point likert scale ranging from 1=very good (asymptomatic and no limitation of normal activities, 2= good (mild symptoms and no limitation of normal activities), 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5= very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Higher scores indicating worse condition.
Time Frame: Baseline, Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo). Missing values were imputed using baseline BOCF. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 284 | 288 | 280 | 285 | 283 | 256 | 254 | 255 | 253 | 254
units on a scale
  Baseline | 3.39 (0.63) | 3.41 (0.62) | 3.39 (0.63) | 3.39 (0.66) | 3.38 (0.63) | 3.44 (0.65) | 3.48 (0.63) | 3.45 (0.67) | 3.41 (0.64) | 3.37 (0.59)
  Change at Week 16 | -0.54 (0.90) | -0.63 (0.91) | -0.61 (0.89) | -0.72 (1.01) | -0.53 (0.75) | -0.69 (0.86) | -0.64 (0.86) | -0.76 (0.95) | -0.75 (0.90) | -0.51 (0.86)
Statistical Analysis 1: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.008, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.32 to -0.05], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.251, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.22 to 0.06], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.251, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.22 to 0.06], Standard Error of Mean 0.07
Statistical Analysis 4: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.961, ANCOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-0.14 to 0.13], Standard Error of Mean 0.07
Statistical Analysis 5: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.272, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.21 to 0.06], Standard Error of Mean 0.07
Statistical Analysis 6: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.271, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.21 to 0.06], Standard Error of Mean 0.07
Statistical Analysis 7: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.128, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.24 to 0.03], Standard Error of Mean 0.07
Statistical Analysis 8: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.133, ANCOVA; LS Mean Difference = -0.10, 95% CI 2-sided [-0.24 to 0.03], Standard Error of Mean 0.07
Statistical Analysis 9: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.35 to -0.08], Standard Error of Mean 0.07
Statistical Analysis 10: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.004, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.34 to -0.06], Standard Error of Mean 0.07
Statistical Analysis 11: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.414, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.20 to 0.08], Standard Error of Mean 0.07
Statistical Analysis 12: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.057, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.27 to 0.00], Standard Error of Mean 0.07
Statistical Analysis 13: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.277, ANCOVA; LS Mean Difference = 0.08, 95% CI 2-sided [-0.06 to 0.21], Standard Error of Mean 0.07
Statistical Analysis 14: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.328, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.21 to 0.07], Standard Error of Mean 0.07
Statistical Analysis 15: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.026, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.30 to -0.02], Standard Error of Mean 0.07
Statistical Analysis 16: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.864, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.15 to 0.13], Standard Error of Mean 0.07

4. Secondary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Weeks 2, 4, 8, 12 and 24: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis of index joint (knee or hip). The WOMAC pain subscale was a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis of index joint (knee or hip) during past 48 hours. It was calculated as mean of the scores from 5 individual questions scored on a NRS of 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Total score range for WOMAC pain subscale score was 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 287 | 280 | 286 | 282 | 254 | 254 | 256 | 254 | 255
units on a scale
  Change at Week 2 | -0.96 (1.98) | -1.00 (2.08) | -1.27 (2.03) | -0.89 (2.21) | -0.90 (1.81) | -1.01 (2.15) | -0.74 (2.08) | -1.08 (2.03) | -0.86 (2.22) | -0.93 (1.66)
  Change at Week 4 | -1.68 (2.05) | -1.87 (1.96) | -2.09 (2.13) | -1.98 (2.22) | -1.14 (2.09) | -1.69 (2.39) | -1.78 (2.06) | -2.07 (2.27) | -2.03 (2.27) | -1.09 (1.94)
  Change at Week 8 | -1.68 (2.27) | -2.08 (2.14) | -2.10 (2.25) | -2.18 (2.26) | -1.13 (2.08) | -1.83 (2.35) | -2.01 (2.26) | -2.23 (2.22) | -2.36 (2.34) | -1.15 (2.03)
  Change at Week 12 | -1.86 (2.32) | -1.95 (2.21) | -2.26 (2.21) | -2.34 (2.35) | -1.23 (2.12) | -2.15 (2.44) | -2.20 (2.54) | -2.28 (2.39) | -2.47 (2.40) | -1.40 (1.96)
  Change at Week 24 | -1.65 (2.33) | -1.82 (2.32) | -1.83 (2.19) | -1.95 (2.38) | -1.32 (2.15) | -1.81 (2.46) | -2.04 (2.33) | -2.10 (2.47) | -2.29 (2.56) | -1.63 (2.07)
Statistical Analysis 1: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; Change at Week 2: Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.927, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.31 to 0.34], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.057, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-0.64 to 0.01], Standard Error of Mean 0.17
Statistical Analysis 3: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.779, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.37 to 0.28], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.798, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.36 to 0.28], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.980, ANCOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-0.33 to 0.32], Standard Error of Mean 0.16
Statistical Analysis 6: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.098, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.60 to 0.05], Standard Error of Mean 0.16
Statistical Analysis 7: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.709, ANCOVA; LS Mean Difference = 0.06, 95% CI 2-sided [-0.26 to 0.38], Standard Error of Mean 0.16
Statistical Analysis 8: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.045, ANCOVA; LS Mean Difference = 0.33, 95% CI 2-sided [0.01 to 0.65], Standard Error of Mean 0.16
Statistical Analysis 9: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.710, ANCOVA; LS Mean Difference = 0.06, 95% CI 2-sided [-0.28 to 0.41], Standard Error of Mean 0.17
Statistical Analysis 10: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.504, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.46 to 0.23], Standard Error of Mean 0.17
Statistical Analysis 11: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.183, ANCOVA; LS Mean Difference = 0.23, 95% CI 2-sided [-0.11 to 0.58], Standard Error of Mean 0.17
Statistical Analysis 12: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.919, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.36 to 0.33], Standard Error of Mean 0.17
Statistical Analysis 13: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.152, ANCOVA; LS Mean Difference = 0.25, 95% CI 2-sided [-0.09 to 0.59], Standard Error of Mean 0.17
Statistical Analysis 14: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.572, ANCOVA; LS Mean Difference = -0.10, 95% CI 2-sided [-0.44 to 0.24], Standard Error of Mean 0.17
Statistical Analysis 15: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.337, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.51 to 0.18], Standard Error of Mean 0.17
Statistical Analysis 16: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.299, ANCOVA; LS Mean Difference = 0.18, 95% CI 2-sided [-0.16 to 0.52], Standard Error of Mean 0.17
Statistical Analysis 17: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; Change at Week 4: Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.84, 95% CI 2-sided [-1.17 to -0.50], Standard Error of Mean 0.17
Statistical Analysis 18: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.89, 95% CI 2-sided [-1.22 to -0.55], Standard Error of Mean 0.17
Statistical Analysis 19: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.68, 95% CI 2-sided [-1.01 to -0.34], Standard Error of Mean 0.17
Statistical Analysis 20: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-0.85 to -0.18], Standard Error of Mean 0.17
Statistical Analysis 21: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.341, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.50 to 0.17], Standard Error of Mean 0.17
Statistical Analysis 22: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.031, ANCOVA; LS Mean Difference = -0.37, 95% CI 2-sided [-0.71 to -0.03], Standard Error of Mean 0.17
Statistical Analysis 23: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.349, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.49 to 0.17], Standard Error of Mean 0.17
Statistical Analysis 24: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.780, ANCOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.29 to 0.38], Standard Error of Mean 0.17
Statistical Analysis 25: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.95, 95% CI 2-sided [-1.31 to -0.58], Standard Error of Mean 0.19
Statistical Analysis 26: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.93, 95% CI 2-sided [-1.29 to -0.56], Standard Error of Mean 0.18
Statistical Analysis 27: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.63, 95% CI 2-sided [-0.99 to -0.26], Standard Error of Mean 0.19
Statistical Analysis 28: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.005, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-0.88 to -0.15], Standard Error of Mean 0.19
Statistical Analysis 29: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.562, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.47 to 0.26], Standard Error of Mean 0.19
Statistical Analysis 30: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.028, ANCOVA; LS Mean Difference = -0.41, 95% CI 2-sided [-0.77 to -0.04], Standard Error of Mean 0.19
Statistical Analysis 31: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.084, ANCOVA; LS Mean Difference = -0.32, 95% CI 2-sided [-0.68 to 0.04], Standard Error of Mean 0.19
Statistical Analysis 32: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.910, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.38 to 0.34], Standard Error of Mean 0.19
Statistical Analysis 33: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; Change at Week 8: Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.05, 95% CI 2-sided [-1.40 to -0.69], Standard Error of Mean 0.18
Statistical Analysis 34: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.91, 95% CI 2-sided [-1.27 to -0.56], Standard Error of Mean 0.18
Statistical Analysis 35: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.90, 95% CI 2-sided [-1.25 to -0.55], Standard Error of Mean 0.18
Statistical Analysis 36: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = -0.53, 95% CI 2-sided [-0.88 to -0.17], Standard Error of Mean 0.18
Statistical Analysis 37: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.039, ANCOVA; LS Mean Difference = -0.37, 95% CI 2-sided [-0.72 to -0.02], Standard Error of Mean 0.18
Statistical Analysis 38: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.032, ANCOVA; LS Mean Difference = -0.39, 95% CI 2-sided [-0.74 to -0.03], Standard Error of Mean 0.18
Statistical Analysis 39: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.409, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.50 to 0.20], Standard Error of Mean 0.18
Statistical Analysis 40: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.461, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.49 to 0.22], Standard Error of Mean 0.18
Statistical Analysis 41: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.21, 95% CI 2-sided [-1.59 to -0.84], Standard Error of Mean 0.19
Statistical Analysis 42: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.03, 95% CI 2-sided [-1.40 to -0.65], Standard Error of Mean 0.19
Statistical Analysis 43: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.80, 95% CI 2-sided [-1.17 to -0.43], Standard Error of Mean 0.19
Statistical Analysis 44: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.59, 95% CI 2-sided [-0.97 to -0.22], Standard Error of Mean 0.19
Statistical Analysis 45: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.281, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.58 to 0.17], Standard Error of Mean 0.19
Statistical Analysis 46: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.023, ANCOVA; LS Mean Difference = -0.43, 95% CI 2-sided [-0.81 to -0.06], Standard Error of Mean 0.19
Statistical Analysis 47: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.031, ANCOVA; LS Mean Difference = -0.41, 95% CI 2-sided [-0.79 to -0.04], Standard Error of Mean 0.19
Statistical Analysis 48: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.331, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.56 to 0.19], Standard Error of Mean 0.19
Statistical Analysis 49: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; Change at Week 12: Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.11, 95% CI 2-sided [-1.47 to -0.75], Standard Error of Mean 0.18
Statistical Analysis 50: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.97, 95% CI 2-sided [-1.33 to -0.60], Standard Error of Mean 0.18
Statistical Analysis 51: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.67, 95% CI 2-sided [-1.03 to -0.31], Standard Error of Mean 0.18
Statistical Analysis 52: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.62, 95% CI 2-sided [-0.98 to -0.26], Standard Error of Mean 0.18
Statistical Analysis 53: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.781, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.41 to 0.31], Standard Error of Mean 0.18
Statistical Analysis 54: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.057, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.71 to 0.01], Standard Error of Mean 0.18
Statistical Analysis 55: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.016, ANCOVA; LS Mean Difference = -0.44, 95% CI 2-sided [-0.80 to -0.08], Standard Error of Mean 0.18
Statistical Analysis 56: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.450, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.50 to 0.22], Standard Error of Mean 0.18
Statistical Analysis 57: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.08, 95% CI 2-sided [-1.47 to -0.69], Standard Error of Mean 0.20
Statistical Analysis 58: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.81, 95% CI 2-sided [-1.20 to -0.42], Standard Error of Mean 0.20
Statistical Analysis 59: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.73, 95% CI 2-sided [-1.12 to -0.34], Standard Error of Mean 0.20
Statistical Analysis 60: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.001, ANCOVA; LS Mean Difference = -0.65, 95% CI 2-sided [-1.04 to -0.26], Standard Error of Mean 0.20
Statistical Analysis 61: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.699, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.47 to 0.31], Standard Error of Mean 0.20
Statistical Analysis 62: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.408, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.55 to 0.22], Standard Error of Mean 0.20
Statistical Analysis 63: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.077, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.74 to 0.04], Standard Error of Mean 0.20
Statistical Analysis 64: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.182, ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-0.65 to 0.12], Standard Error of Mean 0.20

5. Secondary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56: Last Observation Carried Forward (LOCF)
Description: as for outcome 4
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, and 56
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo). Missing values were imputed using LOCF. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 287 | 280 | 286 | 282 | 254 | 254 | 256 | 254 | 255
units on a scale
  Change at Week 2 | -0.96 (1.98) | -1.00 (2.08) | -1.27 (2.03) | -0.89 (2.21) | -0.90 (1.81) | -1.01 (2.15) | -0.74 (2.08) | -1.08 (2.03) | -0.86 (2.22) | -0.93 (1.66)
  Change at Week 4 | -1.66 (2.09) | -1.92 (1.96) | -2.12 (2.13) | -2.05 (2.24) | -1.15 (2.12) | -1.76 (2.45) | -1.73 (2.13) | -2.04 (2.35) | -2.00 (2.31) | -1.10 (1.94)
  Change at Week 8 | -1.76 (2.34) | -2.20 (2.17) | -2.26 (2.25) | -2.36 (2.25) | -1.17 (2.16) | -1.92 (2.45) | -2.07 (2.32) | -2.22 (2.34) | -2.34 (2.42) | -1.17 (2.06)
  Change at Week 12 | -2.04 (2.40) | -2.14 (2.24) | -2.45 (2.18) | -2.56 (2.35) | -1.32 (2.26) | -2.29 (2.53) | -2.32 (2.63) | -2.32 (2.50) | -2.51 (2.47) | -1.40 (2.05)
  Change at Week 16 | -2.00 (2.29) | -2.19 (2.37) | -2.36 (2.20) | -2.56 (2.27) | -1.44 (2.22) | -2.27 (2.59) | -2.23 (2.46) | -2.34 (2.54) | -2.46 (2.59) | -1.50 (2.17)
  Change at Week 24 | -2.04 (2.44) | -2.12 (2.37) | -2.20 (2.26) | -2.33 (2.39) | -1.54 (2.38) | -2.05 (2.56) | -2.25 (2.44) | -2.21 (2.59) | -2.39 (2.64) | -1.69 (2.23)
  Change at Week 32 | -1.94 (2.51) | -2.08 (2.40) | -2.10 (2.32) | -2.33 (2.42) | -1.62 (2.38) | -2.02 (2.57) | -2.14 (2.58) | -2.20 (2.61) | -2.14 (2.67) | -1.62 (2.24)
  Change at Week 40 | -1.90 (2.54) | -1.94 (2.50) | -1.88 (2.38) | -2.12 (2.39) | -1.44 (2.38) | -1.98 (2.49) | -1.99 (2.52) | -1.98 (2.62) | -2.18 (2.60) | -1.54 (2.22)
  Change at Week 48 | -1.86 (2.54) | -1.93 (2.51) | -1.86 (2.44) | -2.08 (2.34) | -1.40 (2.38) | -1.86 (2.47) | -1.93 (2.51) | -2.05 (2.58) | -2.03 (2.63) | -1.45 (2.25)
  Change at Week 56 | -1.84 (2.54) | -1.86 (2.49) | -1.84 (2.44) | -2.03 (2.32) | -1.36 (2.34) | -1.83 (2.38) | -1.72 (2.47) | -1.92 (2.55) | -2.02 (2.61) | -1.48 (2.27)
Statistical Analysis 1: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.798, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.36 to 0.28], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.779, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.37 to 0.28], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.057, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-0.64 to 0.01], Standard Error of Mean 0.17
Statistical Analysis 4: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.927, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.31 to 0.34], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.980, ANCOVA; LS Mean Difference = -0.00, 95% CI 2-sided [-0.33 to 0.32], Standard Error of Mean 0.16
Statistical Analysis 6: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.098, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.60 to 0.05], Standard Error of Mean 0.16
Statistical Analysis 7: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.709, ANCOVA; LS Mean Difference = 0.06, 95% CI 2-sided [-0.26 to 0.38], Standard Error of Mean 0.16
Statistical Analysis 8: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.045, ANCOVA; LS Mean Difference = 0.33, 95% CI 2-sided [0.01 to 0.65], Standard Error of Mean 0.16
Statistical Analysis 9: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.919, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.36 to 0.33], Standard Error of Mean 0.17
Statistical Analysis 10: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.183, ANCOVA; LS Mean Difference = 0.23, 95% CI 2-sided [-0.11 to 0.58], Standard Error of Mean 0.17
Statistical Analysis 11: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.504, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.46 to 0.23], Standard Error of Mean 0.17
Statistical Analysis 12: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.710, ANCOVA; LS Mean Difference = 0.06, 95% CI 2-sided [-0.28 to 0.41], Standard Error of Mean 0.17
Statistical Analysis 13: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.152, ANCOVA; LS Mean Difference = 0.25, 95% CI 2-sided [-0.09 to 0.59], Standard Error of Mean 0.17
Statistical Analysis 14: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.572, ANCOVA; LS Mean Difference = -0.10, 95% CI 2-sided [-0.44 to 0.24], Standard Error of Mean 0.17
Statistical Analysis 15: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.337, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.51 to 0.18], Standard Error of Mean 0.17
Statistical Analysis 16: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.299, ANCOVA; LS Mean Difference = 0.18, 95% CI 2-sided [-0.16 to 0.52], Standard Error of Mean 0.17
Statistical Analysis 17: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.005, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-0.82 to -0.14], Standard Error of Mean 0.17
Statistical Analysis 18: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.71, 95% CI 2-sided [-1.05 to -0.38], Standard Error of Mean 0.17
Statistical Analysis 19: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.91, 95% CI 2-sided [-1.25 to -0.57], Standard Error of Mean 0.17
Statistical Analysis 20: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.90, 95% CI 2-sided [-1.23 to -0.56], Standard Error of Mean 0.17
Statistical Analysis 21: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.177, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.57 to 0.10], Standard Error of Mean 0.17
Statistical Analysis 22: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.014, ANCOVA; LS Mean Difference = -0.42, 95% CI 2-sided [-0.76 to -0.09], Standard Error of Mean 0.17
Statistical Analysis 23: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.286, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.52 to 0.15], Standard Error of Mean 0.17
Statistical Analysis 24: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.952, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.33 to 0.35], Standard Error of Mean 0.17
Statistical Analysis 25: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.58, 95% CI 2-sided [-0.95 to -0.21], Standard Error of Mean 0.19
Statistical Analysis 26: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = -0.57, 95% CI 2-sided [-0.94 to -0.20], Standard Error of Mean 0.19
Statistical Analysis 27: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.89, 95% CI 2-sided [-1.26 to -0.52], Standard Error of Mean 0.19
Statistical Analysis 28: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.92, 95% CI 2-sided [-1.29 to -0.55], Standard Error of Mean 0.19
Statistical Analysis 29: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.972, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.36 to 0.38], Standard Error of Mean 0.19
Statistical Analysis 30: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.096, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-0.69 to 0.06], Standard Error of Mean 0.19
Statistical Analysis 31: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.069, ANCOVA; LS Mean Difference = -0.34, 95% CI 2-sided [-0.72 to 0.03], Standard Error of Mean 0.19
Statistical Analysis 32: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.902, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.39 to 0.35], Standard Error of Mean 0.19
Statistical Analysis 33: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.57, 95% CI 2-sided [-0.93 to -0.22], Standard Error of Mean 0.18
Statistical Analysis 34: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.97, 95% CI 2-sided [-1.33 to -0.61], Standard Error of Mean 0.18
Statistical Analysis 35: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.02, 95% CI 2-sided [-1.38 to -0.66], Standard Error of Mean 0.18
Statistical Analysis 36: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.19, 95% CI 2-sided [-1.55 to -0.84], Standard Error of Mean 0.18
Statistical Analysis 37: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.028, ANCOVA; LS Mean Difference = -0.40, 95% CI 2-sided [-0.75 to -0.04], Standard Error of Mean 0.18
Statistical Analysis 38: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.013, ANCOVA; LS Mean Difference = -0.45, 95% CI 2-sided [-0.81 to -0.09], Standard Error of Mean 0.18
Statistical Analysis 39: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.217, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.58 to 0.13], Standard Error of Mean 0.18
Statistical Analysis 40: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.351, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.53 to 0.19], Standard Error of Mean 0.18
Statistical Analysis 41: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.66, 95% CI 2-sided [-1.05 to -0.28], Standard Error of Mean 0.20
Statistical Analysis 42: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.83, 95% CI 2-sided [-1.22 to -0.45], Standard Error of Mean 0.20
Statistical Analysis 43: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.00, 95% CI 2-sided [-1.38 to -0.62], Standard Error of Mean 0.20
Statistical Analysis 44: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.19, 95% CI 2-sided [-1.57 to -0.80], Standard Error of Mean 0.20
Statistical Analysis 45: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.389, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.55 to 0.22], Standard Error of Mean 0.20
Statistical Analysis 46: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.087, ANCOVA; LS Mean Difference = -0.34, 95% CI 2-sided [-0.72 to 0.05], Standard Error of Mean 0.20
Statistical Analysis 47: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.072, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.74 to 0.03], Standard Error of Mean 0.20
Statistical Analysis 48: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.340, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.57 to 0.20], Standard Error of Mean 0.20
Statistical Analysis 49: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.69, 95% CI 2-sided [-1.06 to -0.33], Standard Error of Mean 0.19
Statistical Analysis 50: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.75, 95% CI 2-sided [-1.11 to -0.39], Standard Error of Mean 0.19
Statistical Analysis 51: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.05, 95% CI 2-sided [-1.42 to -0.69], Standard Error of Mean 0.19
Statistical Analysis 52: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.23, 95% CI 2-sided [-1.59 to -0.87], Standard Error of Mean 0.19
Statistical Analysis 53: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.762, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.42 to 0.31], Standard Error of Mean 0.18
Statistical Analysis 54: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.056, ANCOVA; LS Mean Difference = -0.36, 95% CI 2-sided [-0.72 to 0.01], Standard Error of Mean 0.19
Statistical Analysis 55: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.010, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-0.84 to -0.12], Standard Error of Mean 0.18
Statistical Analysis 56: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.335, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.54 to 0.19], Standard Error of Mean 0.19
Statistical Analysis 57: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.78, 95% CI 2-sided [-1.18 to -0.38], Standard Error of Mean 0.20
Statistical Analysis 58: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.84, 95% CI 2-sided [-1.24 to -0.44], Standard Error of Mean 0.20
Statistical Analysis 59: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.85, 95% CI 2-sided [-1.25 to -0.46], Standard Error of Mean 0.20
Statistical Analysis 60: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.13, 95% CI 2-sided [-1.52 to -0.73], Standard Error of Mean 0.20
Statistical Analysis 61: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.782, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.46 to 0.34], Standard Error of Mean 0.20
Statistical Analysis 62: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.719, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.47 to 0.33], Standard Error of Mean 0.20
Statistical Analysis 63: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.158, ANCOVA; LS Mean Difference = -0.29, 95% CI 2-sided [-0.69 to 0.11], Standard Error of Mean 0.20
Statistical Analysis 64: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.183, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.67 to 0.13], Standard Error of Mean 0.20
Statistical Analysis 65: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; Change at Week 16: Analysis was based on ANCOVA model with treatment, baseline value, index joint (knee or hip) as covariates; Test type: Superiority or Other; p = 0.004, ANCOVA; LS Mean difference = -0.54, 95% CI 2-sided [-0.90 to -0.18], Standard Error of Mean 0.18
Statistical Analysis 66: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean difference = -0.69, 95% CI 2-sided [-1.05 to -0.33], Standard Error of Mean 0.18
Statistical Analysis 67: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean difference = -0.84, 95% CI 2-sided [-1.20 to 0.48], Standard Error of Mean 0.18
Statistical Analysis 68: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean difference = -1.12, 95% CI 2-sided [-1.48 to -0.76], Standard Error of Mean 0.18
Statistical Analysis 69: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p = 0.408, ANCOVA; LS mean difference = -0.15, 95% CI 2-sided [-0.51 to 0.21], Standard Error of Mean 0.18
Statistical Analysis 70: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p = 0.097, ANCOVA; LS mean difference = -0.31, 95% CI 2-sided [-0.67 to 0.06], Standard Error of Mean 0.18
Statistical Analysis 71: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p = 0.018, ANCOVA; LS mean difference = -0.43, 95% CI 2-sided [-0.79 to -0.07], Standard Error of Mean 0.18
Statistical Analysis 72: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p = 0.132, ANCOVA; LS mean difference = -0.28, 95% CI 2-sided [-0.64 to 0.08], Standard Error of Mean 0.18
Statistical Analysis 73: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p = 0.001, ANCOVA; LS Mean Difference = -0.67, 95% CI 2-sided [-1.08 to -0.26], Standard Error of Mean 0.21
Statistical Analysis 74: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.66, 95% CI 2-sided [-1.07 to -0.25], Standard Error of Mean 0.21
Statistical Analysis 75: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.78, 95% CI 2-sided [-1.19 to -0.37], Standard Error of Mean 0.21
Statistical Analysis 76: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.96, 95% CI 2-sided [-1.37 to -0.55], Standard Error of Mean 0.21
Statistical Analysis 77: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p = 0.959, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.40 to 0.42], Standard Error of Mean 0.21
Statistical Analysis 78: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p = 0.618, ANCOVA; LS Mean Difference = -0.10, 95% CI 2-sided [-0.51 to 0.31], Standard Error of Mean 0.21
Statistical Analysis 79: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p = 0.149, ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-0.71 to 0.11], Standard Error of Mean 0.21
Statistical Analysis 80: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p = 0.370, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.60 to 0.22], Standard Error of Mean 0.21

6. Secondary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Score at Weeks 2, 4, 8, 12 and 24: Baseline Observation Carried Forward (BOCF)
Description: as for outcome 2
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 287 | 280 | 286 | 282 | 255 | 253 | 255 | 253 | 254
units on a scale
  Change at Week 2 | -1.10 (1.88) | -1.13 (1.90) | -1.44 (2.02) | -1.06 (2.07) | -0.90 (1.69) | -1.18 (2.01) | -0.95 (1.99) | -1.21 (1.96) | -1.02 (2.13) | -0.90 (1.67)
  Change at Week 4 | -1.71 (2.00) | -1.79 (1.88) | -2.04 (2.16) | -2.00 (2.06) | -1.01 (1.90) | -1.73 (2.23) | -1.78 (2.06) | -1.97 (2.19) | -2.00 (2.13) | -1.07 (1.83)
  Change at Week 8 | -1.62 (2.19) | -2.01 (2.04) | -2.05 (2.26) | -2.15 (2.19) | -1.07 (1.87) | -1.89 (2.27) | -2.00 (2.17) | -2.15 (2.19) | -2.30 (2.22) | -1.13 (1.94)
  Change at Week 12 | -1.85 (2.25) | -1.87 (2.06) | -2.18 (2.17) | -2.29 (2.33) | -1.23 (2.00) | -2.23 (2.34) | -2.13 (2.43) | -2.34 (2.36) | -2.46 (2.32) | -1.36 (1.97)
  Change at Week 24 | -1.66 (2.28) | -1.76 (2.16) | -1.76 (2.11) | -1.96 (2.37) | -1.30 (2.03) | -1.92 (2.29) | -2.00 (2.31) | -2.08 (2.37) | -2.33 (2.45) | -1.57 (2.08)
Statistical Analysis 1: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.887, ANCOVA; LS mean difference = -0.02, 95% CI 2-sided [-0.33 to 0.28], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.046, ANCOVA; LS mean difference = -0.31, 95% CI 2-sided [-0.62 to -0.01], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.771, ANCOVA; LS mean difference = 0.05, 95% CI 2-sided [-0.26 to 0.35], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.032, ANCOVA; LS mean difference = 0.34, 95% CI 2-sided [0.03 to 0.64], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.223, ANCOVA; LS mean difference = 0.21, 95% CI 2-sided [-0.13 to 0.54], Standard Error of Mean 0.17
Statistical Analysis 6: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.718, ANCOVA; LS mean difference = -0.06, 95% CI 2-sided [-0.39 to 0.27], Standard Error of Mean 0.17
Statistical Analysis 7: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.495, ANCOVA; LS mean difference = -0.12, 95% CI 2-sided [-0.45 to 0.22], Standard Error of Mean 0.17
Statistical Analysis 8: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.371, ANCOVA; LS mean difference = 0.15, 95% CI 2-sided [-0.18 to 0.49], Standard Error of Mean 0.17
Statistical Analysis 9: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.647, ANCOVA; LS mean difference = -0.08, 95% CI 2-sided [-0.40 to 0.25], Standard Error of Mean 0.16
Statistical Analysis 10: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.073, ANCOVA; LS mean difference = -0.30, 95% CI 2-sided [-0.62 to 0.03], Standard Error of Mean 0.16
Statistical Analysis 11: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.161, ANCOVA; LS mean difference = -0.23, 95% CI 2-sided [-0.55 to 0.09], Standard Error of Mean 0.16
Statistical Analysis 12: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.961, ANCOVA; LS mean difference = -0.01, 95% CI 2-sided [-0.33 to 0.32], Standard Error of Mean 0.16
Statistical Analysis 13: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.697, ANCOVA; LS mean difference = -0.07, 95% CI 2-sided [-0.42 to 0.28], Standard Error of Mean 0.18
Statistical Analysis 14: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.139, ANCOVA; LS mean difference = -0.27, 95% CI 2-sided [-0.62 to 0.09], Standard Error of Mean 0.18
Statistical Analysis 15: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.120, ANCOVA; LS mean difference = -0.28, 95% CI 2-sided [-0.64 to 0.07], Standard Error of Mean 0.18
Statistical Analysis 16: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.637, ANCOVA; LS mean difference = -0.09, 95% CI 2-sided [-0.44 to 0.27], Standard Error of Mean 0.18
Statistical Analysis 17: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.028, ANCOVA; LS mean difference = -0.38, 95% CI 2-sided [-0.72 to -0.04], Standard Error of Mean 0.17
Statistical Analysis 18: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.024, ANCOVA; LS mean difference = -0.39, 95% CI 2-sided [-0.74 to -0.05], Standard Error of Mean 0.17
Statistical Analysis 19: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.339, ANCOVA; LS mean difference = -0.17, 95% CI 2-sided [-0.51 to 0.17], Standard Error of Mean 0.17
Statistical Analysis 20: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.381, ANCOVA; LS mean difference = -0.15, 95% CI 2-sided [-0.50 to 0.19], Standard Error of Mean 0.17
Statistical Analysis 21: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.438, ANCOVA; LS mean difference = -0.14, 95% CI 2-sided [-0.51 to 0.22], Standard Error of Mean 0.19
Statistical Analysis 22: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.111, ANCOVA; LS mean difference = -0.30, 95% CI 2-sided [-0.66 to 0.07], Standard Error of Mean 0.19
Statistical Analysis 23: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.059, ANCOVA; LS mean difference = -0.35, 95% CI 2-sided [-0.72 to 0.01], Standard Error of Mean 0.19
Statistical Analysis 24: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.282, ANCOVA; LS mean difference = -0.20, 95% CI 2-sided [-0.57 to 0.17], Standard Error of Mean 0.19
Statistical Analysis 25: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.927, ANCOVA; LS mean difference = -0.02, 95% CI 2-sided [-0.37 to 0.33], Standard Error of Mean 0.18
Statistical Analysis 26: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.094, ANCOVA; LS mean difference = -0.30, 95% CI 2-sided [-0.65 to 0.05], Standard Error of Mean 0.18
Statistical Analysis 27: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.012, ANCOVA; LS mean difference = -0.45, 95% CI 2-sided [-0.80 to -0.10], Standard Error of Mean 0.18
Statistical Analysis 28: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.363, ANCOVA; LS mean difference = -0.16, 95% CI 2-sided [-0.51 to 0.19], Standard Error of Mean 0.18
Statistical Analysis 29: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.742, ANCOVA; LS mean difference = 0.06, 95% CI 2-sided [-0.32 to 0.45], Standard Error of Mean 0.20
Statistical Analysis 30: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.436, ANCOVA; LS mean difference = -0.15, 95% CI 2-sided [-0.53 to 0.23], Standard Error of Mean 0.19
Statistical Analysis 31: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.038, ANCOVA; LS mean difference = -0.41, 95% CI 2-sided [-0.79 to -0.02], Standard Error of Mean 0.20
Statistical Analysis 32: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.332, ANCOVA; LS mean difference = -0.19, 95% CI 2-sided [-0.57 to 0.19], Standard Error of Mean 0.20
Statistical Analysis 33: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.284, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.47 to 0.14], Standard Error of Mean 0.16
Statistical Analysis 34: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.224, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.50 to 0.12], Standard Error of Mean 0.16
Statistical Analysis 35: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-0.79 to -0.17], Standard Error of Mean 0.16
Statistical Analysis 36: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.355, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.45 to 0.16], Standard Error of Mean 0.16
Statistical Analysis 37: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.172, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.57 to 0.10], Standard Error of Mean 0.17
Statistical Analysis 38: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.882, ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.36 to 0.31], Standard Error of Mean 0.17
Statistical Analysis 39: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.084, ANCOVA; LS Mean Difference = -0.29, 95% CI 2-sided [-0.63 to 0.04], Standard Error of Mean 0.17
Statistical Analysis 40: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.405, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.47 to 0.19], Standard Error of Mean 0.17
Statistical Analysis 41: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.67, 95% CI 2-sided [-0.99 to -0.34], Standard Error of Mean 0.16
Statistical Analysis 42: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.74, 95% CI 2-sided [-1.06 to -0.42], Standard Error of Mean 0.16
Statistical Analysis 43: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.96, 95% CI 2-sided [-1.29 to -0.64], Standard Error of Mean 0.16
Statistical Analysis 44: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.97, 95% CI 2-sided [-1.29 to -0.65], Standard Error of Mean 0.16
Statistical Analysis 45: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.60, 95% CI 2-sided [-0.95 to -0.25], Standard Error of Mean 0.18
Statistical Analysis 46: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.67, 95% CI 2-sided [-1.02 to -0.32], Standard Error of Mean 0.18
Statistical Analysis 47: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.87, 95% CI 2-sided [-1.22 to -0.51], Standard Error of Mean 0.18
Statistical Analysis 48: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.95, 95% CI 2-sided [-1.31 to -0.60], Standard Error of Mean 0.18
Statistical Analysis 49: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-0.86 to -0.18], Standard Error of Mean 0.17
Statistical Analysis 50: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.90, 95% CI 2-sided [-1.24 to -0.56], Standard Error of Mean 0.17
Statistical Analysis 51: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.92, 95% CI 2-sided [-1.26 to -0.57], Standard Error of Mean 0.18
Statistical Analysis 52: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.07, 95% CI 2-sided [-1.41 to -0.73], Standard Error of Mean 0.17
Statistical Analysis 53: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.70, 95% CI 2-sided [-1.06 to -0.33], Standard Error of Mean 0.19
Statistical Analysis 54: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.84, 95% CI 2-sided [-1.21 to -0.47], Standard Error of Mean 0.19
Statistical Analysis 55: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.99, 95% CI 2-sided [-1.36 to -0.63], Standard Error of Mean 0.19
Statistical Analysis 56: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.19, 95% CI 2-sided [-1.56 to -0.83], Standard Error of Mean 0.19
Statistical Analysis 57: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.001, ANCOVA; LS Mean Difference = -0.58, 95% CI 2-sided [-0.93 to -0.23], Standard Error of Mean 0.18
Statistical Analysis 58: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.88, 95% CI 2-sided [-1.24 to -0.53], Standard Error of Mean 0.18
Statistical Analysis 59: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.88, 95% CI 2-sided [-1.24 to -0.53], Standard Error of Mean 0.18
Statistical Analysis 60: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.05, 95% CI 2-sided [-1.40 to -0.70], Standard Error of Mean 0.18
Statistical Analysis 61: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.79, 95% CI 2-sided [-1.17 to -0.40], Standard Error of Mean 0.20
Statistical Analysis 62: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.72, 95% CI 2-sided [-1.11 to -0.34], Standard Error of Mean 0.20
Statistical Analysis 63: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.94, 95% CI 2-sided [-1.32 to -0.56], Standard Error of Mean 0.19
Statistical Analysis 64: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.13, 95% CI 2-sided [-1.51 to -0.75], Standard Error of Mean 0.20

7. Secondary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Score at Weeks 2, 4, 8, 12, 24, 32, 40, 48 and 56: Last Observation Carried Forward (LOCF)
Description: as for outcome 2
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 32, 40, 48, and 56
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo). Missing values were imputed using LOCF. Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 284 | 287 | 280 | 286 | 282 | 255 | 253 | 255 | 253 | 254
units on a scale
  Baseline | 6.46 (1.72) | 6.47 (1.61) | 6.57 (1.67) | 6.39 (1.62) | 6.32 (1.62) | 6.67 (1.60) | 6.58 (1.58) | 6.57 (1.72) | 6.39 (1.62) | 6.47 (1.59)
  Change at Week 2 | -1.10 (1.88) | -1.13 (1.90) | -1.44 (2.02) | -1.06 (2.07) | -0.90 (1.69) | -1.18 (2.01) | -0.95 (1.99) | -1.21 (1.96) | -1.02 (2.13) | -0.90 (1.67)
  Change at Week 4 | -1.70 (2.02) | -1.84 (1.87) | -2.08 (2.15) | -2.06 (2.11) | -1.04 (1.91) | -1.81 (2.30) | -1.75 (2.10) | -1.95 (2.24) | -1.91 (2.18) | -1.09 (1.83)
  Change at Week 8 | -1.69 (2.23) | -2.13 (2.06) | -2.23 (2.26) | -2.33 (2.21) | -1.11 (1.95) | -2.02 (2.37) | -2.08 (2.19) | -2.13 (2.29) | -2.29 (2.30) | -1.14 (1.96)
  Change at Week 12 | -2.02 (2.31) | -2.08 (2.12) | -2.40 (2.15) | -2.50 (2.36) | -1.31 (2.11) | -2.35 (2.48) | -2.31 (2.46) | -2.37 (2.44) | -2.50 (2.42) | -1.36 (2.05)
  Change at Week 24 | -2.04 (2.37) | -2.08 (2.22) | -2.22 (2.21) | -2.29 (2.46) | -1.49 (2.22) | -2.14 (2.42) | -2.24 (2.31) | -2.20 (2.45) | -2.44 (2.54) | -1.62 (2.22)
  Change at Week 32 | -1.87 (2.40) | -2.01 (2.29) | -2.15 (2.32) | -2.25 (2.46) | -1.53 (2.29) | -2.08 (2.47) | -2.16 (2.42) | -2.22 (2.56) | -2.20 (2.62) | -1.57 (2.23)
  Change at Week 40 | -1.87 (2.37) | -1.90 (2.40) | -1.95 (2.34) | -2.04 (2.48) | -1.44 (2.23) | -2.06 (2.48) | -2.04 (2.40) | -2.00 (2.59) | -2.18 (2.60) | -1.52 (2.24)
  Change at Week 48 | -1.82 (2.36) | -1.93 (2.43) | -1.90 (2.41) | -1.96 (2.39) | -1.39 (2.25) | -1.94 (2.44) | -1.97 (2.42) | -2.03 (2.56) | -2.05 (2.58) | -1.44 (2.23)
  Change at Week 56 | -1.82 (2.36) | -1.84 (2.41) | -1.88 (2.41) | -1.87 (2.38) | -1.34 (2.22) | -1.90 (2.36) | -1.78 (2.36) | -1.92 (2.54) | -2.05 (2.57) | -1.45 (2.24)
Statistical Analysis 1: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.887, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.33 to 0.28], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.046, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-0.62 to -0.01], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.771, ANCOVA; LS mean difference = 0.05, 95% CI 2-sided [-0.26 to 0.35], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.032, ANCOVA; LS mean difference = 0.34, 95% CI 2-sided [0.03 to 0.64], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.223, ANCOVA; LS mean difference = 0.21, 95% CI 2-sided [-0.13 to 0.54], Standard Error of Mean 0.17
Statistical Analysis 6: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.718, ANCOVA; LS mean difference = -0.06, 95% CI 2-sided [-0.39 to 0.27], Standard Error of Mean 0.17
Statistical Analysis 7: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.495, ANCOVA; LS mean difference = -0.12, 95% CI 2-sided [-0.45 to 0.22], Standard Error of Mean 0.17
Statistical Analysis 8: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.389, ANCOVA; LS mean difference = -0.14, 95% CI 2-sided [-0.47 to 0.18], Standard Error of Mean 0.16
Statistical Analysis 9: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.035, ANCOVA; LS mean difference = -0.35, 95% CI 2-sided [-0.68 to -0.02], Standard Error of Mean 0.17
Statistical Analysis 10: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.155, ANCOVA; LS mean difference = -0.23, 95% CI 2-sided [-0.56 to 0.09], Standard Error of Mean 0.16
Statistical Analysis 11: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.876, ANCOVA; LS mean difference = -0.03, 95% CI 2-sided [-0.35 to 0.30], Standard Error of Mean 0.17
Statistical Analysis 12: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.864, ANCOVA; LS mean difference = 0.03, 95% CI 2-sided [-0.33 to 0.39], Standard Error of Mean 0.18
Statistical Analysis 13: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.338, ANCOVA; LS mean difference = -0.18, 95% CI 2-sided [-0.54 to 0.18], Standard Error of Mean 0.18
Statistical Analysis 14: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.101, ANCOVA; LS mean difference = -0.30, 95% CI 2-sided [-0.66 to 0.06], Standard Error of Mean 0.18
Statistical Analysis 15: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.605, ANCOVA; LS mean difference = -0.09, 95% CI 2-sided [-0.46 to 0.27], Standard Error of Mean 0.18
Statistical Analysis 16: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.013, ANCOVA; LS mean difference = -0.43, 95% CI 2-sided [-0.78 to -0.09], Standard Error of Mean 0.17
Statistical Analysis 17: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.005, ANCOVA; LS mean difference = -0.50, 95% CI 2-sided [-0.84 to -0.15], Standard Error of Mean 0.18
Statistical Analysis 18: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.199, ANCOVA; LS mean difference = -0.22, 95% CI 2-sided [-0.57 to 0.12], Standard Error of Mean 0.17
Statistical Analysis 19: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.363, ANCOVA; LS mean difference = -0.16, 95% CI 2-sided [-0.50 to 0.18], Standard Error of Mean 0.18
Statistical Analysis 20: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.613, ANCOVA; LS Mean difference = -0.10, 95% CI 2-sided [-0.47 to 0.28], Standard Error of Mean 0.19
Statistical Analysis 21: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.416, ANCOVA; LS mean difference = -0.16, 95% CI 2-sided [-0.53 to 0.22], Standard Error of Mean 0.19
Statistical Analysis 22: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.143, ANCOVA; LS mean difference = -0.28, 95% CI 2-sided [-0.66 to 0.09], Standard Error of Mean 0.19
Statistical Analysis 23: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.245, ANCOVA; LS mean difference = -0.22, 95% CI 2-sided [-0.60 to 0.15], Standard Error of Mean 0.19
Statistical Analysis 24: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.745, ANCOVA; LS mean difference = -0.06, 95% CI 2-sided [-0.41 to 0.29], Standard Error of Mean 0.18
Statistical Analysis 25: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.062, ANCOVA; LS mean difference = -0.34, 95% CI 2-sided [-0.69 to 0.02], Standard Error of Mean 0.18
Statistical Analysis 26: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.014, ANCOVA; LS mean difference = -0.44, 95% CI 2-sided [-0.80 to -0.09], Standard Error of Mean 0.18
Statistical Analysis 27: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.367, ANCOVA; LS mean difference = -0.16, 95% CI 2-sided [-0.52 to 0.19], Standard Error of Mean 0.18
Statistical Analysis 28: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.995, ANCOVA; LS mean difference = -0.00, 95% CI 2-sided [-0.39 to 0.39], Standard Error of Mean 0.20
Statistical Analysis 29: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.735, ANCOVA; LS mean difference = -0.07, 95% CI 2-sided [-0.46 to 0.32], Standard Error of Mean 0.20
Statistical Analysis 30: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.169, ANCOVA; LS mean difference = -0.28, 95% CI 2-sided [-0.67 to 0.12], Standard Error of Mean 0.20
Statistical Analysis 31: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.295, ANCOVA; LS mean difference = -0.21, 95% CI 2-sided [-0.60 to 0.18], Standard Error of Mean 0.20
Statistical Analysis 32: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.284, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.47 to 0.14], Standard Error of Mean 0.16
Statistical Analysis 33: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.224, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.50 to 0.12], Standard Error of Mean 0.16
Statistical Analysis 34: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-0.79 to -0.17], Standard Error of Mean 0.16
Statistical Analysis 35: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.355, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.45 to 0.16], Standard Error of Mean 0.16
Statistical Analysis 36: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.172, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.57 to 0.10], Standard Error of Mean 0.17
Statistical Analysis 37: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.882, ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.36 to 0.31], Standard Error of Mean 0.17
Statistical Analysis 38: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.084, ANCOVA; LS Mean Difference = -0.29, 95% CI 2-sided [-0.63 to 0.04], Standard Error of Mean 0.17
Statistical Analysis 39: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.405, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.47 to 0.19], Standard Error of Mean 0.17
Statistical Analysis 40: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.62, 95% CI 2-sided [-0.94 to -0.30], Standard Error of Mean 0.17
Statistical Analysis 41: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.76, 95% CI 2-sided [-1.09 to -0.44], Standard Error of Mean 0.17
Statistical Analysis 42: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.97, 95% CI 2-sided [-1.30 to -0.64], Standard Error of Mean 0.17
Statistical Analysis 43: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.00, 95% CI 2-sided [-1.32 to -0.67], Standard Error of Mean 0.17
Statistical Analysis 44: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.66, 95% CI 2-sided [-1.02 to -0.30], Standard Error of Mean 0.18
Statistical Analysis 45: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.63, 95% CI 2-sided [-0.99 to -0.27], Standard Error of Mean 0.18
Statistical Analysis 46: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.83, 95% CI 2-sided [-1.19 to -0.48], Standard Error of Mean 0.18
Statistical Analysis 47: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.93, 95% CI 2-sided [-1.29 to -0.57], Standard Error of Mean 0.18
Statistical Analysis 48: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS Mean Difference = -0.54, 95% CI 2-sided [-0.89 to -0.20], Standard Error of Mean 0.18
Statistical Analysis 49: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.98, 95% CI 2-sided [-1.32 to -0.63], Standard Error of Mean 0.18
Statistical Analysis 50: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.04, 95% CI 2-sided [-1.39 to -0.70], Standard Error of Mean 0.18
Statistical Analysis 51: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.20, 95% CI 2-sided [-1.55 to -0.86], Standard Error of Mean 0.18
Statistical Analysis 52: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.80, 95% CI 2-sided [-1.18 to -0.43], Standard Error of Mean 0.19
Statistical Analysis 53: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.90, 95% CI 2-sided [-1.28 to -0.53], Standard Error of Mean 0.19
Statistical Analysis 54: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.96, 95% CI 2-sided [-1.33 to -0.58], Standard Error of Mean 0.19
Statistical Analysis 55: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.18, 95% CI 2-sided [-1.56 to -0.81], Standard Error of Mean 0.19
Statistical Analysis 56: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.66, 95% CI 2-sided [-1.02 to -0.31], Standard Error of Mean 0.18
Statistical Analysis 57: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.72, 95% CI 2-sided [-1.08 to -0.37], Standard Error of Mean 0.18
Statistical Analysis 58: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.00, 95% CI 2-sided [-1.36 to -0.65], Standard Error of Mean 0.18
Statistical Analysis 59: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -1.17, 95% CI 2-sided [-1.52 to -0.81], Standard Error of Mean 0.18
Statistical Analysis 60: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.90, 95% CI 2-sided [-1.29 to -0.51], Standard Error of Mean 0.20
Statistical Analysis 61: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.90, 95% CI 2-sided [-1.30 to -0.51], Standard Error of Mean 0.20
Statistical Analysis 62: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.97, 95% CI 2-sided [-1.36 to -0.58], Standard Error of Mean 0.20
Statistical Analysis 63: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.01, ANCOVA; LS Mean Difference = -1.18, 95% CI 2-sided [-1.57 to -0.79], Standard Error of Mean 0.20

8. Secondary Outcome: Change From Baseline in the Patient Global Assessment (PGA) of Osteoarthritis at Weeks 2, 4, 8, 12 and 24: Baseline Observation Carried Forward (BOCF)
Description: Patient global assessment of osteoarthritis was assessed by asking a question from participants: "Considering all the ways your osteoarthritis in your knee or hip affects you, how are you doing today?" Participants responded by using a 5-point likert scale ranging from 1=very good (asymptomatic and no limitation of normal activities, 2= mild symptoms and no limitation of normal activities, 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5 = very poor (Very severe symptoms which are intolerable and inability to carry out all normal activities). Higher scores indicating worse condition.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo). Missing values were imputed using BOCF. Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 284 | 288 | 280 | 285 | 283 | 256 | 254 | 255 | 253 | 254
units on a scale
  Change at Week 2 | -0.45 (0.80) | -0.42 (0.83) | -0.50 (0.81) | -0.40 (0.92) | -0.39 (0.71) | -0.46 (0.89) | -0.33 (0.88) | -0.45 (0.89) | -0.26 (0.85) | -0.37 (0.75)
  Change at Week 4 | -0.60 (0.78) | -0.69 (0.81) | -0.74 (0.86) | -0.68 (0.87) | -0.43 (0.80) | -0.68 (0.88) | -0.75 (0.92) | -0.80 (0.92) | -0.75 (0.84) | -0.49 (0.85)
  Change at Week 8 | -0.58 (0.89) | -0.70 (0.84) | -0.69 (0.87) | -0.82 (0.90) | -0.45 (0.81) | -0.63 (0.89) | -0.69 (0.85) | -0.81 (0.92) | -0.79 (0.82) | -0.51 (0.87)
  Change at Week 12 | -0.60 (0.89) | -0.68 (0.85) | -0.69 (0.88) | -0.84 (0.99) | -0.46 (0.89) | -0.71 (0.86) | -0.75 (0.88) | -0.77 (0.93) | -0.83 (0.89) | -0.54 (0.83)
  Change at Week 24 | -0.58 (0.97) | -0.54 (0.93) | -0.50 (0.82) | -0.60 (0.99) | -0.49 (0.82) | -0.57 (0.89) | -0.59 (0.82) | -0.67 (0.99) | -0.74 (0.90) | -0.55 (0.84)
Statistical Analysis 1: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.469, ANCOVA; LS mean difference = 0.04, 95% CI 2-sided [-0.08 to 0.17], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.387, ANCOVA; LS mean difference = -0.05, 95% CI 2-sided [-0.18 to 0.07], Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.887, ANCOVA; LS mean difference = 0.01, 95% CI 2-sided [-0.11 to 0.13], Standard Error of Mean 0.06
Statistical Analysis 4: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.084, ANCOVA; LS mean difference = 0.11, 95% CI 2-sided [-0.01 to 0.23], Standard Error of Mean 0.06
Statistical Analysis 5: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.018, ANCOVA; LS mean difference = 0.16, 95% CI 2-sided [0.03 to 0.29], Standard Error of Mean 0.07
Statistical Analysis 6: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.783, ANCOVA; LS mean difference = 0.02, 95% CI 2-sided [-0.11 to 0.15], Standard Error of Mean 0.07
Statistical Analysis 7: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.762, ANCOVA; LS mean difference = 0.02, 95% CI 2-sided [-0.11 to 0.15], Standard Error of Mean 0.07
Statistical Analysis 8: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.017, ANCOVA; LS mean difference = 0.16, 95% CI 2-sided [0.03 to 0.29], Standard Error of Mean 0.07
Statistical Analysis 9: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.207, ANCOVA; LS mean difference = -0.08, 95% CI 2-sided [-0.20 to 0.04], Standard Error of Mean 0.06
Statistical Analysis 10: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.020, ANCOVA; LS mean difference = -0.15, 95% CI 2-sided [-0.27 to -0.02], Standard Error of Mean 0.06
Statistical Analysis 11: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.941, ANCOVA; LS mean difference = -0.00, 95% CI 2-sided [-0.13 to 0.12], Standard Error of Mean 0.06
Statistical Analysis 12: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.494, ANCOVA; LS mean difference = -0.05, 95% CI 2-sided [-0.18 to 0.09], Standard Error of Mean 0.07
Statistical Analysis 13: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.089, ANCOVA; LS mean difference = -0.11, 95% CI 2-sided [-0.25 to 0.02], Standard Error of Mean 0.07
Statistical Analysis 14: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.467, ANCOVA; LS mean difference = -0.05, 95% CI 2-sided [-0.18 to 0.08], Standard Error of Mean 0.07
Statistical Analysis 15: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.774, ANCOVA; LS mean difference = 0.02, 95% CI 2-sided [-0.11 to 0.15], Standard Error of Mean 0.07
Statistical Analysis 16: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.315, ANCOVA; LS mean difference = 0.06, 95% CI 2-sided [-0.06 to 0.19], Standard Error of Mean 0.06
Statistical Analysis 17: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.088, ANCOVA; LS mean difference = -0.11, 95% CI 2-sided [-0.25 to 0.02], Standard Error of Mean 0.07
Statistical Analysis 18: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.084, ANCOVA; LS mean difference = -0.12, 95% CI 2-sided [-0.25 to 0.02], Standard Error of Mean 0.07
Statistical Analysis 19: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.066, ANCOVA; LS mean difference = -0.12, 95% CI 2-sided [-0.25 to 0.01], Standard Error of Mean 0.07
Statistical Analysis 20: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.073, ANCOVA; LS mean difference = -0.12, 95% CI 2-sided [-0.25 to 0.01], Standard Error of Mean 0.07
Statistical Analysis 21: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.682, ANCOVA; LS mean difference = -0.03, 95% CI 2-sided [-0.16 to 0.10], Standard Error of Mean 0.07
Statistical Analysis 22: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.014, ANCOVA; LS mean difference = -0.17, 95% CI 2-sided [-0.30 to -0.03], Standard Error of Mean 0.07
Statistical Analysis 23: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.027, ANCOVA; LS mean difference = -0.15, 95% CI 2-sided [-0.28 to -0.02], Standard Error of Mean 0.07
Statistical Analysis 24: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.871, ANCOVA; LS mean difference = -0.01, 95% CI 2-sided [-0.14 to 0.12], Standard Error of Mean 0.07
Statistical Analysis 25: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.301, ANCOVA; LS mean difference = -0.07, 95% CI 2-sided [-0.21 to 0.06], Standard Error of Mean 0.07
Statistical Analysis 26: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.181, ANCOVA; LS mean difference = -0.09, 95% CI 2-sided [-0.23 to 0.04], Standard Error of Mean 0.07
Statistical Analysis 27: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.013, ANCOVA; LS mean difference = -0.17, 95% CI 2-sided [-0.30 to -0.04], Standard Error of Mean 0.07
Statistical Analysis 28: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.031, ANCOVA; LS mean difference = -0.15, 95% CI 2-sided [-0.28 to -0.01], Standard Error of Mean 0.07
Statistical Analysis 29: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.874, ANCOVA; LS mean difference = -0.01, 95% CI 2-sided [-0.15 to 0.13], Standard Error of Mean 0.07
Statistical Analysis 30: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.447, ANCOVA; LS mean difference = -0.05, 95% CI 2-sided [-0.19 to 0.08], Standard Error of Mean 0.07
Statistical Analysis 31: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.059, ANCOVA; LS mean difference = -0.13, 95% CI 2-sided [-0.27 to 0.01], Standard Error of Mean 0.07
Statistical Analysis 32: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.196, ANCOVA; LS mean difference = -0.09, 95% CI 2-sided [-0.23 to 0.05], Standard Error of Mean 0.07
Statistical Analysis 33: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.360, ANCOVA; LS mean difference = -0.06, 95% CI 2-sided [-0.18 to 0.06], Standard Error of Mean 0.06
Statistical Analysis 34: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.845, ANCOVA; LS mean difference = -0.01, 95% CI 2-sided [-0.13 to 0.11], Standard Error of Mean 0.06
Statistical Analysis 35: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.076, ANCOVA; LS mean difference = -0.11, 95% CI 2-sided [-0.23 to 0.01], Standard Error of Mean 0.06
Statistical Analysis 36: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.957, ANCOVA; LS mean difference = -0.00, 95% CI 2-sided [-0.12 to 0.12], Standard Error of Mean 0.06
Statistical Analysis 37: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.404, ANCOVA; LS mean difference = -0.06, 95% CI 2-sided [-0.19 to 0.08], Standard Error of Mean 0.07
Statistical Analysis 38: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.128, ANCOVA; LS mean difference = 0.10, 95% CI 2-sided [-0.03 to 0.23], Standard Error of Mean 0.07
Statistical Analysis 39: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.577, ANCOVA; LS mean difference = -0.04, 95% CI 2-sided [-0.17 to 0.09], Standard Error of Mean 0.07
Statistical Analysis 40: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.068, ANCOVA; LS mean difference = 0.12, 95% CI 2-sided [-0.01 to 0.25], Standard Error of Mean 0.07
Statistical Analysis 41: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.011, ANCOVA; LS mean difference = -0.16, 95% CI 2-sided [-0.28 to -0.04], Standard Error of Mean 0.06
Statistical Analysis 42: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = -0.24, 95% CI 2-sided [-0.36 to -0.11], Standard Error of Mean 0.06
Statistical Analysis 43: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = -0.30, 95% CI 2-sided [-0.43 to -0.18], Standard Error of Mean 0.06
Statistical Analysis 44: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = -0.24, 95% CI 2-sided [-0.36 to -0.12], Standard Error of Mean 0.06
Statistical Analysis 45: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.043, ANCOVA; LS mean difference = -0.14, 95% CI 2-sided [-0.27 to -0.00], Standard Error of Mean 0.07
Statistical Analysis 46: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.007, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.31 to -0.05], Standard Error of Mean 0.07
Statistical Analysis 47: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.25, 95% CI 2-sided [-0.38 to -0.12], Standard Error of Mean 0.07
Statistical Analysis 48: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.36 to -0.10], Standard Error of Mean 0.07
Statistical Analysis 49: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.074, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.25 to 0.01], Standard Error of Mean 0.07
Statistical Analysis 50: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.37 to -0.10], Standard Error of Mean 0.07
Statistical Analysis 51: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.37 to -0.10], Standard Error of Mean 0.07
Statistical Analysis 52: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.36, 95% CI 2-sided [-0.49 to -0.23], Standard Error of Mean 0.07
Statistical Analysis 53: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.236, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.21 to 0.05], Standard Error of Mean 0.07
Statistical Analysis 54: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.112, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.24 to 0.02], Standard Error of Mean 0.07
Statistical Analysis 55: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.38 to -0.11], Standard Error of Mean 0.07
Statistical Analysis 56: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-0.39 to -0.12], Standard Error of Mean 0.07
Statistical Analysis 57: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.059, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.26 to 0.01], Standard Error of Mean 0.07
Statistical Analysis 58: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.33 to -0.07], Standard Error of Mean 0.07
Statistical Analysis 59: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.001, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.36 to -0.09], Standard Error of Mean 0.07
Statistical Analysis 60: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.37, 95% CI 2-sided [-0.51 to -0.24], Standard Error of Mean 0.07
Statistical Analysis 61: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.055, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.27 to 0.00], Standard Error of Mean 0.07
Statistical Analysis 62: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.038, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.28 to -0.01], Standard Error of Mean 0.07
Statistical Analysis 63: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.007, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.33 to -0.05], Standard Error of Mean 0.07
Statistical Analysis 64: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = -0.28, 95% CI 2-sided [-0.42 to -0.14], Standard Error of Mean 0.07

9. Secondary Outcome: Change From Baseline in the Patient Global Assessment (PGA) of Osteoarthritis at Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56: Last Observation Carried Forward (LOCF)
Description: as for outcome 8
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, and 56
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (tanezumab or matching placebo). Missing values were imputed using LOCF. Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 284 | 288 | 280 | 285 | 283 | 256 | 254 | 255 | 253 | 254
units on a scale
  Change at Week 2 | -0.45 (0.80) | -0.42 (0.83) | -0.50 (0.81) | -0.40 (0.92) | -0.39 (0.71) | -0.46 (0.89) | -0.33 (0.88) | -0.45 (0.89) | -0.26 (0.85) | -0.37 (0.75)
  Change at Week 4 | -0.60 (0.80) | -0.72 (0.82) | -0.76 (0.86) | -0.72 (0.90) | -0.44 (0.80) | -0.70 (0.91) | -0.76 (0.93) | -0.78 (0.95) | -0.74 (0.86) | -0.51 (0.85)
  Change at Week 8 | -0.63 (0.91) | -0.77 (0.87) | -0.75 (0.88) | -0.86 (0.95) | -0.48 (0.83) | -0.68 (0.91) | -0.74 (0.87) | -0.81 (0.94) | -0.81 (0.85) | -0.54 (0.90)
  Change at Week 12 | -0.67 (0.91) | -0.79 (0.89) | -0.78 (0.90) | -0.91 (1.04) | -0.49 (0.93) | -0.77 (0.90) | -0.84 (0.89) | -0.81 (0.95) | -0.86 (0.93) | -0.57 (0.88)
  Change at Week 16 | -0.63 (0.93) | -0.74 (0.95) | -0.72 (0.92) | -0.79 (1.07) | -0.57 (0.81) | -0.76 (0.91) | -0.73 (0.88) | -0.80 (0.96) | -0.77 (0.94) | -0.54 (0.92)
  Change at Week 24 | -0.69 (1.02) | -0.68 (1.00) | -0.64 (0.87) | -0.69 (1.07) | -0.57 (0.89) | -0.66 (0.96) | -0.69 (0.87) | -0.73 (1.02) | -0.77 (0.96) | -0.59 (0.93)
  Change at Week 32 | -0.60 (0.97) | -0.66 (0.95) | -0.60 (0.93) | -0.68 (1.16) | -0.57 (0.96) | -0.63 (1.02) | -0.66 (0.92) | -0.73 (0.91) | -0.66 (1.00) | -0.57 (0.92)
  Change at Week 40 | -0.58 (0.98) | -0.60 (0.98) | -0.53 (0.93) | -0.56 (1.10) | -0.50 (0.91) | -0.61 (1.03) | -0.67 (0.87) | -0.59 (1.00) | -0.66 (1.01) | -0.57 (0.94)
  Change at Week 48 | -0.53 (0.99) | -0.60 (0.98) | -0.51 (0.92) | -0.48 (1.09) | -0.49 (0.91) | -0.53 (1.04) | -0.62 (0.91) | -0.63 (0.98) | -0.59 (1.01) | -0.54 (0.95)
  Change at Week 56 | -0.53 (1.00) | -0.55 (0.95) | -0.49 (0.94) | -0.46 (1.09) | -0.47 (0.89) | -0.51 (1.01) | -0.56 (0.85) | -0.61 (1.00) | -0.58 (1.02) | -0.54 (0.96)
Statistical Analysis 1: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.469, ANCOVA; LS mean difference = 0.04, 95% CI 2-sided [-0.08 to 0.17], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.387, ANCOVA; LS mean difference = -0.05, 95% CI 2-sided [-0.18 to 0.07], Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.887, ANCOVA; LS mean difference = 0.01, 95% CI 2-sided [-0.11 to 0.13], Standard Error of Mean 0.06
Statistical Analysis 4: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.084, ANCOVA; LS mean difference = 0.11, 95% CI 2-sided [-0.01 to 0.23], Standard Error of Mean 0.06
Statistical Analysis 5: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.018, ANCOVA; LS mean difference = 0.16, 95% CI 2-sided [0.03 to 0.29], Standard Error of Mean 0.07
Statistical Analysis 6: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.783, ANCOVA; LS mean difference = 0.02, 95% CI 2-sided [-0.11 to 0.15], Standard Error of Mean 0.07
Statistical Analysis 7: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.762, ANCOVA; LS mean difference = 0.02, 95% CI 2-sided [-0.11 to 0.15], Standard Error of Mean 0.07
Statistical Analysis 8: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.017, ANCOVA; LS mean difference = 0.16, 95% CI 2-sided [0.03 to 0.29], Standard Error of Mean 0.07
Statistical Analysis 9: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.091, ANCOVA; LS mean difference = -0.11, 95% CI 2-sided [-0.23 to 0.02], Standard Error of Mean 0.06
Statistical Analysis 10: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.009, ANCOVA; LS mean difference = -0.16, 95% CI 2-sided [-0.29 to -0.04], Standard Error of Mean 0.06
Statistical Analysis 11: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.835, ANCOVA; LS mean difference = -0.01, 95% CI 2-sided [-0.13 to 0.11], Standard Error of Mean 0.06
Statistical Analysis 12: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.463, ANCOVA; LS mean difference = 0.05, 95% CI 2-sided [-0.08 to 0.17], Standard Error of Mean 0.06
Statistical Analysis 13: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.713, ANCOVA; LS mean difference = -0.02, 95% CI 2-sided [-0.16 to 0.11], Standard Error of Mean 0.07
Statistical Analysis 14: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.267, ANCOVA; LS mean difference = -0.08, 95% CI 2-sided [-0.21 to 0.06], Standard Error of Mean 0.07
Statistical Analysis 15: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.552, ANCOVA; LS mean difference = -0.04, 95% CI 2-sided [-0.17 to 0.09], Standard Error of Mean 0.07
Statistical Analysis 16: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.885, ANCOVA; LS mean difference = 0.01, 95% CI 2-sided [-0.12 to 0.14], Standard Error of Mean 0.07
Statistical Analysis 17: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.47, ANCOVA; LS mean difference = -0.13, 95% CI 2-sided [-0.26 to -0.00], Standard Error of Mean 0.07
Statistical Analysis 18: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.056, ANCOVA; LS mean difference = -0.13, 95% CI 2-sided [-0.26 to 0.00], Standard Error of Mean 0.07
Statistical Analysis 19: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.117, ANCOVA; LS mean difference = -0.10, 95% CI 2-sided [-0.24 to 0.03], Standard Error of Mean 0.07
Statistical Analysis 20: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.106, ANCOVA; LS mean difference = -0.11, 95% CI 2-sided [-0.24 to 0.02], Standard Error of Mean 0.07
Statistical Analysis 21: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.673, ANCOVA; LS mean difference = -0.03, 95% CI 2-sided [-0.16 to 0.10], Standard Error of Mean 0.07
Statistical Analysis 22: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.089, ANCOVA; LS mean difference = -0.11, 95% CI 2-sided [-0.25 to 0.02], Standard Error of Mean 0.07
Statistical Analysis 23: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.065, ANCOVA; LS mean difference = -0.12, 95% CI 2-sided [-0.26 to 0.01], Standard Error of Mean 0.07
Statistical Analysis 24: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.567, ANCOVA; LS mean difference = -0.04, 95% CI 2-sided [-0.17 to 0.09], Standard Error of Mean 0.07
Statistical Analysis 25: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 10 mg (Naproxen Exposure); [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.135, ANCOVA; LS mean difference = -0.10, 95% CI 2-sided [-0.24 to 0.03], Standard Error of Mean 0.07
Statistical Analysis 26: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Tanezumab 5 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.094, ANCOVA; LS mean difference = -0.12, 95% CI 2-sided [-0.25 to 0.02], Standard Error of Mean 0.07
Statistical Analysis 27: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.055, ANCOVA; LS mean difference = -0.13, 95% CI 2-sided [-0.27 to 0.00], Standard Error of Mean 0.07
Statistical Analysis 28: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Tanezumab 10 mg + Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.087, ANCOVA; LS mean difference = -0.12, 95% CI 2-sided [-0.25 to 0.02], Standard Error of Mean 0.07
Statistical Analysis 29: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 10 mg (Celecoxib Exposure); [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.542, ANCOVA; LS mean difference = -0.04, 95% CI 2-sided [-0.18 to 0.10], Standard Error of Mean 0.07
Statistical Analysis 30: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Tanezumab 5 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.643, ANCOVA; LS mean difference = -0.03, 95% CI 2-sided [-0.17 to 0.11], Standard Error of Mean 0.07
Statistical Analysis 31: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.301, ANCOVA; LS mean difference = -0.07, 95% CI 2-sided [-0.21 to 0.07], Standard Error of Mean 0.07
Statistical Analysis 32: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Tanezumab 10 mg + Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.237, ANCOVA; LS mean difference = -0.08, 95% CI 2-sided [-0.22 to 0.05], Standard Error of Mean 0.07
Statistical Analysis 33: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.360, ANCOVA; LS mean difference = -0.06, 95% CI 2-sided [-0.18 to 0.06], Standard Error of Mean 0.06
Statistical Analysis 34: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.854, ANCOVA; LS mean difference = -0.01, 95% CI 2-sided [-0.13 to 0.11], Standard Error of Mean 0.06
Statistical Analysis 35: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.076, ANCOVA; LS mean difference = -0.11, 95% CI 2-sided [-0.23 to 0.01], Standard Error of Mean 0.06
Statistical Analysis 36: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.957, ANCOVA; LS mean difference = -0.00, 95% CI 2-sided [-0.12 to 0.12], Standard Error of Mean 0.06
Statistical Analysis 37: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.404, ANCOVA; LS mean difference = -0.06, 95% CI 2-sided [-0.19 to 0.08], Standard Error of Mean 0.07
Statistical Analysis 38: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.128, ANCOVA; LS mean difference = 0.10, 95% CI 2-sided [-0.03 to 0.23], Standard Error of Mean 0.07
Statistical Analysis 39: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.577, ANCOVA; LS mean difference = -0.04, 95% CI 2-sided [-0.17 to 0.09], Standard Error of Mean 0.07
Statistical Analysis 40: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.068, ANCOVA; LS mean difference = 0.12, 95% CI 2-sided [-0.01 to 0.25], Standard Error of Mean 0.07
Statistical Analysis 41: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.016, ANCOVA; LS mean difference = -0.15, 95% CI 2-sided [-0.27 to -0.03], Standard Error of Mean 0.06
Statistical Analysis 42: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = -0.26, 95% CI 2-sided [-0.38 to -0.13], Standard Error of Mean 0.06
Statistical Analysis 43: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = -0.31, 95% CI 2-sided [-0.44 to -0.19], Standard Error of Mean 0.06
Statistical Analysis 44: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = -0.27, 95% CI 2-sided [-0.39 to -0.15], Standard Error of Mean 0.06
Statistical Analysis 45: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.037, ANCOVA; LS mean difference = -0.14, 95% CI 2-sided [-0.27 to -0.01], Standard Error of Mean 0.07
Statistical Analysis 46: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.015, ANCOVA; LS mean difference = -0.17, 95% CI 2-sided [-0.30 to -0.03], Standard Error of Mean 0.07
Statistical Analysis 47: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.001, ANCOVA; 0.07 = -0.22, 95% CI 2-sided [-0.35 to -0.08]
Statistical Analysis 48: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS mean difference = -0.21, 95% CI 2-sided [-0.34 to -0.07], Standard Error of Mean 0.07
Statistical Analysis 49: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.042, ANCOVA; LS mean difference = -0.14, 95% CI 2-sided [-0.27 to -0.00], Standard Error of Mean 0.07
Statistical Analysis 50: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = -0.27, 95% CI 2-sided [-0.40 to -0.14], Standard Error of Mean 0.07
Statistical Analysis 51: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = -0.26, 95% CI 2-sided [-0.40 to -0.13], Standard Error of Mean 0.07
Statistical Analysis 52: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = -0.37, 95% CI 2-sided [-0.50 to -0.24], Standard Error of Mean 0.07
Statistical Analysis 53: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.182, ANCOVA; LS mean difference = -0.09, 95% CI 2-sided [-0.22 to 0.04], Standard Error of Mean 0.07
Statistical Analysis 54: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.080, ANCOVA; LS mean difference = -0.12, 95% CI 2-sided [-0.25 to 0.01], Standard Error of Mean 0.07
Statistical Analysis 55: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p = 0.002, ANCOVA; LS mean difference = -0.20, 95% CI 2-sided [-0.34 to -0.07], Standard Error of Mean 0.07
Statistical Analysis 56: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 33]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = -0.24, 95% CI 2-sided [-0.37 to -0.11], Standard Error of Mean 0.07
Statistical Analysis 57: Comparison: Tanezumab 5 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.016, ANCOVA; LS mean difference = -0.17, 95% CI 2-sided [-0.30 to -0.03], Standard Error of Mean 0.07
Statistical Analysis 58: Comparison: Tanezumab 10 mg (Naproxen Exposure) vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = -0.27, 95% CI 2-sided [-0.40 to -0.13], Standard Error of Mean 0.07
Statistical Analysis 59: Comparison: Tanezumab 5 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = -0.28, 95% CI 2-sided [-0.42 to -0.15], Standard Error of Mean 0.07
Statistical Analysis 60: Comparison: Tanezumab 10 mg + Naproxen 500 mg vs Naproxen 500 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = -0.40, 95% CI 2-sided [-0.53 to -0.27], Standard Error of Mean 0.07
Statistical Analysis 61: Comparison: Tanezumab 5 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.032, ANCOVA; LS mean difference = -0.15, 95% CI 2-sided [-0.29 to -0.01], Standard Error of Mean 0.07
Statistical Analysis 62: Comparison: Tanezumab 10 mg (Celecoxib Exposure) vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.006, ANCOVA; LS mean difference = -0.19, 95% CI 2-sided [-0.33 to -0.06], Standard Error of Mean 0.07
Statistical Analysis 63: Comparison: Tanezumab 5 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p = 0.009, ANCOVA; LS mean difference = -0.18, 95% CI 2-sided [-0.32 to -0.05], Standard Error of Mean 0.07
Statistical Analysis 64: Comparison: Tanezumab 10 mg + Celecoxib 100 mg vs Celecoxib 100 mg; [analysis description as in outcome 4, analysis 49]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference = -0.27, 95% CI 2-sided [-0.41 to -0.13], Standard Error of Mean 0.07

10. Secondary Outcome: Percentage of Participants With Outcome Measures in Rheumatology - Osteoarthritis Research Society International (OMERACT-OARSI) Response: Baseline Observation Carried Forward (BOCF)
Description: Participants were considered as OMERACT-OARSI responder: if the improvement from baseline to week of interest was greater than or equal to (>=) 50 percent and >=2 units in WOMAC pain subscale or WOMAC physical function subscale score, or at least 2 of the following 3 being true: improvement from baseline to week of interest was >=20 percent and >=1 unit in 1) WOMAC pain subscale score, 2) WOMAC physical function subscale score, 3) PGA of osteoarthritis. WOMAC pain subscale assess amount of pain experienced (score: 0 [no pain] to 10 [worst possible pain], higher score = more pain), WOMAC physical function subscale assess degree of difficulty experienced (score: 0 [minimum difficulty] to 10 [maximum difficulty], higher score = worse physical function) and PGA of osteoarthritis (score: 1 [very good] to 5 [very poor], higher score = worse condition).
Time Frame: Weeks 2, 4, 8, 12, 16, and 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo). Missing values were imputed using BOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
percentage of participants
  Week 2 | 40.4 | 35.5 | 43.2 | 36.1 | 31.8 | 39.6 | 33.9 | 39.5 | 33.1 | 32.4
  Week 4 | 53.0 | 57.6 | 60.7 | 54.5 | 39.7 | 51.6 | 55.5 | 57.4 | 57.5 | 41.0
  Week 8 | 49.5 | 58.9 | 60.4 | 58.3 | 39.0 | 53.9 | 57.5 | 59.4 | 65.0 | 42.6
  Week 12 | 54.0 | 56.1 | 61.4 | 61.1 | 42.9 | 56.6 | 59.1 | 62.1 | 65.7 | 45.3
  Week 16 | 52.3 | 53.0 | 56.8 | 60.1 | 45.2 | 55.1 | 55.9 | 59.8 | 63.4 | 47.3
  Week 24 | 48.1 | 50.9 | 51.4 | 51.0 | 41.1 | 49.8 | 53.5 | 54.7 | 59.4 | 49.2

11. Secondary Outcome: Percentage of Participants With Outcome Measures in Rheumatology - Osteoarthritis Research Society International (OMERACT-OARSI) Response: Last Observation Carried Forward (LOCF)
Description: Participants were considered as OMERACT-OARSI responder: if the improvement from baseline to week of interest was >=50 percent and >=2 units in WOMAC pain subscale or WOMAC physical function subscale score, or at least 2 of the following 3 being true: improvement from baseline to week of interest was >=20 percent and >=1 unit in 1) WOMAC pain subscale score, 2) WOMAC physical function subscale score, 3) PGA of osteoarthritis. WOMAC pain subscale assess amount of pain experienced (score: 0 [no pain] to 10 [worst possible pain], higher score = more pain), WOMAC physical function subscale assess degree of difficulty experienced (score: 0 [minimum difficulty] to 10 [maximum difficulty], higher score = worse physical function) and PGA of osteoarthritis (score: 1 [very good] to 5 [very poor], higher score = worse condition).
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, and 56
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (tanezumab or matching placebo). Missing values were imputed using LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
percentage of participants
  Week 2 | 40.4 | 35.5 | 43.2 | 36.1 | 31.8 | 39.6 | 33.9 | 39.5 | 33.1 | 32.4
  Week 4 | 53.7 | 59.0 | 62.5 | 57.6 | 41.0 | 53.1 | 55.9 | 57.8 | 57.9 | 41.8
  Week 8 | 53.3 | 62.2 | 65.7 | 64.2 | 41.0 | 56.3 | 61.4 | 61.3 | 66.5 | 43.8
  Week 12 | 60.4 | 61.8 | 68.2 | 68.4 | 46.6 | 60.9 | 65.0 | 65.6 | 68.1 | 47.7
  Week 16 | 59.3 | 59.7 | 65.7 | 69.1 | 49.5 | 60.5 | 62.2 | 64.1 | 66.5 | 51.2
  Week 24 | 60.4 | 60.1 | 63.2 | 62.2 | 48.4 | 58.6 | 63.4 | 60.5 | 64.2 | 55.1
  Week 32 | 60.7 | 57.6 | 61.4 | 63.2 | 52.3 | 57.4 | 56.3 | 62.5 | 60.6 | 53.1
  Week 40 | 57.9 | 56.3 | 58.9 | 59.0 | 50.9 | 58.2 | 56.3 | 57.4 | 62.2 | 49.2
  Week 48 | 58.2 | 57.6 | 57.9 | 58.0 | 49.5 | 57.4 | 55.9 | 58.2 | 58.3 | 49.2
  Week 56 | 57.2 | 54.9 | 57.5 | 58.0 | 50.5 | 56.6 | 53.5 | 57.0 | 59.4 | 49.2

12. Secondary Outcome: Percentage of Participants With at Least 30 Percent (%), 50%, 70% and 90% Reduction in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score From Baseline at Weeks 2, 4, 8, 12, 16, and 24: BOCF
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis in index joint (knee or hip). The WOMAC pain subscale was a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in index joint (knee or hip) during past 48 hours. It was calculated as mean of the scores from 5 individual questions scored on a NRS of 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Total score range for WOMAC pain subscale score was 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Percentage of participants who experienced an improvement (reduction) of >=30%, >=50%, >=70%, or >=90% in the WOMAC pain subscale scores from Baseline were reported.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, and 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (tanezumab or matching placebo). Missing values were imputed using BOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
percentage of participants
  Week 2: >=30% Reduction | 28.4 | 26.8 | 35.0 | 24.9 | 22.7 | 28.0 | 22.8 | 30.6 | 26.0 | 24.7
  Week 2: >=50% Reduction | 17.5 | 17.1 | 20.4 | 16.1 | 12.8 | 12.6 | 13.8 | 17.3 | 18.5 | 11.0
  Week 2: >=70% Reduction | 5.6 | 8.7 | 6.4 | 7.4 | 5.3 | 7.1 | 6.3 | 7.8 | 8.3 | 5.5
  Week 2: >=90% Reduction | 1.1 | 1.4 | 2.9 | 1.8 | 1.1 | 2.4 | 1.2 | 1.2 | 3.1 | 1.6
  Week 4: >=30% Reduction | 40.7 | 45.6 | 52.1 | 47.7 | 29.8 | 39.8 | 41.7 | 49.0 | 50.4 | 31.0
  Week 4: >=50% Reduction | 24.6 | 30.0 | 27.5 | 32.3 | 19.5 | 22.4 | 26.0 | 30.2 | 32.7 | 18.4
  Week 4: >=70% Reduction | 11.9 | 12.5 | 15.0 | 17.5 | 6.7 | 13.8 | 11.4 | 16.5 | 19.3 | 7.1
  Week 4: >=90% Reduction | 2.1 | 3.1 | 6.8 | 4.2 | 2.5 | 4.3 | 3.9 | 6.3 | 5.5 | 1.0
  Week 8: >=30% Reduction | 43.9 | 49.8 | 49.3 | 49.8 | 29.8 | 44.1 | 45.7 | 51.0 | 55.9 | 30.2
  Week 8: >=50% Reduction | 27.7 | 33.8 | 29.6 | 35.1 | 16.7 | 27.2 | 29.9 | 33.7 | 36.2 | 18.8
  Week 8: >=70% Reduction | 13.7 | 16.4 | 18.2 | 21.1 | 8.2 | 13.8 | 16.5 | 18.8 | 23.2 | 9.0
  Week 8: >=90% Reduction | 4.2 | 3.8 | 6.4 | 7.7 | 2.1 | 5.1 | 6.7 | 6.3 | 7.1 | 2.7
  Week 12: >=30% Reduction | 45.6 | 46.3 | 53.2 | 54.4 | 34.0 | 48.0 | 52.0 | 53.7 | 58.3 | 36.5
  Week 12: >=50% Reduction | 30.2 | 32.8 | 32.1 | 39.3 | 19.5 | 33.5 | 35.8 | 37.6 | 41.7 | 21.6
  Week 12: >=70% Reduction | 14.4 | 16.0 | 18.6 | 23.9 | 7.8 | 19.3 | 19.3 | 20.8 | 23.6 | 9.0
  Week 12: >=90% Reduction | 6.3 | 6.3 | 6.8 | 9.8 | 2.8 | 4.7 | 7.9 | 7.1 | 10.6 | 2.4
  Week 16: >=30% Reduction | 44.6 | 47.0 | 49.6 | 54.0 | 36.2 | 48.0 | 48.8 | 52.9 | 54.3 | 39.2
  Week 16: >=50% Reduction | 27.4 | 32.8 | 34.3 | 36.5 | 19.9 | 35.0 | 35.0 | 37.6 | 42.5 | 24.3
  Week 16: >=70% Reduction | 15.1 | 17.4 | 15.0 | 24.9 | 7.8 | 20.1 | 18.1 | 22.0 | 24.8 | 9.8
  Week 16: >=90% Reduction | 6.0 | 6.3 | 6.8 | 8.4 | 2.5 | 7.5 | 5.9 | 7.8 | 12.6 | 2.7
  Week 24: >=30% Reduction | 40.4 | 44.9 | 44.3 | 46.0 | 36.5 | 42.5 | 46.5 | 47.1 | 53.5 | 41.6
  Week 24: >=50% Reduction | 27.7 | 31.7 | 28.2 | 34.4 | 21.3 | 30.3 | 33.5 | 35.3 | 41.3 | 25.9
  Week 24: >=70% Reduction | 14.0 | 17.4 | 16.4 | 21.4 | 11.7 | 15.4 | 18.5 | 21.6 | 23.6 | 11.4
  Week 24: >=90% Reduction | 6.7 | 7.3 | 6.4 | 6.0 | 3.5 | 7.5 | 7.1 | 7.5 | 11.8 | 3.9

13. Secondary Outcome: Percentage of Participants With at Least 30%, 50%, 70% and 90% Reduction in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score: Last Observation Carried Forward (LOCF)
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis of index joint (knee or hip). The WOMAC pain subscale was a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis of index joint (knee or hip) during past 48 hours. It was calculated as mean of the scores from 5 individual questions scored on a NRS of 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Total score range for WOMAC pain subscale score was 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Percentage of participants who experienced an improvement (reduction) of >=30 percent, >=50%, >=70%, or >=90% in the WOMAC pain subscale scores from Baseline were reported.
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, and 56
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
percentage of participants
  Week 2: >=30% Reduction | 28.4 | 26.8 | 35.0 | 24.9 | 22.7 | 28.0 | 22.8 | 30.6 | 26.0 | 24.7
  Week 2: >=50% Reduction | 17.5 | 17.1 | 20.4 | 16.1 | 12.8 | 12.6 | 13.8 | 17.3 | 18.5 | 11.0
  Week 2: >=70% Reduction | 5.6 | 8.7 | 6.4 | 7.4 | 5.3 | 7.1 | 6.3 | 7.8 | 8.3 | 5.5
  Week 2: >=90% Reduction | 1.1 | 1.4 | 2.9 | 1.8 | 1.1 | 2.4 | 1.2 | 1.2 | 3.1 | 1.6
  Week 4: >=30% Reduction | 41.1 | 46.3 | 53.2 | 49.8 | 30.5 | 41.3 | 41.7 | 49.8 | 50.4 | 31.0
  Week 4: >=50% Reduction | 24.6 | 30.7 | 27.9 | 33.7 | 20.2 | 23.6 | 26.0 | 30.6 | 32.7 | 18.4
  Week 4: >=70% Reduction | 11.9 | 12.5 | 15.0 | 17.9 | 6.7 | 14.2 | 11.4 | 16.9 | 19.3 | 7.1
  Week 4: >=90% Reduction | 2.1 | 3.1 | 6.8 | 4.6 | 2.5 | 4.7 | 3.9 | 6.3 | 5.5 | 1.0
  Week 8: >=30% Reduction | 46.3 | 51.9 | 53.9 | 55.1 | 31.2 | 46.5 | 48.8 | 52.9 | 56.7 | 31.0
  Week 8: >=50% Reduction | 29.1 | 35.2 | 31.4 | 38.9 | 17.7 | 28.7 | 30.7 | 34.5 | 37.0 | 18.8
  Week 8: >=70% Reduction | 14.4 | 16.7 | 19.3 | 22.8 | 8.5 | 14.6 | 17.3 | 19.2 | 23.6 | 9.0
  Week 8: >=90% Reduction | 4.2 | 4.2 | 6.4 | 8.4 | 2.1 | 5.9 | 7.1 | 6.3 | 7.5 | 2.7
  Week 12: >=30% Reduction | 49.8 | 50.9 | 59.3 | 60.7 | 36.9 | 52.8 | 57.1 | 57.3 | 60.2 | 37.6
  Week 12: >=50% Reduction | 32.6 | 35.5 | 34.3 | 43.5 | 21.3 | 36.6 | 37.8 | 39.2 | 42.9 | 22.0
  Week 12: >=70% Reduction | 15.4 | 16.4 | 19.6 | 26.0 | 8.5 | 20.5 | 20.9 | 21.6 | 24.0 | 9.0
  Week 12: >=90% Reduction | 6.3 | 6.6 | 7.1 | 10.5 | 2.8 | 5.1 | 8.7 | 7.1 | 11.0 | 2.4
  Week 16: >=30% Reduction | 49.1 | 52.3 | 56.8 | 61.8 | 39.7 | 52.4 | 53.9 | 56.9 | 57.1 | 41.6
  Week 16: >=50% Reduction | 30.2 | 35.9 | 37.5 | 41.8 | 21.6 | 38.2 | 36.6 | 39.2 | 43.7 | 25.5
  Week 16: >=70% Reduction | 16.1 | 18.1 | 16.8 | 27.4 | 8.5 | 20.9 | 19.7 | 22.7 | 24.8 | 9.8
  Week 16: >=90% Reduction | 6.0 | 6.6 | 7.5 | 9.1 | 2.5 | 7.9 | 6.7 | 7.8 | 12.6 | 2.7
  Week 24: >=30% Reduction | 49.5 | 53.0 | 54.3 | 55.8 | 42.9 | 49.2 | 53.9 | 52.5 | 57.9 | 45.5
  Week 24: >=50% Reduction | 34.0 | 36.2 | 33.2 | 40.7 | 25.2 | 34.3 | 35.4 | 37.6 | 43.3 | 27.8
  Week 24: >=70% Reduction | 16.8 | 18.5 | 19.6 | 24.6 | 13.1 | 16.5 | 20.5 | 22.7 | 24.0 | 11.4
  Week 24: >=90% Reduction | 7.4 | 7.7 | 7.5 | 7.4 | 4.3 | 7.9 | 7.9 | 7.8 | 11.8 | 3.9
  Week 32: >=30% Reduction | 49.5 | 52.3 | 53.6 | 56.5 | 44.3 | 49.6 | 51.6 | 52.5 | 53.5 | 43.1
  Week 32: >=50% Reduction | 30.2 | 33.8 | 33.9 | 42.5 | 27.3 | 35.4 | 36.2 | 39.2 | 39.4 | 28.2
  Week 32: >=70% Reduction | 18.2 | 17.8 | 16.1 | 22.1 | 12.1 | 19.3 | 21.7 | 21.6 | 22.0 | 12.5
  Week 32: >=90% Reduction | 5.6 | 7.0 | 5.4 | 8.4 | 5.0 | 7.9 | 9.1 | 10.6 | 12.6 | 2.4
  Week 40: >=30% Reduction | 49.5 | 50.9 | 51.8 | 52.6 | 42.2 | 49.2 | 50.8 | 49.8 | 53.9 | 41.6
  Week 40: >=50% Reduction | 31.9 | 31.7 | 30.4 | 38.2 | 25.5 | 34.3 | 31.1 | 33.3 | 39.0 | 29.0
  Week 40: >=70% Reduction | 16.1 | 17.4 | 15.7 | 19.3 | 9.2 | 17.7 | 20.5 | 19.6 | 21.7 | 11.4
  Week 40: >=90% Reduction | 5.3 | 5.6 | 4.6 | 5.6 | 3.2 | 7.5 | 5.9 | 8.6 | 9.4 | 2.4
  Week 48: >=30% Reduction | 48.8 | 51.6 | 51.4 | 51.9 | 40.4 | 48.4 | 49.2 | 50.2 | 51.2 | 42.0
  Week 48: >=50% Reduction | 30.9 | 30.7 | 30.4 | 36.5 | 23.4 | 30.7 | 31.9 | 33.7 | 37.0 | 27.1
  Week 48: >=70% Reduction | 17.2 | 16.0 | 15.4 | 18.9 | 11.0 | 16.1 | 18.9 | 20.4 | 20.5 | 11.8
  Week 48: >=90% Reduction | 5.6 | 5.9 | 4.6 | 6.7 | 3.9 | 5.9 | 5.5 | 7.5 | 9.4 | 2.7
  Week 56: >=30% Reduction | 47.7 | 50.2 | 51.4 | 52.6 | 40.4 | 46.9 | 46.5 | 47.8 | 52.0 | 41.6
  Week 56: >=50% Reduction | 30.2 | 28.9 | 28.6 | 36.1 | 22.7 | 29.9 | 28.7 | 31.8 | 37.8 | 27.5
  Week 56: >=70% Reduction | 16.5 | 15.3 | 16.1 | 17.9 | 9.9 | 14.2 | 16.5 | 18.4 | 20.5 | 12.5
  Week 56: >=90% Reduction | 6.0 | 5.2 | 4.6 | 6.3 | 3.2 | 5.1 | 4.7 | 7.5 | 8.7 | 2.4

14. Secondary Outcome: Number of Participants With Cumulative Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis of index joint (knee or hip). The WOMAC pain subscale was a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis of index joint (knee or hip) during past 48 hours. It was calculated as mean of the scores from 5 individual questions scored on a NRS of 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Total score range for WOMAC pain subscale score was 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Number of participants who experienced reduction (as percent) of >0% to >=100% from Baseline in WOMAC pain subscale scores at Week 16 were reported.
Time Frame: Baseline, Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (tanezumab or matching placebo). Missing values were imputed using BOCF. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 287 | 280 | 285 | 282 | 254 | 254 | 255 | 254 | 255
Participants
  >0% | 198 | 201 | 199 | 203 | 172 | 177 | 182 | 193 | 194 | 170
  >=10% | 179 | 184 | 183 | 194 | 153 | 162 | 167 | 176 | 184 | 150
  >=20% | 148 | 162 | 158 | 174 | 130 | 142 | 150 | 151 | 162 | 124
  >=30% | 127 | 135 | 139 | 154 | 102 | 122 | 124 | 135 | 138 | 100
  >=40% | 103 | 117 | 118 | 132 | 81 | 108 | 114 | 115 | 123 | 81
  >=50% | 78 | 94 | 96 | 104 | 56 | 89 | 89 | 96 | 108 | 62
  >=60% | 53 | 75 | 61 | 82 | 39 | 70 | 68 | 72 | 79 | 44
  >=70% | 43 | 50 | 42 | 71 | 22 | 51 | 46 | 56 | 63 | 25
  >=80% | 29 | 29 | 31 | 45 | 14 | 31 | 34 | 36 | 50 | 13
  >=90% | 17 | 18 | 19 | 24 | 7 | 19 | 15 | 20 | 32 | 7
  100% | 4 | 11 | 12 | 10 | 3 | 5 | 8 | 7 | 11 | 5

15. Secondary Outcome: Number of Participants With Cumulative Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score: Last Observation Carried Forward (LOCF)
Description: as for outcome 14
Time Frame: Baseline, Week 16
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
Participants
  >0% | 228 | 234 | 233 | 245 | 201 | 197 | 202 | 208 | 208 | 188
  >=10% | 203 | 210 | 215 | 229 | 175 | 179 | 184 | 188 | 197 | 162
  >=20% | 167 | 183 | 181 | 201 | 144 | 157 | 167 | 163 | 173 | 134
  >=30% | 140 | 150 | 159 | 176 | 112 | 133 | 137 | 145 | 145 | 106
  >=40% | 114 | 129 | 132 | 150 | 88 | 117 | 120 | 120 | 127 | 84
  >=50% | 86 | 103 | 105 | 119 | 61 | 97 | 93 | 100 | 111 | 65
  >=60% | 58 | 79 | 68 | 92 | 43 | 77 | 72 | 75 | 80 | 45
  >=70% | 46 | 52 | 47 | 78 | 24 | 53 | 50 | 58 | 63 | 25
  >=80% | 31 | 30 | 36 | 48 | 16 | 32 | 38 | 37 | 50 | 13
  >=90% | 17 | 19 | 21 | 26 | 7 | 20 | 17 | 20 | 32 | 7
  100% | 4 | 12 | 14 | 12 | 3 | 5 | 8 | 7 | 11 | 5

16. Secondary Outcome: Percentage of Participants With Improvement of At Least 2 Points in Patient's Global Assessment (PGA) of Osteoarthritis at Weeks 2, 4, 8, 12, 16, and 24: Baseline Observation Carried Forward (BOCF)
Description: Patient global assessment of osteoarthritis was assessed by asking a question from participants: "Considering all the ways your osteoarthritis in your knee or hip affects you, how are you doing today?" Participants responded by using a 5-point likert scale ranging from 1=very good (asymptomatic and no limitation of normal activities, 2= mild symptoms and no limitation of normal activities, 3= fair (moderate symptoms and limitation of some normal activities), 4= poor (severe symptoms and inability to carry out most normal activities), and 5 = very poor (Very severe symptoms which are intolerable and inability to carry out all normal activities). Higher scores indicating worse condition. Improvement signifies a decrease of at least 2 points on the 5-point scale relative to baseline value. Percentage of participants who showed an improvement of >=2 points on scale were reported.
Time Frame: Weeks 2, 4, 8, 12, 16, and 24
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
percentage of participants
  Week 2 | 9.9 | 10.1 | 8.2 | 10.9 | 6.4 | 11.3 | 9.4 | 12.5 | 5.9 | 6.3
  Week 4 | 10.2 | 13.5 | 17.5 | 15.1 | 10.6 | 19.1 | 18.5 | 18.8 | 14.6 | 10.6
  Week 8 | 14.1 | 18.4 | 18.2 | 19.3 | 9.2 | 15.6 | 16.5 | 19.6 | 17.4 | 11.8
  Week 12 | 15.5 | 17.4 | 18.2 | 25.3 | 12.7 | 17.2 | 17.7 | 20.8 | 22.1 | 12.2
  Week 16 | 14.8 | 19.1 | 16.4 | 22.5 | 10.6 | 18.4 | 15.4 | 20.0 | 18.2 | 13.4
  Week 24 | 17.6 | 18.1 | 12.1 | 18.6 | 14.1 | 13.3 | 12.6 | 18.8 | 20.9 | 13.0

17. Secondary Outcome: Percentage of Participants With Improvement of Atleast 2 Points in Patient's Global Assessment (PGA) of Osteoarthritis at Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, and 56: Last Observation Carried Forward (LOCF)
Description: as for outcome 16
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, and 56
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo). Missing values were imputed using LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
percentage of participants
  Week 2 | 9.9 | 10.1 | 8.2 | 10.9 | 6.4 | 11.3 | 9.4 | 12.5 | 5.9 | 6.3
  Week 4 | 10.6 | 14.2 | 17.9 | 16.1 | 10.6 | 20.3 | 18.9 | 18.8 | 14.6 | 11.0
  Week 8 | 15.1 | 20.5 | 19.3 | 20.7 | 9.9 | 17.2 | 18.5 | 19.6 | 18.2 | 13.0
  Week 12 | 16.9 | 20.8 | 20.4 | 27.0 | 13.8 | 19.1 | 20.9 | 21.6 | 23.3 | 13.4
  Week 16 | 16.5 | 22.6 | 18.9 | 24.2 | 12.0 | 21.1 | 18.1 | 20.8 | 19.4 | 14.6
  Week 24 | 20.1 | 22.2 | 15.4 | 21.4 | 16.3 | 16.8 | 15.4 | 20.4 | 22.5 | 15.0
  Week 32 | 14.4 | 18.8 | 16.4 | 23.2 | 15.5 | 19.1 | 16.5 | 19.2 | 20.2 | 15.0
  Week 40 | 14.8 | 17.4 | 13.9 | 18.9 | 14.1 | 18.4 | 15.0 | 18.4 | 20.6 | 15.4
  Week 48 | 14.4 | 16.7 | 12.9 | 16.1 | 14.5 | 17.2 | 14.6 | 18.8 | 17.4 | 14.6
  Week 56 | 14.4 | 15.3 | 13.6 | 15.8 | 13.4 | 14.8 | 11.8 | 18.4 | 17.8 | 15.0

18. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score at Weeks 2, 4, 8, 12, 16 and 24: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis of index joint (knee or hip). The WOMAC stiffness subscale was a 2-item questionnaire used to assess the amount of stiffness experienced due to osteoarthritis of the index joint (knee or hip) during the past 48 hours. Stiffness was defined as a sensation of decreased ease of movement in the index joint (knee or hip). It was calculated as mean of the scores from 2 individual questions scored on NRS of 0 (no stiffness) to 10 (worst stiffness), with higher scores indicate more stiffness. Total score range for WOMAC stiffness subscale score was 0 (no stiffness) to 10 (worst stiffness), where higher scores indicated more stiffness.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, and 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 284 | 287 | 280 | 286 | 281 | 255 | 254 | 255 | 254 | 255
units on a scale
  Baseline | 6.50 (2.00) | 6.66 (1.85) | 6.70 (1.88) | 6.42 (2.05) | 6.60 (1.73) | 6.62 (2.14) | 6.58 (2.04) | 6.47 (2.14) | 6.33 (2.01) | 6.39 (1.89)
  Change at Week 2 | -1.35 (2.43) | -1.32 (2.18) | -1.65 (2.44) | -1.19 (2.29) | -1.02 (1.98) | -1.35 (2.52) | -1.21 (2.40) | -1.41 (2.31) | -1.11 (2.44) | -0.82 (2.04)
  Change at Week 4 | -1.85 (2.46) | -2.10 (2.34) | -2.31 (2.51) | -2.19 (2.44) | -1.23 (2.17) | -1.94 (2.65) | -2.05 (2.49) | -2.15 (2.48) | -2.25 (2.43) | -1.00 (2.18)
  Change at Week 8 | -1.76 (2.60) | -2.26 (2.38) | -2.26 (2.66) | -2.31 (2.54) | -1.29 (2.24) | -2.02 (2.66) | -2.22 (2.59) | -2.28 (2.51) | -2.60 (2.51) | -1.13 (2.16)
  Change at Week 12 | -1.98 (2.64) | -2.14 (2.38) | -2.49 (2.52) | -2.42 (2.69) | -1.40 (2.27) | -2.38 (2.75) | -2.36 (2.87) | -2.42 (2.70) | -2.72 (2.54) | -1.23 (2.16)
  Change at Week 16 | -1.93 (2.55) | -2.15 (2.40) | -2.31 (2.57) | -2.40 (2.65) | -1.42 (2.22) | -2.14 (2.74) | -2.28 (2.68) | -2.35 (2.62) | -2.62 (2.64) | -1.34 (2.13)
  Change at Week 24 | -1.80 (2.62) | -1.96 (2.52) | -1.98 (2.57) | -2.04 (2.74) | -1.46 (2.28) | -1.97 (2.56) | -2.10 (2.64) | -2.08 (2.59) | -2.39 (2.59) | -1.38 (2.18)

19. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score at Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56: Last Observation Carried Forward (LOCF)
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis of index joint (knee or hip). The WOMAC stiffness subscale was a 2-item questionnaire used to assess the amount of stiffness experienced due to osteoarthritis in the index joint (knee or hip) during the past 48 hours. Stiffness was defined as a sensation of decreased ease of movement in the index joint (knee or hip). It was calculated as mean of the scores from 2 individual questions scored on NRS of 0 (no stiffness) to 10 (worst stiffness), with higher scores indicate more stiffness. Total score range for WOMAC stiffness subscale score was 0 (no stiffness) to 10 (worst stiffness), where higher scores indicated more stiffness.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, and 56
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 284 | 287 | 280 | 286 | 281 | 255 | 254 | 255 | 254 | 255
units on a scale
  Change at Week 2 | -1.35 (2.43) | -1.32 (2.18) | -1.65 (2.44) | -1.19 (2.29) | -1.02 (1.98) | -1.35 (2.52) | -1.21 (2.40) | -1.41 (2.31) | -1.11 (2.44) | -0.82 (2.04)
  Change at Week 4 | -1.88 (2.49) | -2.17 (2.33) | -2.34 (2.50) | -2.27 (2.46) | -1.26 (2.20) | -2.04 (2.71) | -2.03 (2.52) | -2.13 (2.53) | -2.22 (2.49) | -1.01 (2.18)
  Change at Week 8 | -1.88 (2.67) | -2.43 (2.38) | -2.44 (2.66) | -2.52 (2.53) | -1.35 (2.32) | -2.15 (2.75) | -2.30 (2.62) | -2.30 (2.62) | -2.58 (2.60) | -1.15 (2.18)
  Change at Week 12 | -2.18 (2.71) | -2.39 (2.38) | -2.71 (2.50) | -2.68 (2.69) | -1.52 (2.40) | -2.55 (2.92) | -2.49 (2.90) | -2.49 (2.79) | -2.76 (2.64) | -1.24 (2.23)
  Change at Week 16 | -2.16 (2.62) | -2.44 (2.38) | -2.64 (2.58) | -2.70 (2.67) | -1.58 (2.35) | -2.35 (2.91) | -2.41 (2.71) | -2.43 (2.77) | -2.68 (2.72) | -1.38 (2.25)
  Change at Week 24 | -2.22 (2.75) | -2.36 (2.50) | -2.48 (2.65) | -2.46 (2.81) | -1.75 (2.45) | -2.28 (2.78) | -2.37 (2.66) | -2.23 (2.78) | -2.55 (2.68) | -1.43 (2.33)
  Change at Week 32 | -2.07 (2.86) | -2.23 (2.51) | -2.36 (2.62) | -2.48 (2.80) | -1.80 (2.52) | -2.18 (2.79) | -2.31 (2.73) | -2.46 (2.79) | -2.31 (2.68) | -1.41 (2.37)
  Change at Week 40 | -2.05 (2.85) | -2.15 (2.63) | -2.13 (2.63) | -2.24 (2.76) | -1.69 (2.52) | -2.10 (2.83) | -2.20 (2.74) | -2.16 (2.74) | -2.26 (2.68) | -1.43 (2.47)
  Change at Week 48 | -2.03 (2.90) | -2.23 (2.71) | -2.11 (2.71) | -2.20 (2.71) | -1.69 (2.54) | -2.01 (2.80) | -2.10 (2.73) | -2.22 (2.80) | -2.17 (2.67) | -1.34 (2.45)
  Change at Week 56 | -1.99 (2.86) | -2.10 (2.66) | -2.07 (2.72) | -2.08 (2.74) | -1.63 (2.49) | -1.97 (2.80) | -1.94 (2.72) | -2.10 (2.76) | -2.14 (2.69) | -1.34 (2.47)

20. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Weeks 2, 4, 8, 12, 16 and 24: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis of index joint (knee or hip). Each item is scored on a 0 to 10 NRS scale, where higher scores indicate higher pain/stiffness or worse function. WOMAC average score was calculated as the mean of 3 WOMAC subscale scores (pain, physical function and stiffness). Total score range was 0 (no response) to 10 (worse response), where higher score indicated worse response.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, and 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (tanezumab or matching placebo). Missing values were imputed using BOCF. Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 286 | 283 | 255 | 254 | 256 | 254 | 255
units on a scale
  Baseline | 6.45 (1.62) | 6.54 (1.53) | 6.60 (1.58) | 6.38 (1.63) | 6.41 (1.51) | 6.60 (1.58) | 6.54 (1.54) | 6.48 (1.70) | 6.33 (1.59) | 6.38 (1.55)
  Change at Week 2 | -1.13 (1.90) | -1.15 (1.86) | -1.46 (2.03) | -1.04 (2.03) | -0.93 (1.69) | -1.17 (2.05) | -0.98 (2.01) | -1.23 (1.94) | -0.99 (2.12) | -0.89 (1.65)
  Change at Week 4 | -1.74 (2.04) | -1.92 (1.91) | -2.15 (2.15) | -2.06 (2.11) | -1.13 (1.91) | -1.79 (2.30) | -1.87 (2.07) | -2.08 (2.20) | -2.10 (2.17) | -1.06 (1.85)
  Change at Week 8 | -1.68 (2.21) | -2.11 (2.05) | -2.14 (2.27) | -2.22 (2.20) | -1.15 (1.94) | -1.93 (2.30) | -2.08 (2.22) | -2.23 (2.19) | -2.42 (2.25) | -1.14 (1.91)
  Change at Week 12 | -1.90 (2.26) | -1.98 (2.08) | -2.31 (2.18) | -2.35 (2.33) | -1.27 (2.02) | -2.26 (2.40) | -2.24 (2.52) | -2.35 (2.36) | -2.55 (2.30) | -1.33 (1.89)
  Change at Week 16 | -1.84 (2.17) | -1.98 (2.17) | -2.17 (2.19) | -2.28 (2.29) | -1.34 (1.99) | -2.13 (2.39) | -2.17 (2.35) | -2.30 (2.36) | -2.48 (2.42) | -1.42 (1.94)
  Change at Week 24 | -1.70 (2.29) | -1.84 (2.19) | -1.87 (2.17) | -1.99 (2.38) | -1.34 (2.06) | -1.90 (2.28) | -2.05 (2.31) | -2.09 (2.35) | -2.33 (2.42) | -1.53 (2.00)

21. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56: Last Observation Carried Forward (LOCF)
Description: as for outcome 20
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, and 56
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 286 | 283 | 255 | 254 | 256 | 254 | 255
units on a scale
  Change at Week 2 | -1.13 (1.90) | -1.15 (1.86) | -1.46 (2.03) | -1.04 (2.03) | -0.93 (1.69) | -1.17 (2.05) | -0.98 (2.01) | -1.23 (1.94) | -0.99 (2.12) | -0.89 (1.65)
  Change at Week 4 | -1.74 (2.06) | -1.98 (1.90) | -2.18 (2.13) | -2.13 (2.13) | -1.15 (1.95) | -1.87 (2.36) | -1.84 (2.12) | -2.06 (2.26) | -2.07 (2.23) | -1.07 (1.85)
  Change at Week 8 | -1.78 (2.26) | -2.25 (2.05) | -2.31 (2.26) | -2.41 (2.19) | -1.20 (2.01) | -2.03 (2.39) | -2.15 (2.25) | -2.22 (2.29) | -2.41 (2.34) | -1.16 (1.94)
  Change at Week 12 | -2.08 (2.31) | -2.20 (2.09) | -2.52 (2.14) | -2.58 (2.32) | -1.37 (2.14) | -2.40 (2.52) | -2.37 (2.55) | -2.40 (2.44) | -2.59 (2.39) | -1.33 (1.97)
  Change at Week 16 | -2.05 (2.22) | -2.24 (2.16) | -2.48 (2.17) | -2.57 (2.27) | -1.45 (2.10) | -2.31 (2.51) | -2.29 (2.38) | -2.36 (2.46) | -2.53 (2.48) | -1.45 (2.03)
  Change at Week 24 | -2.10 (2.37) | -2.18 (2.19) | -2.30 (2.22) | -2.36 (2.40) | -1.58 (2.24) | -2.16 (2.41) | -2.28 (2.33) | -2.22 (2.45) | -2.46 (2.49) | -1.58 (2.13)
  Change at Week 32 | -1.96 (2.44) | -2.10 (2.24) | -2.20 (2.26) | -2.35 (2.42) | -1.64 (2.29) | -2.10 (2.44) | -2.20 (2.44) | -2.30 (2.51) | -2.22 (2.52) | -1.53 (2.15)
  Change at Week 40 | -1.94 (2.43) | -1.99 (2.35) | -1.99 (2.31) | -2.14 (2.40) | -1.51 (2.26) | -2.05 (2.43) | -2.07 (2.39) | -2.05 (2.50) | -2.20 (2.48) | -1.49 (2.16)
  Change at Week 48 | -1.91 (2.44) | -2.02 (2.39) | -1.96 (2.36) | -2.08 (2.33) | -1.48 (2.28) | -1.94 (2.40) | -2.00 (2.40) | -2.10 (2.50) | -2.08 (2.48) | -1.40 (2.16)
  Change at Week 56 | -1.89 (2.43) | -1.93 (2.36) | -1.93 (2.36) | -1.99 (2.32) | -1.43 (2.25) | -1.90 (2.33) | -1.81 (2.36) | -1.98 (2.46) | -2.07 (2.48) | -1.42 (2.18)

22. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item: Pain When Walking on a Flat Surface at Weeks 2, 4, 8, 12, 16 and 24: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis in index joint (knee or hip). Participants responded about the amount of pain they experienced when walking on a flat surface by answering the question: "How much pain have you had when walking on a flat surface?". Participants responded by using a NRS of 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, and 24
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 287 | 280 | 286 | 282 | 254 | 254 | 256 | 254 | 255
units on a scale
  Baseline | 6.22 (1.83) | 6.37 (1.97) | 6.34 (1.87) | 6.13 (1.96) | 6.12 (2.08) | 6.28 (1.83) | 6.30 (1.88) | 6.21 (1.97) | 6.14 (1.97) | 6.10 (1.83)
  Change at Week 2 | -1.05 (2.24) | -1.02 (2.43) | -1.31 (2.24) | -0.87 (2.43) | -0.80 (2.08) | -1.04 (2.34) | -0.68 (2.49) | -1.01 (2.24) | -0.86 (2.51) | -0.86 (2.04)
  Change at Week 4 | -1.67 (2.37) | -1.88 (2.39) | -1.98 (2.19) | -1.92 (2.34) | -1.04 (2.47) | -1.49 (2.58) | -1.64 (2.44) | -1.88 (2.53) | -1.93 (2.45) | -0.95 (2.27)
  Change at Week 8 | -1.57 (2.64) | -1.95 (2.51) | -1.93 (2.53) | -2.09 (2.50) | -1.05 (2.33) | -1.67 (2.50) | -1.84 (2.50) | -2.11 (2.44) | -2.26 (2.58) | -1.11 (2.40)
  Change at Week 12 | -1.74 (2.53) | -1.78 (2.38) | -2.15 (2.38) | -2.22 (2.51) | -1.10 (2.34) | -2.04 (2.54) | -2.02 (2.84) | -2.20 (2.73) | -2.25 (2.61) | -1.35 (2.24)
  Change at Week 16 | -1.71 (2.40) | -1.77 (2.61) | -1.95 (2.49) | -2.19 (2.49) | -1.23 (2.32) | -1.94 (2.69) | -1.91 (2.66) | -2.08 (2.75) | -2.22 (2.69) | -1.38 (2.28)
  Change at Week 24 | -1.56 (2.49) | -1.65 (2.47) | -1.64 (2.47) | -1.83 (2.51) | -1.20 (2.33) | -1.63 (2.61) | -1.88 (2.65) | -1.96 (2.71) | -2.06 (2.72) | -1.55 (2.33)

23. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item: Pain When Walking on a Flat Surface at Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56: Last Observation Carried Forward (LOCF)
Description: as for outcome 22
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, and 56
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 287 | 280 | 286 | 282 | 254 | 254 | 256 | 254 | 255
units on a scale
  Change at Week 2 | -1.05 (2.24) | -1.02 (2.43) | -1.31 (2.24) | -0.87 (2.43) | -0.80 (2.08) | -1.04 (2.34) | -0.68 (2.49) | -1.01 (2.24) | -0.86 (2.51) | -0.86 (2.04)
  Change at Week 4 | -1.65 (2.40) | -1.92 (2.41) | -2.01 (2.18) | -1.99 (2.36) | -1.04 (2.51) | -1.54 (2.65) | -1.59 (2.51) | -1.84 (2.62) | -1.91 (2.51) | -0.96 (2.28)
  Change at Week 8 | -1.65 (2.69) | -2.09 (2.62) | -2.08 (2.53) | -2.26 (2.52) | -1.07 (2.45) | -1.73 (2.64) | -1.85 (2.62) | -2.06 (2.60) | -2.22 (2.71) | -1.13 (2.45)
  Change at Week 12 | -1.93 (2.62) | -1.98 (2.53) | -2.32 (2.38) | -2.41 (2.57) | -1.20 (2.54) | -2.11 (2.71) | -2.08 (2.97) | -2.20 (2.86) | -2.27 (2.76) | -1.36 (2.33)
  Change at Week 16 | -1.93 (2.50) | -2.00 (2.74) | -2.20 (2.55) | -2.44 (2.51) | -1.33 (2.52) | -2.03 (2.85) | -1.98 (2.81) | -2.11 (2.91) | -2.25 (2.83) | -1.42 (2.41)
  Change at Week 24 | -1.95 (2.64) | -1.94 (2.68) | -1.98 (2.61) | -2.15 (2.59) | -1.36 (2.62) | -1.79 (2.79) | -1.97 (2.86) | -2.04 (2.89) | -2.15 (2.87) | -1.64 (2.52)
  Change at Week 32 | -1.78 (2.72) | -1.80 (2.85) | -1.91 (2.61) | -2.12 (2.67) | -1.45 (2.71) | -1.78 (2.87) | -1.80 (2.99) | -1.96 (2.89) | -1.89 (3.00) | -1.56 (2.48)
  Change at Week 40 | -1.69 (2.76) | -1.78 (2.92) | -1.69 (2.69) | -1.77 (2.71) | -1.23 (2.66) | -1.72 (2.75) | -1.75 (2.84) | -1.73 (2.92) | -1.89 (2.95) | -1.40 (2.53)
  Change at Week 48 | -1.63 (2.81) | -1.72 (2.92) | -1.68 (2.76) | -1.78 (2.64) | -1.22 (2.67) | -1.62 (2.72) | -1.64 (2.92) | -1.79 (2.90) | -1.74 (2.98) | -1.33 (2.60)
  Change at Week 56 | -1.65 (2.79) | -1.64 (2.92) | -1.68 (2.76) | -1.73 (2.63) | -1.15 (2.62) | -1.61 (2.62) | -1.42 (2.89) | -1.67 (2.92) | -1.72 (2.94) | -1.36 (2.63)

24. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item: Pain When Going Up or Down Stairs at Weeks 2, 4, 8, 12, 16 and 24: Baseline Observation Carried Forward (BOCF)
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness and physical function in participants with osteoarthritis of index joint (knee or hip). Participants responded about the amount of pain they experienced when going up or down stairs by answering the question: "How much pain have you had when going up or down the stairs?" Participants responded by using a NRS of 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, and 24
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 287 | 280 | 286 | 282 | 254 | 254 | 256 | 254 | 255
units on a scale
  Baseline | 7.55 (1.80) | 7.68 (1.78) | 7.72 (1.69) | 7.50 (1.73) | 7.40 (1.87) | 7.80 (1.71) | 7.59 (1.77) | 7.55 (1.77) | 7.54 (1.78) | 7.52 (1.70)
  Change at Week 2 | -1.29 (2.23) | -1.34 (2.33) | -1.67 (2.39) | -1.36 (2.42) | -0.94 (2.19) | -1.41 (2.39) | -1.23 (2.31) | -1.45 (2.43) | -1.37 (2.18) | -1.05 (2.08)
  Change at Week 4 | -1.78 (2.31) | -2.13 (2.30) | -2.46 (2.55) | -2.32 (2.44) | -1.22 (2.38) | -2.05 (2.65) | -2.07 (2.35) | -2.43 (2.63) | -2.36 (2.43) | -1.29 (2.21)
  Change at Week 8 | -1.79 (2.50) | -2.32 (2.49) | -2.41 (2.62) | -2.53 (2.60) | -1.34 (2.27) | -2.17 (2.63) | -2.26 (2.58) | -2.48 (2.56) | -2.65 (2.59) | -1.33 (2.04)
  Change at Week 12 | -2.09 (2.69) | -2.16 (2.59) | -2.49 (2.57) | -2.67 (2.66) | -1.37 (2.37) | -2.45 (2.71) | -2.52 (2.78) | -2.48 (2.72) | -2.79 (2.64) | -1.50 (2.10)
  Change at Week 16 | -1.99 (2.60) | -2.20 (2.65) | -2.35 (2.47) | -2.53 (2.64) | -1.53 (2.29) | -2.39 (2.71) | -2.35 (2.68) | -2.52 (2.76) | -2.76 (2.77) | -1.66 (2.17)
  Change at Week 24 | -1.82 (2.66) | -2.01 (2.67) | -2.02 (2.52) | -2.22 (2.74) | -1.51 (2.28) | -2.02 (2.74) | -2.28 (2.63) | -2.47 (2.90) | -2.63 (2.76) | -1.73 (2.33)

25. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Item: Pain When Going Up or Down Stairs at Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56: Last Observation Carried Forward (LOCF)
Description: as for outcome 24
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, and 56
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 287 | 280 | 286 | 282 | 254 | 254 | 256 | 254 | 255
units on a scale
  Change at Week 2 | -1.29 (2.23) | -1.34 (2.33) | -1.67 (2.39) | -1.36 (2.42) | -0.94 (2.19) | -1.41 (2.39) | -1.23 (2.31) | -1.45 (2.43) | -1.37 (2.18) | -1.05 (2.08)
  Change at Week 4 | -1.80 (2.31) | -2.20 (2.31) | -2.51 (2.55) | -2.41 (2.44) | -1.26 (2.39) | -2.14 (2.68) | -2.05 (2.39) | -2.43 (2.70) | -2.37 (2.44) | -1.30 (2.20)
  Change at Week 8 | -1.90 (2.55) | -2.48 (2.52) | -2.62 (2.61) | -2.75 (2.59) | -1.35 (2.37) | -2.27 (2.68) | -2.37 (2.61) | -2.50 (2.67) | -2.71 (2.60) | -1.35 (2.08)
  Change at Week 12 | -2.29 (2.70) | -2.40 (2.60) | -2.76 (2.52) | -2.94 (2.65) | -1.47 (2.52) | -2.64 (2.78) | -2.69 (2.83) | -2.57 (2.81) | -2.90 (2.64) | -1.55 (2.17)
  Change at Week 16 | -2.23 (2.63) | -2.47 (2.65) | -2.70 (2.45) | -2.88 (2.59) | -1.63 (2.46) | -2.62 (2.78) | -2.53 (2.73) | -2.59 (2.87) | -2.89 (2.75) | -1.75 (2.24)
  Change at Week 24 | -2.26 (2.73) | -2.38 (2.71) | -2.48 (2.55) | -2.66 (2.73) | -1.74 (2.53) | -2.35 (2.84) | -2.57 (2.71) | -2.60 (2.99) | -2.83 (2.78) | -1.84 (2.44)
  Change at Week 32 | -2.12 (2.75) | -2.28 (2.74) | -2.43 (2.72) | -2.62 (2.84) | -1.70 (2.52) | -2.27 (2.80) | -2.50 (2.84) | -2.52 (2.98) | -2.55 (2.90) | -1.78 (2.48)
  Change at Week 40 | -2.06 (2.66) | -2.21 (2.73) | -2.09 (2.59) | -2.41 (2.80) | -1.51 (2.45) | -2.31 (2.78) | -2.28 (2.77) | -2.26 (2.95) | -2.47 (2.87) | -1.76 (2.46)
  Change at Week 48 | -1.99 (2.69) | -2.17 (2.74) | -2.10 (2.74) | -2.29 (2.74) | -1.48 (2.47) | -2.20 (2.79) | -2.24 (2.84) | -2.30 (2.91) | -2.31 (2.89) | -1.64 (2.47)
  Change at Week 56 | -2.00 (2.70) | -2.08 (2.76) | -2.10 (2.72) | -2.24 (2.70) | -1.43 (2.45) | -2.16 (2.75) | -1.98 (2.78) | -2.16 (2.89) | -2.34 (2.84) | -1.71 (2.51)

26. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) at Week 12 and 24: Baseline Observation Carried Forward (BOCF)
Description: The SF-36 health survey is a self-administered questionnaire that measures each of the following 8 health domains: domain 1= general health, domain 2= physical function, domain 3= role physical, domain 4= bodily pain, domain 5= vitality, domain 6= social function, domain 7= role emotional, domain 8= mental health. Total score for each domain are scaled 0 (minimum) to 100 (maximum), where higher scores represent better health status.
Time Frame: Baseline, Weeks 12 and 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo). Missing values were imputed using BOCF. 'Number analyzed' signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
units on a scale
  General health at baseline: number analyzed (Participants) | 284 | 288 | 280 | 285 | 279 | 254 | 254 | 255 | 253 | 255
  General health at baseline | 56.76 (20.74) | 57.41 (21.03) | 60.66 (20.88) | 57.92 (22.08) | 57.61 (21.97) | 56.20 (20.62) | 56.93 (20.48) | 56.34 (20.39) | 58.27 (20.65) | 55.69 (22.22)
  Physical function at baseline: number analyzed (Participants) | 282 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Physical function at baseline | 32.82 (19.12) | 32.74 (21.34) | 34.79 (20.63) | 33.88 (18.66) | 35.46 (19.94) | 33.43 (20.62) | 34.79 (19.21) | 33.41 (22.07) | 35.11 (20.48) | 32.81 (19.57)
  Role physical at baseline: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Role physical at baseline | 43.29 (25.54) | 43.88 (23.81) | 44.58 (23.90) | 44.69 (23.60) | 46.09 (24.57) | 42.59 (23.69) | 42.86 (23.46) | 42.65 (24.90) | 45.60 (22.57) | 43.55 (22.70)
  Bodily pain at baseline: number analyzed (Participants) | 284 | 287 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 255
  Bodily pain at baseline | 36.91 (17.91) | 35.90 (17.87) | 37.80 (17.49) | 37.67 (17.89) | 35.72 (16.34) | 34.14 (16.39) | 35.57 (18.00) | 34.11 (16.66) | 36.47 (16.93) | 36.96 (17.60)
  Vitality at baseline: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 253 | 255 | 253 | 255
  Vitality at baseline | 51.58 (19.45) | 51.28 (20.10) | 53.73 (19.83) | 52.57 (19.76) | 50.78 (18.94) | 50.52 (18.21) | 51.52 (21.07) | 51.45 (19.16) | 53.63 (18.42) | 51.52 (17.90)
  Social function at baseline: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 255
  Social function at baseline | 65.63 (25.65) | 65.97 (26.68) | 68.13 (24.43) | 64.47 (25.28) | 62.23 (26.33) | 63.19 (24.26) | 63.68 (25.44) | 64.51 (24.58) | 66.90 (24.16) | 64.31 (24.07)
  Role emotional at baseline: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 254 | 253 | 255
  Role emotional at baseline | 66.08 (29.30) | 66.35 (28.15) | 67.74 (29.39) | 67.92 (29.42) | 68.45 (28.65) | 63.02 (28.66) | 64.07 (28.31) | 62.68 (29.21) | 65.05 (28.53) | 63.39 (28.73)
  Mental health at baseline: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 253 | 255 | 253 | 255
  Mental health at baseline | 70.42 (19.16) | 70.23 (19.71) | 72.20 (19.67) | 70.40 (18.77) | 70.34 (19.78) | 70.95 (17.94) | 71.08 (19.16) | 68.25 (19.23) | 71.07 (19.83) | 69.08 (18.69)
  Change at Week 12: General health: number analyzed (Participants) | 284 | 288 | 280 | 285 | 279 | 254 | 254 | 255 | 253 | 255
  Change at Week 12: General health | 3.29 (14.32) | 4.66 (15.19) | 3.66 (15.27) | 5.14 (15.96) | 3.88 (15.25) | 5.46 (14.25) | 3.37 (15.13) | 5.18 (13.96) | 5.66 (16.53) | 4.68 (16.00)
  Change at Week 12: Physical function: number analyzed (Participants) | 282 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 12: Physical function | 11.68 (22.48) | 12.88 (21.49) | 14.23 (25.26) | 14.38 (24.59) | 5.76 (21.38) | 12.70 (22.24) | 9.05 (22.01) | 13.84 (24.37) | 12.99 (24.30) | 7.48 (18.88)
  Change at Week 12: Role physical: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 12: Role physical | 9.73 (25.90) | 12.59 (24.75) | 13.13 (24.85) | 15.39 (26.13) | 6.70 (23.58) | 13.36 (25.67) | 10.04 (26.31) | 15.51 (26.62) | 13.71 (25.39) | 7.58 (23.58)
  Change at Week 12: Bodily pain: number analyzed (Participants) | 284 | 287 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 255
  Change at Week 12: Bodily pain | 11.44 (21.66) | 13.08 (21.93) | 14.41 (22.41) | 16.53 (22.55) | 7.83 (19.22) | 16.74 (21.52) | 12.50 (22.60) | 17.15 (23.61) | 16.83 (22.01) | 8.01 (19.68)
  Change at Week 12: Vitality: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 253 | 255 | 253 | 255
  Change at Week 12: Vitality | 5.68 (17.68) | 5.14 (17.69) | 6.47 (17.84) | 6.12 (18.16) | 3.97 (15.62) | 7.41 (17.89) | 4.35 (17.88) | 6.32 (17.13) | 6.47 (17.88) | 2.43 (15.51)
  Change at Week 12: Social function: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 255
  Change at Week 12: Social function | 5.90 (24.79) | 5.25 (23.40) | 5.36 (23.74) | 7.76 (23.66) | 7.41 (24.36) | 10.19 (25.95) | 5.36 (25.97) | 8.14 (24.30) | 8.94 (23.90) | 3.33 (23.87)
  Change at Week 12: Role emotional: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 12: Role emotional | 5.08 (26.90) | 5.50 (25.83) | 4.91 (25.97) | 4.47 (24.64) | 0.92 (23.38) | 8.23 (28.14) | 3.64 (28.43) | 8.63 (26.82) | 6.82 (26.37) | 4.13 (24.69)
  Change at Week 12: Mental health: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 253 | 255 | 253 | 255
  Change at Week 12: Mental health | 2.85 (17.25) | 3.28 (15.58) | 0.96 (16.77) | 3.04 (15.36) | 1.57 (15.44) | 3.00 (15.55) | 0.36 (16.85) | 3.78 (17.45) | 3.17 (17.39) | 0.67 (15.99)
  Change at Week 24: General health: number analyzed (Participants) | 284 | 288 | 280 | 285 | 279 | 254 | 254 | 255 | 253 | 255
  Change at Week 24: General health | 3.08 (13.39) | 2.95 (15.61) | 3.77 (14.43) | 4.54 (14.38) | 2.90 (14.43) | 4.07 (15.59) | 4.25 (16.34) | 3.46 (14.82) | 4.28 (15.77) | 3.90 (15.80)
  Change at Week 24: Physical function: number analyzed (Participants) | 282 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 24: Physical function | 10.52 (21.56) | 9.50 (22.90) | 9.83 (22.63) | 12.30 (24.18) | 5.75 (19.12) | 10.40 (22.45) | 9.33 (19.85) | 11.83 (23.45) | 12.00 (23.60) | 8.00 (18.72)
  Change at Week 24: Role physical: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 24: Role physical | 9.40 (25.04) | 7.42 (26.32) | 9.58 (25.13) | 11.54 (25.10) | 7.28 (22.16) | 10.24 (23.60) | 10.46 (25.88) | 10.93 (25.86) | 10.50 (23.87) | 7.70 (20.85)
  Change at Week 24: Bodily pain: number analyzed (Participants) | 284 | 287 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 255
  Change at Week 24: Bodily pain | 10.73 (21.66) | 9.63 (22.77) | 10.41 (21.52) | 13.04 (21.24) | 8.87 (19.60) | 10.69 (21.07) | 10.22 (23.32) | 14.02 (23.34) | 13.47 (21.19) | 8.72 (19.45)
  Change at Week 24: Vitality: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 253 | 255 | 253 | 255
  Change at Week 24: Vitality | 5.94 (16.70) | 3.93 (18.24) | 3.77 (16.18) | 4.52 (16.59) | 1.90 (14.77) | 5.71 (17.61) | 4.00 (18.26) | 2.84 (17.03) | 4.15 (16.64) | 2.87 (16.25)
  Change at Week 24: Social function: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 255
  Change at Week 24: Social function | 4.01 (25.13) | 3.21 (26.84) | 3.21 (22.32) | 6.14 (22.56) | 6.16 (23.26) | 7.63 (23.13) | 6.25 (25.58) | 7.06 (25.35) | 5.78 (22.67) | 4.07 (21.74)
  Change at Week 24: Role emotional: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 24: Role emotional | 3.35 (23.83) | 0.58 (25.64) | 2.38 (22.42) | 2.16 (22.64) | 2.92 (22.96) | 5.81 (26.42) | 4.95 (25.97) | 6.47 (24.20) | 3.39 (24.12) | 2.23 (23.18)
  Change at Week 24: Mental health: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 253 | 255 | 253 | 255
  Change at Week 24: Mental health | 2.31 (17.07) | 1.48 (16.93) | 0.95 (15.78) | 2.26 (15.92) | 1.52 (14.67) | 1.33 (14.50) | 0.42 (15.32) | 0.94 (15.01) | 0.87 (16.48) | 0.00 (16.15)

27. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) at Weeks 12, 24, 40 and 56: Last Observation Carried Forward (LOCF)
Description: as for outcome 26
Time Frame: Baseline, Weeks 12, 24, 40, and 56
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (either tanezumab or matching placebo). Missing values were imputed using LOCF. 'Number analyzed' signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
units on a scale
  Change at Week 12: General health: number analyzed (Participants) | 284 | 288 | 280 | 285 | 279 | 254 | 254 | 255 | 253 | 255
  Change at Week 12: General health | 3.29 (14.32) | 4.66 (15.19) | 3.66 (15.27) | 5.14 (15.96) | 3.88 (15.25) | 5.46 (14.25) | 3.37 (15.13) | 5.18 (13.96) | 5.66 (16.53) | 4.68 (16.00)
  Change at Week 12: Physical function: number analyzed (Participants) | 282 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 12: Physical function | 32.82 (19.12) | 32.74 (21.34) | 34.79 (20.63) | 33.88 (18.66) | 35.46 (19.94) | 12.70 (22.24) | 9.05 (22.01) | 13.84 (24.37) | 12.99 (24.30) | 7.48 (18.88)
  Change at Week 12: Role physical: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 12: Role physical | 43.29 (25.54) | 43.88 (23.81) | 44.58 (23.90) | 44.69 (23.60) | 46.09 (24.57) | 13.36 (25.67) | 10.04 (26.31) | 15.51 (26.62) | 13.71 (25.39) | 7.58 (23.58)
  Change at Week 12: Bodily pain: number analyzed (Participants) | 284 | 287 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 255
  Change at Week 12: Bodily pain | 11.44 (21.66) | 13.08 (21.93) | 14.41 (22.41) | 16.53 (22.55) | 7.83 (19.22) | 16.74 (21.52) | 12.50 (22.60) | 17.15 (23.61) | 16.83 (22.01) | 8.01 (19.68)
  Change at Week 12: Vitality: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 253 | 255 | 253 | 255
  Change at Week 12: Vitality | 5.68 (17.68) | 5.14 (17.69) | 6.47 (17.84) | 6.12 (18.16) | 3.97 (15.62) | 7.41 (17.89) | 4.35 (17.88) | 6.32 (17.13) | 6.47 (17.88) | 2.43 (15.51)
  Change at Week 12: Social function: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 255
  Change at Week 12: Social function | 5.90 (24.79) | 5.25 (23.40) | 5.36 (23.74) | 7.76 (23.66) | 7.41 (24.36) | 10.19 (25.95) | 5.36 (25.97) | 8.14 (24.30) | 8.94 (23.90) | 3.33 (23.87)
  Change at Week 12: Role emotional: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 12: Role emotional | 5.08 (26.90) | 5.50 (25.83) | 4.91 (25.97) | 4.47 (24.64) | 0.92 (23.38) | 8.23 (28.14) | 3.64 (28.43) | 8.63 (26.82) | 6.82 (26.37) | 4.13 (24.69)
  Change at Week 12: Mental health: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 253 | 255 | 253 | 255
  Change at Week 12: Mental health | 2.85 (17.25) | 3.28 (15.58) | 0.96 (16.77) | 3.04 (15.36) | 1.57 (15.44) | 3.00 (15.55) | 0.36 (16.85) | 3.78 (17.45) | 3.17 (17.39) | 0.67 (15.99)
  Change at Week 24: General health: number analyzed (Participants) | 284 | 288 | 280 | 285 | 279 | 254 | 254 | 255 | 253 | 255
  Change at Week 24: General health | 3.95 (14.92) | 3.18 (16.54) | 3.93 (16.09) | 4.66 (15.46) | 3.77 (16.48) | 4.42 (15.98) | 4.59 (17.08) | 3.72 (15.54) | 4.62 (16.60) | 4.45 (16.75)
  Change at Week 24: Physical function: number analyzed (Participants) | 282 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 24: Physical function | 11.70 (22.93) | 11.35 (24.40) | 10.85 (24.77) | 13.73 (24.60) | 6.43 (21.08) | 11.23 (23.56) | 10.00 (21.47) | 12.92 (24.02) | 12.91 (24.35) | 8.41 (20.14)
  Change at Week 24: Role physical: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 24: Role physical | 11.14 (26.65) | 9.53 (28.68) | 10.71 (26.82) | 13.03 (26.16) | 7.97 (24.14) | 11.74 (24.66) | 11.84 (27.30) | 11.84 (27.49) | 12.45 (24.96) | 8.27 (22.89)
  Change at Week 24: Bodily pain: number analyzed (Participants) | 284 | 287 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 255
  Change at Week 24: Bodily pain | 12.95 (22.92) | 11.63 (24.07) | 11.75 (23.05) | 14.73 (21.67) | 9.19 (21.10) | 12.24 (21.85) | 12.00 (24.21) | 15.22 (24.37) | 14.83 (21.76) | 9.09 (20.09)
  Change at Week 24: Vitality: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 253 | 255 | 253 | 255
  Change at Week 24: Vitality | 7.17 (18.11) | 4.34 (18.95) | 4.42 (18.09) | 5.48 (18.13) | 2.57 (16.19) | 5.95 (18.32) | 4.87 (19.75) | 3.09 (17.82) | 4.50 (18.07) | 2.40 (17.96)
  Change at Week 24: Social function: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 255
  Change at Week 24: Social function | 5.19 (27.51) | 3.56 (28.56) | 2.81 (24.00) | 7.11 (23.55) | 7.32 (25.07) | 8.51 (24.64) | 7.09 (27.25) | 7.35 (26.34) | 6.57 (24.56) | 3.97 (24.47)
  Change at Week 24: Role emotional: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 24: Role emotional | 5.22 (26.39) | 1.56 (27.95) | 3.63 (24.03) | 3.10 (24.18) | 2.59 (25.68) | 6.73 (28.21) | 5.09 (28.41) | 6.83 (25.37) | 4.58 (26.67) | 2.76 (25.33)
  Change at Week 24: Mental health: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 253 | 255 | 253 | 255
  Change at Week 24: Mental health | 2.90 (18.22) | 1.51 (17.97) | 0.45 (17.97) | 2.65 (16.96) | 1.38 (16.71) | 1.37 (15.33) | 0.30 (16.71) | 1.39 (15.75) | 1.06 (18.13) | 0.20 (18.25)
  Change at Week 40: General health: number analyzed (Participants) | 284 | 288 | 280 | 285 | 279 | 254 | 254 | 255 | 253 | 255
  Change at Week 40: General health | 3.40 (15.54) | 2.45 (16.52) | 2.83 (16.57) | 3.87 (16.28) | 3.47 (16.07) | 3.74 (15.63) | 3.31 (16.35) | 3.20 (15.93) | 3.45 (16.95) | 4.09 (16.42)
  Change at Week 40: Physical function: number analyzed (Participants) | 282 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 40: Physical function | 10.00 (22.96) | 10.23 (24.17) | 10.49 (24.89) | 11.96 (25.30) | 6.23 (19.34) | 9.91 (22.72) | 8.74 (21.92) | 12.32 (24.17) | 11.78 (25.11) | 7.24 (20.71)
  Change at Week 40: Role physical: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 40: Role physical | 9.64 (26.06) | 8.79 (27.05) | 10.98 (26.99) | 10.00 (26.77) | 7.01 (23.65) | 11.32 (25.78) | 10.53 (26.49) | 12.38 (28.71) | 12.13 (24.46) | 7.58 (23.43)
  Change at Week 40: Bodily pain: number analyzed (Participants) | 284 | 287 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 255
  Change at Week 40: Bodily pain | 11.27 (23.45) | 10.73 (23.77) | 10.79 (23.42) | 12.42 (21.98) | 7.11 (19.38) | 11.45 (21.91) | 10.87 (23.44) | 13.96 (23.88) | 13.28 (21.69) | 8.17 (19.11)
  Change at Week 40: Vitality: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 253 | 255 | 253 | 255
  Change at Week 40: Vitality | 5.92 (17.95) | 3.30 (19.26) | 4.42 (18.61) | 4.45 (18.58) | 2.32 (17.09) | 5.29 (18.95) | 4.40 (19.47) | 3.24 (17.68) | 4.17 (16.83) | 2.67 (18.06)
  Social function at Week 40: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 255
  Social function at Week 40 | 4.05 (27.36) | 3.21 (28.09) | 2.19 (23.43) | 4.56 (25.07) | 7.23 (24.46) | 7.43 (25.14) | 6.20 (27.82) | 6.03 (25.56) | 6.23 (25.29) | 2.65 (25.28)
  Change at Week 40: Role emotional: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 40: Role emotional | 4.08 (27.04) | 1.91 (26.29) | 2.80 (24.30) | 0.76 (25.47) | 1.61 (26.00) | 6.69 (27.88) | 2.99 (30.27) | 5.98 (27.72) | 5.47 (26.06) | 3.41 (27.05)
  Change at Week 40: Mental health: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 253 | 255 | 253 | 255
  Change at Week 40: Mental health | 2.16 (19.27) | 1.41 (17.56) | 0.25 (18.14) | 1.76 (16.34) | 0.49 (16.26) | 1.22 (16.42) | 0.26 (18.11) | 1.22 (15.48) | 1.11 (17.41) | 0.82 (18.76)
  Change at Week 56: General health: number analyzed (Participants) | 284 | 288 | 280 | 285 | 279 | 254 | 254 | 255 | 253 | 255
  Change at Week 56: General health | 3.12 (15.53) | 2.31 (16.84) | 2.59 (16.83) | 3.69 (16.54) | 3.33 (16.26) | 3.75 (14.82) | 3.41 (16.14) | 3.10 (15.85) | 3.75 (16.71) | 3.99 (16.87)
  Change at Week 56: Physical function: number analyzed (Participants) | 282 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 56: Physical function | 9.95 (22.78) | 9.19 (24.31) | 10.19 (24.94) | 11.15 (25.00) | 5.95 (19.75) | 10.12 (22.91) | 8.25 (21.73) | 12.07 (24.08) | 11.48 (24.80) | 6.91 (20.39)
  Change at Week 56: Role physical: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 56: Role physical | 9.13 (26.00) | 8.01 (27.09) | 10.49 (26.86) | 9.01 (26.81) | 7.19 (23.29) | 11.20 (25.54) | 10.46 (26.83) | 11.96 (28.82) | 12.06 (24.38) | 7.28 (23.78)
  Change at Week 56: Bodily pain: number analyzed (Participants) | 284 | 287 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 255
  Change at Week 56: Bodily pain | 11.58 (23.00) | 10.21 (24.18) | 10.38 (23.28) | 11.92 (22.25) | 7.47 (19.17) | 11.52 (21.79) | 10.32 (23.48) | 13.53 (24.12) | 13.36 (21.53) | 8.69 (19.35)
  Change at Week 56: Vitality: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 253 | 255 | 253 | 255
  Change at Week 56: Vitality | 5.70 (18.10) | 3.10 (19.16) | 4.17 (18.73) | 3.82 (18.90) | 2.68 (16.53) | 4.82 (18.47) | 4.47 (19.74) | 3.41 (17.70) | 4.15 (16.66) | 2.08 (17.89)
  Change at Week 56: Social function: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 255
  Change at Week 56: Social function | 4.53 (26.95) | 2.95 (28.04) | 1.65 (23.40) | 3.99 (24.98) | 7.23 (23.97) | 7.73 (25.15) | 6.10 (27.69) | 6.23 (26.15) | 6.67 (24.59) | 2.84 (25.01)
  Change at Week 56: Role emotional: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 254 | 255 | 253 | 254
  Change at Week 56: Role emotional | 4.23 (28.30) | 1.53 (26.76) | 1.99 (24.59) | 0.47 (25.50) | 1.67 (25.90) | 6.10 (28.74) | 3.25 (30.06) | 6.11 (28.11) | 5.07 (26.11) | 3.51 (27.41)
  Change at Week 56: Mental health: number analyzed (Participants) | 284 | 288 | 280 | 285 | 280 | 254 | 253 | 255 | 253 | 255
  Change at Week 56: Mental health | 2.28 (19.24) | 1.42 (17.72) | -0.11 (18.49) | 1.53 (16.55) | 0.41 (16.13) | 1.10 (16.47) | 0.18 (18.05) | 1.47 (15.63) | 1.25 (17.22) | 0.96 (18.44)

28. Secondary Outcome: Number of Participants Who Had Discontinued Study Due to Lack of Efficacy
Time Frame: Baseline up to Week 56
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (tanezumab or matching placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
Participants | 23 | 23 | 22 | 15 | 40 | 19 | 21 | 15 | 18 | 38

29. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Time to discontinuation due to lack of efficacy was defined as the time interval from the date of study drug administration up to the date of discontinuation of participant from study due to lack of efficacy.
Time Frame: Baseline up to Week 56
Population: as for outcome 28
Measure: Mean (Standard Error); unit: days
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
days | 319.87 (3.74) | 331.69 (3.65) | 394.80 (5.08) | 271.89 (2.66) | 306.11 (4.94) | 329.79 (3.68) | 314.16 (4.15) | 334.84 (3.08) | 324.25 (3.32) | 303.08 (5.10)

30. Secondary Outcome: Change From Baseline in Percent Work Time Missed Due to Osteoarthritis at Week 24 Assessed Using Work Productivity and Activity Impairment Questionnaire- Specific Health Problem (WPAI-SHP): Baseline Observation Carried Forward (BOCF)
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which a specified health problem affected work productivity and regular activities over the past 7 days. The questions (Q) are: Q1 = currently employed. Q2 = hours missed due to health problems. Q3 = hours missed other reasons. Q4 = hours actually worked. Q5 = degree health affected productivity while working (0-10 scale). Q6 = degree health affected regular activities (0-10 scale). Subscale scores are calculated: Percent work time missed due to health problem: Q2/(Q2+Q4). The computed percentage range for each sub-scale is 0-100, where higher numbers indicate greater impairment and less productivity.
Time Frame: Baseline, Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (tanezumab or matching placebo). Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: change in percent work time missed
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 101 | 103 | 99 | 121 | 114 | 76 | 77 | 92 | 84 | 90
change in percent work time missed | -0.88 (11.54) | 0.04 (8.16) | 0.63 (6.23) | -0.77 (15.75) | 1.11 (12.55) | -2.85 (10.19) | -0.42 (12.87) | 1.51 (11.21) | -1.64 (9.60) | -0.61 (8.36)

31. Secondary Outcome: Change From Baseline in Percent Work Time Missed Due to Osteoarthritis at Week 24 and 56 Assessed Using Work Productivity and Activity Impairment Questionnaire- Specific Health Problem (WPAI-SHP): Last Observation Carried Forward (LOCF)
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which a specified health problem affected work productivity and regular activities over the past 7 days. The questions are: Q1 = currently employed. Q2 = hours missed due to health problems. Q3 = hours missed other reasons. Q4 = hours actually worked. Q5 = degree health affected productivity while working (0-10 scale). Q6 = degree health affected regular activities (0-10 scale). Subscale scores are calculated: Percent work time missed due to health problem: Q2/(Q2+Q4). The computed percentage range for each sub-scale is 0-100, where higher numbers indicate greater impairment and less productivity.
Time Frame: Baseline, Week 24 and 56
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: change in percent work time missed
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 101 | 103 | 99 | 121 | 114 | 76 | 77 | 92 | 84 | 90
change in percent work time missed
  Change at Week 24 | -0.88 (11.54) | 0.04 (8.16) | 0.63 (6.23) | 0.77 (15.75) | 1.11 (12.55) | -2.85 (10.19) | -0.42 (12.87) | 1.51 (11.21) | -1.64 (9.60) | -0.61 (8.36)
  Change at Week 56 | -1.10 (11.30) | -0.39 (9.29) | 1.08 (7.57) | -0.41 (16.46) | 2.26 (13.76) | -3.06 (9.98) | -0.46 (12.88) | 1.51 (11.21) | -1.64 (9.60) | -0.82 (7.94)

32. Secondary Outcome: Change From Baseline in Percent Impairment While Working Due to Osteoarthritis at Week 24 Assessed Using Work Productivity and Activity Impairment Questionnaire- Specific Health Problem (WPAI-SHP): Baseline Observation Carried Forward (BOCF)
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which a specified health problem affected work productivity and regular activities over the past 7 days. The questions are: Q1 = currently employed. Q2 = hours missed due to health problems. Q3 = hours missed other reasons. Q4 = hours actually worked. Q5 = degree health affected productivity while working (0-10 scale). Q6 = degree health affected regular activities (0-10 scale). Subscale scores are calculated: Percent impairment while working due to health problem: Q5/10. The computed percentage range for each sub-scale is 0-100, where higher numbers indicate greater impairment and less productivity.
Time Frame: Baseline, Week 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: change in percent impairment
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 100 | 101 | 98 | 120 | 113 | 73 | 73 | 89 | 80 | 86
change in percent impairment | -11.90 (22.32) | -11.68 (24.74) | -5.51 (26.33) | -13.00 (27.34) | -7.35 (29.03) | -17.81 (22.00) | -13.01 (25.91) | -9.33 (22.40) | -9.63 (23.68) | -5.81 (22.62)

33. Secondary Outcome: Change From Baseline in Percent Impairment While Working Due to Osteoarthritis at Week 24 and 56 Assessed Using Work Productivity and Activity Impairment Questionnaire- Specific Health Problem (WPAI-SHP): Last Observation Carried Forward (LOCF)
Description: as for outcome 32
Time Frame: Baseline, Weeks 24 and 56
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: change in percent impairment
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 100 | 101 | 98 | 120 | 113 | 73 | 73 | 89 | 80 | 86
change in percent impairment
  Change at Week 24 | -11.90 (22.32) | -11.68 (24.74) | -5.51 (26.33) | -13.00 (27.34) | -7.35 (29.03) | -17.81 (22.00) | -13.01 (25.91) | -9.33 (22.40) | -9.63 (23.68) | -5.81 (22.62)
  Change at Week 56 | -10.30 (23.11) | -11.88 (24.85) | -4.08 (25.92) | -11.33 (27.19) | -5.31 (28.51) | -16.99 (22.09) | -12.88 (27.00) | -8.09 (24.58) | -4.25 (42.03) | -5.93 (22.30)

34. Secondary Outcome: Change From Baseline in the Percent Overall Work Impairment Due to Osteoarthritis at Week 24 Assessed Using Work Productivity and Activity Impairment Questionnaire- Specific Health Problem (WPAI-SHP): BOCF
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which a specified health problem affected work productivity and regular activities over the past 7 days. The questions are: Q1 = currently employed. Q2 = hours missed due to health problems. Q3 = hours missed other reasons. Q4 = hours actually worked. Q5 = degree health affected productivity while working (0-10 scale). Q6 = degree health affected regular activities (0-10 scale). Subscale scores are calculated: Percent overall work impairment due to health problem: Q2/(Q2+Q4)+[(1-Q2/(Q2+Q4))*(Q5/10)]. The computed percentage range for each sub-scale is 0-100, where higher numbers indicate greater impairment and less productivity.
Time Frame: Baseline, Week 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: change in percent work impairment
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 101 | 103 | 99 | 121 | 114 | 77 | 254 | 92 | 84 | 90
change in percent work impairment | -5.40 (31.08) | -1.46 (24.95) | -0.75 (18.60) | -1.35 (29.85) | 2.09 (28.55) | -10.17 (26.46) | -0.22 (22.51) | 1.25 (26.81) | -4.30 (24.16) | -2.29 (23.87)

35. Secondary Outcome: Change From Baseline in the Percent Overall Work Impairment Due to Osteoarthritis at Week 24 and 56 Assessed Using Work Productivity and Activity Impairment Questionnaire- Specific Health Problem (WPAI-SHP): LOCF
Description: as for outcome 34
Time Frame: Baseline, Weeks 24 and 56
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: change in percent work impairment
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 101 | 103 | 99 | 121 | 114 | 76 | 77 | 92 | 84 | 90
change in percent work impairment
  Change at Week 24 | -5.40 (31.08) | -1.46 (24.95) | -0.75 (18.60) | -1.35 (29.85) | 2.09 (28.55) | -10.17 (26.46) | -0.22 (22.51) | 1.25 (26.81) | -4.30 (24.16) | -2.29 (23.87)
  Change at Week 56 | -6.08 (30.20) | -1.88 (26.61) | 0.77 (22.05) | -0.85 (31.85) | 4.11 (27.38) | -10.32 (26.52) | -1.01 (23.22) | 1.25 (26.81) | -4.30 (24.16) | -3.02 (21.60)

36. Secondary Outcome: Change From Baseline in the Percent Activity Impairment Due to Osteoarthritis at Week 24 Assessed Using Work Productivity and Activity Impairment Questionnaire - Specific Health Problem (WPAI-SHP): Baseline Observation Carried Forward (BOCF)
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which a specified health problem affected work productivity and regular activities over the past 7 days. The questions are: Q1 = currently employed. Q2 = hours missed due to health problems. Q3 = hours missed other reasons. Q4 = hours actually worked. Q5 = degree health affected productivity while working (0-10 scale). Q6 = degree health affected regular activities (0-10 scale). Subscale scores are calculated: Percent activity impairment due to health problem: Q6/10. The computed percentage range for each sub-scale is 0-100, where higher numbers indicate greater impairment and less productivity.
Time Frame: Baseline, Week 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: change in percent activity impairment
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 283 | 287 | 279 | 284 | 280 | 254 | 250 | 255 | 249 | 253
change in percent activity impairment | -12.30 (25.61) | -15.51 (26.17) | -13.55 (26.42) | -14.96 (26.74) | -10.00 (25.92) | -17.24 (25.11) | -17.84 (25.81) | -18.04 (25.47) | -17.31 (26.28) | -11.90 (26.06)

37. Secondary Outcome: Change From Baseline in the Percent Activity Impairment Due to Osteoarthritis at Week 24 and 56 Assessed Using Work Productivity and Activity Impairment Questionnaire - Specific Health Problem (WPAI-SHP): Last Observation Carried Forward (LOCF)
Description: as for outcome 36
Time Frame: Baseline, Weeks 24, and 56
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: change in percent activity impairment
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 283 | 287 | 279 | 284 | 280 | 254 | 250 | 255 | 249 | 253
change in percent activity impairment
  Change at Week 24 | -12.30 (25.61) | -15.51 (26.17) | -13.55 (26.42) | -14.96 (26.74) | -10.00 (25.92) | -17.24 (25.11) | -17.84 (25.81) | -18.04 (25.47) | -17.31 (26.28) | -11.90 (26.06)
  Change at Week 56 | -12.12 (25.37) | -14.77 (26.72) | -12.19 (27.03) | -13.20 (26.58) | -9.32 (24.93) | -15.39 (23.53) | -15.76 (27.09) | -18.04 (25.93) | -15.86 (26.91) | -11.19 (26.55)

38. Secondary Outcome: Percentage of Participants Who Used Rescue Medication: Observed Data
Description: In case of inadequate pain relief for osteoarthritis, acetaminophen up to 4000 mg per day for maximum of 3 days within a week could be taken as rescue medication. Percentage of participants with any use of rescue medication during each study interval were summarized.
Time Frame: Weeks 1-2, 3-4, 5-8, 9-12, 13-16, 17-24, 25-32, 33-40, 41-48 and 49-56
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (tanezumab or matching placebo). 'Number analyzed' signifies participants evaluable at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
percentage of participants
  Weeks 1-2: number analyzed (Participants) | 266 | 275 | 264 | 267 | 273 | 241 | 240 | 241 | 240 | 250
  Weeks 1-2 | 60.5 | 59.3 | 57.6 | 62.9 | 61.9 | 69.7 | 64.2 | 60.2 | 62.5 | 63.2
  Weeks 3-4: number analyzed (Participants) | 256 | 262 | 256 | 254 | 260 | 244 | 231 | 241 | 234 | 247
  Weeks 3-4 | 63.3 | 61.8 | 55.1 | 60.6 | 62.3 | 68.4 | 64.9 | 59.3 | 60.3 | 66.0
  Weeks 5-8: number analyzed (Participants) | 251 | 249 | 243 | 240 | 247 | 228 | 224 | 232 | 230 | 234
  Weeks 5-8 | 67.7 | 64.7 | 55.1 | 57.9 | 68.8 | 68.0 | 61.2 | 62.5 | 63.9 | 66.7
  Weeks 9-12: number analyzed (Participants) | 242 | 245 | 229 | 236 | 230 | 221 | 220 | 229 | 224 | 223
  Weeks 9-12 | 67.8 | 65.3 | 56.3 | 61.4 | 64.8 | 62.9 | 64.5 | 60.3 | 57.1 | 65.9
  Weeks 13-16: number analyzed (Participants) | 231 | 234 | 224 | 225 | 216 | 215 | 204 | 220 | 218 | 208
  Weeks 13-16 | 66.7 | 63.7 | 62.1 | 57.8 | 68.1 | 64.2 | 61.3 | 62.3 | 57.8 | 68.8
  Weeks 17-24: number analyzed (Participants) | 206 | 209 | 207 | 206 | 197 | 200 | 189 | 207 | 198 | 196
  Weeks 17-24 | 68.9 | 67.0 | 64.7 | 66.0 | 76.6 | 67.0 | 65.1 | 59.4 | 66.2 | 66.3
  Weeks 25-32: number analyzed (Participants) | 162 | 153 | 159 | 156 | 151 | 158 | 151 | 156 | 148 | 156
  Weeks 25-32 | 66.0 | 67.3 | 59.1 | 59.6 | 69.5 | 66.5 | 70.2 | 63.5 | 66.2 | 71.2
  Weeks 33-40: number analyzed (Participants) | 90 | 82 | 91 | 76 | 76 | 80 | 73 | 71 | 76 | 86
  Weeks 33-40 | 64.4 | 69.5 | 58.2 | 61.8 | 73.7 | 63.8 | 71.2 | 64.8 | 61.8 | 61.6
  Weeks 41-48: number analyzed (Participants) | 51 | 40 | 49 | 46 | 47 | 39 | 41 | 30 | 40 | 43
  Weeks 41-48 | 66.7 | 62.5 | 59.2 | 60.9 | 66.0 | 64.1 | 70.7 | 63.3 | 52.5 | 65.1
  Weeks 49-56: number analyzed (Participants) | 91 | 90 | 89 | 89 | 87 | 79 | 85 | 76 | 87 | 89
  Weeks 49-56 | 69.2 | 71.1 | 62.9 | 74.2 | 78.2 | 75.9 | 74.1 | 72.4 | 79.3 | 77.5

39. Secondary Outcome: Percentage of Participants Who Used Rescue Medication: Last Observation Carried Forward (LOCF)
Description: as for outcome 38
Time Frame: Weeks 1-2, 3-4, 5-8, 9-12, 13-16, 17-24, 25-32, 33-40, 41-48 and 49-56
Population: as for outcome 38
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
percentage of participants
  Weeks 1-2: number analyzed (Participants) | 278 | 286 | 274 | 284 | 281 | 253 | 250 | 253 | 249 | 255
  Weeks 1-2 | 60.4 | 59.4 | 56.9 | 63.0 | 63.0 | 70.0 | 64.4 | 60.5 | 62.7 | 63.1
  Weeks 3-4: number analyzed (Participants) | 281 | 287 | 278 | 285 | 281 | 255 | 250 | 255 | 251 | 256
  Weeks 3-4 | 63.0 | 61.7 | 54.7 | 60.7 | 63.0 | 69.4 | 64.4 | 59.2 | 61.1 | 66.0
  Weeks 5-8: number analyzed (Participants) | 284 | 287 | 280 | 287 | 281 | 255 | 251 | 255 | 252 | 256
  Weeks 5-8 | 66.5 | 63.8 | 55.0 | 58.9 | 69.8 | 69.8 | 61.0 | 62.4 | 64.3 | 67.6
  Weeks 9-12: number analyzed (Participants) | 284 | 288 | 280 | 287 | 281 | 255 | 252 | 256 | 253 | 256
  Weeks 9-12 | 65.8 | 64.2 | 55.4 | 60.3 | 66.2 | 65.1 | 63.9 | 60.5 | 59.3 | 68.4
  Weeks 13-16: number analyzed (Participants) | 285 | 288 | 280 | 287 | 281 | 255 | 252 | 256 | 253 | 256
  Weeks 13-16 | 65.3 | 62.5 | 60.0 | 57.8 | 69.4 | 67.5 | 62.3 | 62.5 | 59.7 | 70.7
  Weeks 17-24: number analyzed (Participants) | 285 | 288 | 280 | 287 | 281 | 255 | 252 | 256 | 253 | 256
  Weeks 17-24 | 68.1 | 64.6 | 63.2 | 64.5 | 75.8 | 69.8 | 64.3 | 60.9 | 65.6 | 69.1
  Weeks 25-32: number analyzed (Participants) | 285 | 288 | 280 | 287 | 281 | 255 | 252 | 256 | 253 | 256
  Weeks 25-32 | 66.7 | 64.9 | 60.0 | 63.1 | 70.8 | 71.8 | 67.5 | 63.7 | 66.4 | 74.2
  Weeks 33-40: number analyzed (Participants) | 285 | 288 | 280 | 287 | 281 | 255 | 252 | 256 | 253 | 256
  Weeks 33-40 | 68.1 | 66.3 | 61.8 | 64.1 | 71.9 | 71.4 | 67.5 | 62.9 | 65.2 | 71.5
  Weeks 41-48: number analyzed (Participants) | 285 | 288 | 280 | 287 | 281 | 255 | 252 | 256 | 254 | 256
  Weeks 41-48 | 69.5 | 66.0 | 63.9 | 64.8 | 71.5 | 71.4 | 67.9 | 63.7 | 65.0 | 72.3
  Weeks 49-56: number analyzed (Participants) | 285 | 288 | 280 | 287 | 281 | 256 | 253 | 256 | 254 | 256
  Weeks 49-56 | 71.2 | 69.1 | 65.4 | 67.6 | 72.6 | 71.5 | 70.0 | 66.8 | 68.1 | 71.5

40. Secondary Outcome: Amount of Rescue Medication Used
Description: In case of inadequate pain relief for osteoarthritis, acetaminophen up to 4000 mg per day up to 3 days in a week could be taken as rescue medication. The total dosage of acetaminophen in mg used during the specified time intervals were summarized.
Time Frame: Weeks 1-2, 3-4, 5-8, 9-12, 13-16, 17-24, 25-32, 33-40, 41-48, and 49-56
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: milligram (mg)
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
milligram (mg)
  Weeks 1-2: number analyzed (Participants) | 278 | 286 | 274 | 284 | 281 | 253 | 250 | 253 | 249 | 255
  Weeks 1-2 | 3144.66 (6878.90) | 3365.46 (8829.47) | 2739.96 (7060.72) | 3524.27 (5665.78) | 3543.99 (5541.14) | 3132.30 (4047.15) | 3834.79 (7152.17) | 2910.68 (4285.74) | 3250.69 (4846.02) | 3455.85 (8154.84)
  Weeks 3-4: number analyzed (Participants) | 281 | 287 | 278 | 285 | 281 | 255 | 250 | 255 | 252 | 256
  Weeks 3-4 | 3411.93 (6929.86) | 3582.77 (8814.22) | 2660.11 (6782.71) | 3066.65 (5206.51) | 3415.52 (5260.63) | 3255.16 (4142.25) | 3769.17 (7131.76) | 2672.18 (4108.60) | 3011.67 (4412.94) | 3281.23 (6981.13)
  Weeks 5-8: number analyzed (Participants) | 284 | 287 | 280 | 287 | 281 | 255 | 251 | 255 | 252 | 256
  Weeks 5-8 | 2846.58 (6532.40) | 2875.55 (8372.63) | 2131.45 (6429.73) | 2396.99 (4684.26) | 2991.01 (4634.26) | 2571.99 (3240.96) | 2969.34 (6656.34) | 2140.44 (3585.06) | 2223.15 (3624.98) | 3182.45 (6991.76)
  Weeks 9-12: number analyzed (Participants) | 284 | 288 | 280 | 287 | 281 | 255 | 252 | 256 | 253 | 256
  Weeks 9-12 | 2863.10 (6547.23) | 2955.84 (8403.06) | 2291.41 (6478.22) | 2415.93 (4630.96) | 2919.20 (4643.38) | 2380.78 (3162.61) | 3008.85 (6675.65) | 2166.23 (3632.39) | 2266.13 (3753.34) | 3067.56 (6962.68)
  Weeks 13-16: number analyzed (Participants) | 285 | 288 | 280 | 287 | 281 | 255 | 252 | 256 | 253 | 256
  Weeks 13-16 | 2993.63 (6587.61) | 2912.14 (8426.72) | 2562.94 (6525.59) | 2551.21 (4793.92) | 2920.39 (4659.70) | 2450.55 (3280.41) | 2938.95 (6667.26) | 2244.74 (3642.93) | 2486.23 (3933.41) | 3269.78 (7040.71)
  Weeks 17-24: number analyzed (Participants) | 285 | 288 | 280 | 287 | 281 | 255 | 252 | 256 | 253 | 256
  Weeks 17-24 | 2733.43 (6432.63) | 2778.55 (8311.86) | 2525.71 (6490.27) | 2261.93 (4517.29) | 2759.90 (4426.38) | 2261.84 (2980.00) | 2725.86 (6619.25) | 2235.23 (3702.39) | 2370.30 (3599.96) | 2816.00 (6854.35)
  Weeks 25-32: number analyzed (Participants) | 285 | 288 | 280 | 287 | 281 | 255 | 252 | 256 | 253 | 256
  Weeks 25-32 | 2823.39 (6441.86) | 2824.83 (8313.77) | 2548.20 (6512.08) | 2289.28 (4563.36) | 2792.04 (4555.75) | 2383.27 (3102.23) | 2927.44 (6606.26) | 2432.81 (3783.30) | 2723.26 (3891.04) | 3126.26 (6906.75)
  Weeks 33-40: number analyzed (Participants) | 285 | 288 | 280 | 287 | 281 | 255 | 252 | 256 | 253 | 256
  Weeks 33-40 | 2810.18 (6445.83) | 2900.69 (8319.96) | 2608.91 (6529.78) | 2361.40 (4541.68) | 2755.66 (4503.88) | 2449.87 (3126.73) | 2976.37 (6607.95) | 2428.51 (3758.09) | 2682.35 (3925.96) | 3032.17 (6889.07)
  Weeks 41-48: number analyzed (Participants) | 285 | 288 | 280 | 287 | 281 | 255 | 252 | 256 | 254 | 256
  Weeks 41-48 | 2927.31 (6460.58) | 2906.70 (8324.75) | 2673.48 (6517.91) | 2373.66 (4547.39) | 2746.29 (4498.19) | 2521.27 (3163.27) | 3033.87 (6627.43) | 2408.58 (3706.60) | 2618.83 (3864.42) | 3101.63 (6912.29)
  Weeks 49-56: number analyzed (Participants) | 285 | 288 | 280 | 287 | 281 | 256 | 253 | 256 | 254 | 256
  Weeks 49-56 | 2979.89 (6413.29) | 2910.73 (6626.26) | 2938.47 (6717.61) | 2545.36 (4465.07) | 3106.46 (4908.02) | 2840.21 (3627.85) | 2770.28 (3810.98) | 2511.61 (3797.81) | 2842.74 (3642.86) | 3035.33 (4124.28)

41. Secondary Outcome: Change From Baseline in Medial Minimum Joint Space Width of the Index Knee at Week 56
Time Frame: Baseline, Week 56
Population: Analysis was performed on ITT analysis set. Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this outcome measure. Data was planned to be assessed and reported for combined population of naproxen and celecoxib cohort.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Groups:
- Tanezumab 5 mg (Naproxen or Celecoxib Exposure): Participants were administered with tanezumab 5 mg IV infusion, once every 8 weeks up to Week 48, beginning from Day 1 of Week 1. Additionally, participants received naproxen 500 mg/celecoxib 100 mg tablet orally twice daily on Days 1-7 followed by naproxen 500 mg/celecoxib 100 mg tablet orally once daily in the morning along with placebo matching to naproxen/celecoxib tablet once daily in the evening of Days 8-14. From Day 15, participants received placebo matched to naproxen 500 mg/celecoxib 100 mg tablet orally twice daily up to Week 48.
- Tanezumab 10 mg (Naproxen or Celecoxib Exposure): Participants were administered with tanezumab 10 mg IV infusion, once every 8 weeks up to Week 48, beginning from Day 1 of Week 1. Additionally, participants received naproxen 500 mg/celecoxib 100 mg tablet orally twice daily on Days 1-7 followed by naproxen 500 mg/celecoxib 100 mg tablet orally once daily in the morning along with placebo matching to naproxen/celecoxib tablet once daily in the evening of Days 8-14. From Day 15, participants received placebo matched to naproxen 500 mg/celecoxib 100 mg tablet orally twice daily up to Week 48.
- Tanezumab 5 mg + NSAID: Tanezumab 5 mg IV infusion, once every 8 weeks plus NSAID (naproxen 500 mg or celecoxib 100 mg) tablet orally twice daily up to Week 48.
- Tanezumab 10 mg + NSAID: Tanezumab 10 mg IV infusion, once every 8 weeks plus NSAID (naproxen 500 mg or celecoxib 100 mg) tablet orally twice daily up to Week 48.
- NSAID: Placebo matched to tanezumab infusion, IV once every 8 weeks plus NSAID (naproxen 500 mg or celecoxib 100 mg) tablet orally twice daily up to Week 48.
Arm/Group | Tanezumab 5 mg (Naproxen or Celecoxib Exposure) | Tanezumab 10 mg (Naproxen or Celecoxib Exposure) | Tanezumab 5 mg + NSAID | Tanezumab 10 mg + NSAID | NSAID
Number analyzed (Participants) | 448 | 449 | 446 | 452 | 446
millimeter (mm)
  Baseline: number analyzed (Participants) | 371 | 370 | 369 | 368 | 375
  Baseline | 2.769 (2.077) | 2.850 (2.077) | 3.005 (2.068) | 2.982 (2.106) | 3.022 (2.090)
  Change at Week 56: number analyzed (Participants) | 255 | 256 | 262 | 239 | 275
  Change at Week 56 | -0.189 (0.970) | -0.213 (1.069) | -0.162 (1.069) | -0.172 (1.096) | -0.041 (0.850)

42. Secondary Outcome: Change From Baseline in Minimum Joint Space Width of the Index Hip at Week 56
Time Frame: Baseline, Week 56
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Tanezumab 5 mg (Naproxen or Celecoxib Exposure) | Tanezumab 10 mg (Naproxen or Celecoxib Exposure) | Tanezumab 5 mg + NSAID | Tanezumab 10 mg + NSAID | NSAID
Number analyzed (Participants) | 92 | 93 | 90 | 90 | 93
millimeter
  Baseline: number analyzed (Participants) | 91 | 92 | 87 | 87 | 90
  Baseline | 2.447 (1.364) | 2.372 (1.433) | 2.346 (1.424) | 2.195 (1.561) | 2.724 (1.525)
  Change at Week 56: number analyzed (Participants) | 69 | 67 | 65 | 59 | 71
  Change at Week 56 | -0.075 (0.587) | -0.137 (0.619) | -0.240 (0.599) | -0.136 (0.437) | -0.028 (0.477)

43. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Week 64 that were absent before treatment or that worsened relative to pre-treatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline up to Week 64
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
Participants
  AEs | 203 | 211 | 205 | 207 | 192 | 202 | 188 | 185 | 193 | 172
  SAEs | 22 | 23 | 28 | 30 | 22 | 22 | 23 | 26 | 34 | 21

44. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56: Observed Data
Description: The Neuropathy Impairment Score is the sum of scores over all 37 items from both the left and right side. The neurological impairment score assessed strength of groups of muscles of the head and neck, upper limbs and lower limbs, deep tendon reflexes and sensation (tactile, vibration, joint position sense, and pin prick) of index fingers and great toes through neurological examination. NIS calculated scoring muscle weakness (0=normal, 1=25% weak, 2=50% weak, 3=75% week, 3.25= move against gravity, 3.5=movement gravity eliminated, 3.75= muscle flicker no movement, 4=paralysis), scoring reflexes (0=normal, 1=reduced. 2=absent), scoring sensation (0=normal, 1=decreased, 2=absent). For NIS possible overall score (combined of both left and right sides of each domain), ranged from 0 (no impairment) to 244 (maximum impairment), higher scores indicated increased/more neuropathic deficits.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, and 56
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
units on a scale
  Baseline: number analyzed (Participants) | 285 | 288 | 280 | 287 | 282 | 256 | 254 | 256 | 253 | 255
  Baseline | 2.64 (5.96) | 2.56 (5.82) | 1.93 (4.34) | 2.54 (6.43) | 2.31 (6.34) | 2.04 (4.55) | 2.09 (4.00) | 2.24 (4.84) | 2.08 (4.86) | 2.18 (5.20)
  Change at Week 2: number analyzed (Participants) | 278 | 284 | 272 | 274 | 271 | 251 | 251 | 252 | 247 | 251
  Change at Week 2 | -0.20 (1.61) | -0.25 (2.27) | -0.30 (1.78) | -0.16 (1.98) | -0.11 (1.94) | -0.11 (1.87) | -0.29 (2.03) | -0.14 (1.60) | -0.33 (1.55) | -0.34 (1.17)
  Change at Week 4: number analyzed (Participants) | 269 | 274 | 263 | 268 | 264 | 244 | 239 | 245 | 242 | 248
  Change at Week 4 | -0.40 (1.93) | -0.42 (2.37) | -0.18 (1.68) | -0.29 (2.01) | -0.11 (2.20) | -0.20 (1.51) | -0.30 (1.93) | -0.41 (1.98) | -0.39 (2.27) | -0.11 (2.80)
  Change at Week 8: number analyzed (Participants) | 257 | 257 | 251 | 248 | 257 | 237 | 227 | 238 | 233 | 240
  Change at Week 8 | -0.47 (2.17) | -0.42 (2.40) | -0.22 (1.98) | -0.30 (2.05) | -0.12 (2.31) | -0.32 (2.05) | -0.36 (2.29) | -0.55 (2.08) | -0.22 (3.84) | -0.35 (2.06)
  Change at Week 12: number analyzed (Participants) | 248 | 253 | 248 | 236 | 240 | 230 | 222 | 232 | 228 | 232
  Change at Week 12 | -0.53 (2.38) | -0.38 (2.95) | -0.34 (2.28) | -0.62 (3.94) | -0.29 (2.65) | -0.52 (1.98) | -0.56 (2.37) | -0.72 (2.29) | -0.38 (3.84) | -0.44 (2.21)
  Change at Week 16: number analyzed (Participants) | 246 | 244 | 233 | 231 | 228 | 222 | 216 | 229 | 223 | 221
  Change at Week 16 | -0.81 (2.91) | -0.41 (2.62) | -0.38 (2.70) | -0.58 (2.82) | -0.26 (2.61) | -0.41 (2.25) | -0.64 (233) | -0.83 (2.41) | -0.48 (3.18) | -0.50 (2.47)
  Change at Week 24: number analyzed (Participants) | 224 | 224 | 219 | 223 | 212 | 198 | 217 | 211 | 211 | 207
  Change at Week 24 | -0.78 (3.26) | -0.50 (2.70) | -0.57 (2.27) | -0.57 (2.88) | -0.43 (2.52) | -0.37 (2.42) | -0.46 (2.47) | -0.99 (2.66) | -0.47 (2.83) | -0.50 (2.73)
  Change at Week 32: number analyzed (Participants) | 208 | 195 | 200 | 201 | 194 | 195 | 187 | 197 | 192 | 191
  Change at Week 32 | -0.56 (2.71) | -0.53 (2.64) | -0.78 (2.97) | -0.47 (3.51) | -0.39 (2.27) | -0.50 (2.61) | -0.71 (2.44) | -1.05 (2.97) | -0.49 (2.85) | -0.63 (2.72)
  Change at Week 40: number analyzed (Participants) | 186 | 174 | 179 | 175 | 178 | 179 | 173 | 177 | 172 | 179
  Change at Week 40 | -0.61 (2.37) | -0.47 (2.91) | -0.63 (2.75) | -0.38 (3.82) | -0.42 (2.77) | -0.42 (2.94) | -0.58 (2.37) | -1.06 (3.09) | -0.71 (2.73) | -0.73 (2.91)
  Change at Week 48: number analyzed (Participants) | 151 | 143 | 144 | 138 | 138 | 153 | 141 | 145 | 137 | 149
  Change at Week 48 | -0.55 (3.44) | -0.81 (2.56) | -0.67 (2.77) | -0.80 (3.46) | -0.48 (2.83) | -0.56 (2.74) | -0.65 (2.74) | -1.07 (3.49) | -0.50 (2.74) | -0.69 (3.14)
  Change at Week 56: number analyzed (Participants) | 83 | 83 | 83 | 70 | 72 | 76 | 69 | 69 | 72 | 83
  Change at Week 56 | -0.30 (5.01) | -0.70 (2.91) | -0.83 (4.14) | -0.10 (3.27) | -0.36 (2.68) | -0.53 (2.54) | -0.42 (2.51) | -1.01 (3.45) | -0.38 (2.04) | -0.54 (2.58)

45. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56: Last Observation Carried Forward (LOCF)
Description: as for outcome 44
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
units on a scale
  Baseline: number analyzed (Participants) | 285 | 288 | 280 | 287 | 282 | 256 | 254 | 256 | 253 | 255
  Baseline | 2.64 (5.96) | 2.56 (5.82) | 1.93 (4.34) | 2.54 (6.43) | 2.31 (6.34) | 2.04 (4.55) | 2.09 (4.00) | 2.24 (4.84) | 2.08 (4.86) | 2.18 (5.20)
  Change at Week 2: number analyzed (Participants) | 278 | 284 | 272 | 274 | 271 | 251 | 251 | 252 | 247 | 251
  Change at Week 2 | -0.20 (1.61) | -0.25 (2.27) | -0.30 (1.78) | -0.16 (1.98) | -0.11 (1.94) | -0.11 (1.87) | -0.29 (2.03) | -0.14 (1.60) | -0.33 (1.55) | -0.34 (1.71)
  Change at Week 4: number analyzed (Participants) | 282 | 287 | 275 | 284 | 277 | 253 | 251 | 254 | 250 | 252
  Change at Week 4 | -0.37 (1.88) | -0.46 (2.41) | -0.20 (1.66) | -0.33 (2.42) | -0.08 (2.20) | -0.21 (1.50) | -0.30 (1.90) | -0.40 (1.99) | -0.40 (2.24) | -0.13 (2.79)
  Change at Week 8: number analyzed (Participants) | 282 | 287 | 277 | 284 | 277 | 254 | 251 | 254 | 250 | 252
  Change at Week 8 | -0.49 (2.14) | -0.46 (2.38) | -0.25 (1.98) | -0.38 (2.51) | -0.12 (2.29) | -0.32 (2.00) | -0.35 (2.20) | -0.53 (2.06) | -0.33 (3.79) | -0.22 (2.96)
  Change at Week 12: number analyzed (Participants) | 282 | 287 | 277 | 284 | 277 | 254 | 251 | 254 | 250 | 252
  Change at Week 12 | -0.52 (2.33) | -0.43 (2.88) | -0.38 (2.25) | -0.65 (3.93) | -0.26 (2.54) | -0.53 (1.93) | -0.50 (2.34) | -0.69 (2.25) | -0.26 (4.78) | -0.28 (3.05)
  Change at Week 16: number analyzed (Participants) | 283 | 287 | 277 | 284 | 277 | 254 | 251 | 254 | 250 | 252
  Change at Week 16 | -0.77 (2.77) | -0.48 (2.58) | -0.35 (2.67) | -0.58 (3.02) | -0.18 (2.62) | -0.43 (2.15) | -0.56 (2.28) | -0.79 (2.35) | -0.30 (4.34) | -0.34 (3.20)
  Change at Week 24: number analyzed (Participants) | 283 | 287 | 277 | 284 | 277 | 254 | 251 | 254 | 250 | 252
  Change at Week 24 | -0.73 (3.07) | -0.57 (2.67) | -0.44 (2.21) | -0.60 (3.02) | -0.31 (2.49) | -0.35 (2.28) | -0.38 (2.31) | -0.90 (2.53) | -0.22 (4.47) | -0.36 (3.37)
  Change at Week 32: number analyzed (Participants) | 283 | 287 | 277 | 284 | 277 | 254 | 251 | 254 | 250 | 252
  Change at Week 32 | -0.56 (2.77) | -0.57 (2.77) | -0.52 (2.76) | -0.53 (3.41) | -0.32 (2.32) | -0.44 (2.38) | -0.56 (2.40) | -0.93 (2.72) | -0.26 (4.44) | -0.34 (3.46)
  Change at Week 40: number analyzed (Participants) | 283 | 287 | 278 | 284 | 277 | 254 | 251 | 254 | 250 | 252
  Change at Week 40 | -0.50 (2.65) | -0.55 (2.82) | -0.32 (2.56) | -0.49 (3.57) | -0.40 (2.73) | -0.41 (2.66) | -0.50 (2.37) | -0.50 (2.72) | -0.33 (4.34) | -0.39 (3.52)
  Change at Week 48: number analyzed (Participants) | 283 | 283 | 278 | 284 | 277 | 254 | 251 | 254 | 250 | 252
  Change at Week 48 | -0.43 (3.27) | -0.58 (2.71) | -0.38 (2.56) | -0.65 (3.20) | -0.43 (2.63) | -0.44 (2.40) | -0.52 (2.48) | -0.87 (2.90) | -0.34 (4.40) | -0.36 (3.51)
  Change at Week 56: number analyzed (Participants) | 283 | 287 | 278 | 284 | 277 | 254 | 251 | 254 | 250 | 252
  Change at Week 56 | -0.48 (3.83) | -0.53 (2.76) | -0.45 (2.95) | -0.58 (3.30) | -0.46 (2.72) | -0.41 (2.31) | -0.44 (2.58) | -0.89 (2.90) | -0.43 (4.45) | -0.41 (3.40)

46. Other Pre Specified Outcome: Number of Participants With Anti-Drug Antibody (ADA) Response
Description: Human serum ADA samples were analyzed for the presence or absence of anti--tanezumab antibodies by using a semi quantitative enzyme -linked immunosorbent assay (ELISA). Participants tested positive for ADA response on at least one post-baseline visit were reported. Participants with ADA titer level >=4.32 for tanezumab were considered ADA positive.
Time Frame: Baseline, Weeks 16, 40, 24, and 56
Population: ITT analysis set included all randomized participants who received at least 1 dose of IV study medication (tanezumab or matching placebo). Data was planned to be assessed and reported for combined population of naproxen and celecoxib cohort. This outcome measure was planned not to be analyzed for placebo reporting arms (Naproxen 500 mg and Celecoxib 100 mg).
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg (Naproxen or Celecoxib Exposure) | Tanezumab 10 mg (Naproxen or Celecoxib Exposure) | Tanezumab 5 mg + NSAID | Tanezumab 10 mg + NSAID
Number analyzed (Participants) | 541 | 542 | 536 | 542
Participants
  Baseline | 3 | 2 | 4 | 2
  Week 16 | 5 | 3 | 4 | 0
  Week 24 | 4 | 2 | 1 | 1
  Week 40 | 2 | 2 | 5 | 2
  Week 56 | 3 | 2 | 1 | 2

47. Secondary Outcome: Plasma Trough (Pre-dose) Concentration of Tanezumab
Time Frame: Predose on Day 1, Weeks 16, 24, 40, and 56
Population: Analysis was performed on ITT analysis set. Here, 'overall number of participants analyzed' signifies those participants who were evaluable for this outcome measure and Number analyzed' signifies participants evaluable at specified time points. Data was planned to be assessed and reported for combined population of naproxen and celecoxib cohort. This outcome measure was planned not to be analyzed for placebo reporting arms (Naproxen 500 mg and Celecoxib 100 mg).
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | Tanezumab 5 mg (Naproxen or Celecoxib Exposure) | Tanezumab 10 mg (Naproxen or Celecoxib Exposure) | Tanezumab 5 mg + NSAID | Tanezumab 10 mg + NSAID
Number analyzed (Participants) | 512 | 517 | 502 | 507
nanogram/milliliter
  Day 1 | 48.4570 (241.4173) | 164.068 (1045.628) | 102.398 (543.2856) | 96.4720 (481.0747)
  Week 16: number analyzed (Participants) | 426 | 413 | 421 | 410
  Week 16 | 222.779 (228.0336) | 556.854 (599.8115) | 255.246 (400.3175) | 723.316 (2791.080)
  Week 24: number analyzed (Participants) | 395 | 387 | 398 | 391
  Week 24 | 250.813 (375.3960) | 545.672 (375.3960) | 271.632 (368.0965) | 538.756 (481.1859)
  Week 40: number analyzed (Participants) | 295 | 259 | 272 | 257
  Week 40 | 231.840 (211.3920) | 523.214 (365.6468) | 263.049 (289.5641) | 527.108 (442.1378)
  Week 56: number analyzed (Participants) | 391 | 390 | 389 | 370
  Week 56 | 168.673 (307.1740) | 385.733 (456.5163) | 138.159 (253.3517) | 377.231 (422.0123)

48. Other Pre Specified Outcome: Number of Participants With Positive Urine or Serum Pregnancy Test
Description: Female participants, who reported positive in urine or serum pregnancy test were reported.
Time Frame: Baseline up to Week 56
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 200 | 208 | 184 | 192 | 199 | 192 | 184 | 179 | 177 | 189
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

49. Secondary Outcome: Number of Participants With Intravenous (IV) Doses of Study Medication
Description: Number of participants are reported based on the maximum number of IV doses of either tanezumab or placebo received.
Time Frame: Baseline up to Week 48
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Number analyzed (Participants) | 285 | 288 | 280 | 288 | 283 | 256 | 254 | 256 | 254 | 256
Participants
  Number of IV Doses: 1 | 32 | 36 | 36 | 44 | 35 | 25 | 30 | 22 | 21 | 22
  Number of IV Doses: 2 | 19 | 18 | 19 | 16 | 30 | 15 | 19 | 12 | 12 | 24
  Number of IV Doses: 3 | 27 | 28 | 17 | 21 | 21 | 13 | 16 | 18 | 22 | 12
  Number of IV Doses: 4 | 41 | 51 | 51 | 55 | 44 | 39 | 35 | 44 | 48 | 37
  Number of IV Doses: 5 | 71 | 70 | 66 | 74 | 74 | 82 | 78 | 84 | 72 | 73
  Number of IV Doses: 6 | 45 | 44 | 45 | 31 | 33 | 41 | 34 | 43 | 38 | 44
  Number of IV Doses: 7 | 50 | 41 | 46 | 47 | 46 | 41 | 42 | 33 | 41 | 44

ADVERSE EVENTS:
Description: Cases of osteonecrosis (ON) reported in this and other studies conducted up to 2010 were adjudicated post-hoc by an expert committee (2010-2012). Few of these events (2 of 87 reported ON cases), were confirmed as ON by the committee. Source: https://doi.org/10.1002/art.39492
Arm/Group | Tanezumab 5 mg (Naproxen Exposure) | Tanezumab 10 mg (Naproxen Exposure) | Tanezumab 5 mg + Naproxen 500 mg | Tanezumab 10 mg + Naproxen 500 mg | Naproxen 500 mg | Tanezumab 5 mg (Celecoxib Exposure) | Tanezumab 10 mg (Celecoxib Exposure) | Tanezumab 5 mg + Celecoxib 100 mg | Tanezumab 10 mg + Celecoxib 100 mg | Celecoxib 100 mg
Serious Adverse Events (participants affected / at risk) | 22/285 | 23/288 | 28/280 | 30/288 | 22/283 | 22/256 | 23/254 | 26/256 | 34/254 | 21/256
Other Adverse Events (participants affected / at risk) | 201/285 | 205/288 | 201/280 | 202/288 | 188/283 | 195/256 | 181/254 | 182/256 | 187/254 | 170/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 5 mg (Naproxen Exposure) (N=285) | Tanezumab 10 mg (Naproxen Exposure) (N=288) | Tanezumab 5 mg + Naproxen 500 mg (N=280) | Tanezumab 10 mg + Naproxen 500 mg (N=288) | Naproxen 500 mg (N=283) | Tanezumab 5 mg (Celecoxib Exposure) (N=256) | Tanezumab 10 mg (Celecoxib Exposure) (N=254) | Tanezumab 5 mg + Celecoxib 100 mg (N=256) | Tanezumab 10 mg + Celecoxib 100 mg (N=254) | Celecoxib 100 mg (N=256)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 2
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gallbladder pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2 | 2 | 0 | 1 | 3 | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 5 | 2 | 9 | 2 | 2 | 1 | 2 | 1 | 5 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nerve root compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 6 | 7 | 6 | 5 | 3 | 5 | 9 | 11 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 5 mg (Naproxen Exposure) (N=285) | Tanezumab 10 mg (Naproxen Exposure) (N=288) | Tanezumab 5 mg + Naproxen 500 mg (N=280) | Tanezumab 10 mg + Naproxen 500 mg (N=288) | Naproxen 500 mg (N=283) | Tanezumab 5 mg (Celecoxib Exposure) (N=256) | Tanezumab 10 mg (Celecoxib Exposure) (N=254) | Tanezumab 5 mg + Celecoxib 100 mg (N=256) | Tanezumab 10 mg + Celecoxib 100 mg (N=254) | Celecoxib 100 mg (N=256)
Anaemia (Blood and lymphatic system disorders) | 6 | 3 | 7 | 5 | 4 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 5 | 6 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 6 | 4 | 4 | 10 | 7 | 13 | 11 | 8
Nausea (Gastrointestinal disorders) | 8 | 2 | 8 | 1 | 3 | 6 | 1 | 4 | 5 | 9
Fatigue (General disorders) | 2 | 4 | 6 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 15 | 14 | 20 | 23 | 6 | 18 | 13 | 18 | 27 | 6
Bronchitis (Infections and infestations) | 8 | 5 | 5 | 2 | 4 | 7 | 6 | 5 | 9 | 6
Influenza (Infections and infestations) | 8 | 7 | 6 | 4 | 8 | 8 | 9 | 4 | 6 | 8
Nasopharyngitis (Infections and infestations) | 7 | 9 | 12 | 7 | 8 | 15 | 10 | 18 | 14 | 15
Sinusitis (Infections and infestations) | 6 | 6 | 6 | 4 | 11 | 8 | 6 | 5 | 6 | 10
Upper respiratory tract infection (Infections and infestations) | 11 | 11 | 14 | 10 | 14 | 11 | 8 | 8 | 13 | 16
Urinary tract infection (Infections and infestations) | 9 | 14 | 13 | 9 | 16 | 21 | 13 | 12 | 15 | 13
Fall (Injury, poisoning and procedural complications) | 5 | 10 | 12 | 14 | 8 | 13 | 8 | 12 | 11 | 7
Joint sprain (Injury, poisoning and procedural complications) | 1 | 6 | 3 | 8 | 2 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 7 | 10 | 13 | 7 | 9 | 6 | 5 | 5 | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 | 50 | 37 | 32 | 26 | 39 | 39 | 34 | 27 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 12 | 9 | 12 | 12 | 15 | 9 | 11 | 12 | 8
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 | 6 | 8 | 6 | 0 | 7 | 5 | 4 | 7 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 8 | 17 | 9 | 11 | 5 | 14 | 10 | 9 | 6 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 6 | 9 | 7 | 6 | 5 | 2 | 7 | 5 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 7 | 14 | 5 | 7 | 6 | 10 | 6 | 10 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 10 | 3 | 6 | 0 | 7 | 5 | 7 | 9 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 | 11 | 12 | 14 | 7 | 12 | 16 | 17 | 12 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 22 | 9 | 14 | 7 | 10 | 13 | 12 | 16 | 11
Carpal tunnel syndrome (Nervous system disorders) | 3 | 11 | 4 | 8 | 3 | 6 | 12 | 7 | 3 | 1
Decreased vibratory sense (Nervous system disorders) | 8 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 8 | 5 | 11 | 6 | 5 | 7 | 9 | 5 | 5 | 7
Headache (Nervous system disorders) | 9 | 18 | 7 | 7 | 5 | 20 | 13 | 15 | 9 | 16
Hypoaesthesia (Nervous system disorders) | 16 | 17 | 16 | 17 | 7 | 9 | 14 | 19 | 18 | 7
Paraesthesia (Nervous system disorders) | 14 | 28 | 17 | 35 | 8 | 19 | 11 | 31 | 25 | 9
Anxiety (Psychiatric disorders) | 2 | 6 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 6 | 2 | 2 | 2 | 7 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 2 | 8 | 5 | 8 | 6 | 10 | 4 | 6
Rash (Skin and subcutaneous tissue disorders) | 3 | 5 | 7 | 6 | 5 | 4 | 4 | 6 | 6 | 2
Hypertension (Vascular disorders) | 6 | 9 | 11 | 5 | 9 | 5 | 7 | 8 | 8 | 13
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 6 | 1 | 4
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 7 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 4 | 2 | 5
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 2 | 6 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 4 | 6 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 5 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.